CLINICAL TRIAL: NCT04040192
Title: A Phase 3, Randomized, Double-Blind, Vehicle-Controlled Study to Evaluate the Efficacy and Safety of Maintenance Treatment and Flare Reduction With Crisaborole Ointment, 2%, Once Daily Over 52 Weeks in Pediatric and Adult Participants (Ages 3 Months and Older) With Mild-to-Moderate Atopic Dermatitis, Who Responded to Twice Daily Crisaborole Ointment, 2%, Treatment
Brief Title: A Study to Evaluate Long-Term Maintenance Treatment With Once Daily Crisaborole Ointment 2% in Pediatric and Adult Participants With Mild-to-Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C3291035; 2019-000443-28 (EudraCT Number); CRISADE CONTROL (Other: Alias Study Number)
Record Dates: First submitted 2019-07-30; First posted 2019-07-31 (Actual); Results first posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Atopic Dermatitis
Keywords: Eczema; Crisaborole
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Crisaborole 2% (Experimental): Crisaborole 2% ointment applied once daily (QD)
  Interventions: Drug: Crisaborole 2%
- Vehicle (Placebo Comparator): Vehicle ointment applied once daily (QD)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Crisaborole 2% — Crisaborole ointment 2%
  Arms: Crisaborole 2%
Drug: Vehicle — Vehicle ointment
  Arms: Vehicle

SUMMARY:
This study will evaluate crisaborole therapy once daily (QD) as a long-term topical maintenance therapy for the reduction of flare in responders to crisaborole twice daily (BID) treatment.

DETAILED DESCRIPTION:
Approximately 700 participants will be enrolled in an run-in period to receive crisaborole, BID for up to a maximum of 8 weeks to identify crisaborole responders. A responder is defined as a participant who achieves both ISGA and EASI50 success. ISGA success is defined as achieving a score of 0 or 1 with at least 2 grade improvement from baseline; and the EASI50 success is defined as at least 50% improvement from baseline. Non responders at the end of the 8-week run-in period will be discontinued from the study.

Approximately 250 responders will be randomized (1:1 ratio) to enter the double-blind maintenance treatment period to receive crisaborole or vehicle QD for 52 weeks, with follow-up assessments every 4 weeks. If a flare occurs and if the participant meets the criteria for having a flare (ISGA ≥2), the participant will switch to enter a flare treatment period to receive open-label crisaborole BID for up to 12 weeks with follow-up assessments every 4 weeks. If the flare has resolved (ISGA ≤1) the participant will resume maintenance treatment and respective visit schedule. If a flare does not resolve after 3 consecutive treatment courses the participant will discontinue the study. A flare treatment period may comprise up to 3 consecutive treatment courses with crisaborole BID (each course is 4 weeks).

An end of study (EOS) safety follow-up is required 4 weeks after the last study treatment of any treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 3 months of age and older
* Confirmed diagnosis of atopic dermatitis according to Hanifin and Rajka criteria
* Minimum of 5% BSA affected by atopic dermatitis
* ISGA score of Mild (2) or Moderate (3)

Exclusion Criteria:

- Has any clinically significant medical disorder, condition, or disease (including active or potentially recurrent non AD dermatological conditions and known genetic dermatological conditions that overlap with AD, such as Netherton syndrome).

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 620 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (44):
- United States (25):
  - First OC Dermatology, Fountain Valley, California
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - Asthma and Allergy Associates, PC, Colorado Springs, Colorado
  - Colorado Springs Dermatology Clinic, PC, Colorado Springs, Colorado
  - Skin Care Research LLC, Boca Raton, Florida
  - Clinical Neuroscience Solutions, Inc, Jacksonville, Florida
  - Olympian Clinical Research, Largo, Florida
  - Baumann Cosmetic and Research Institute, Miami, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - Meridian Clinical Research, LLC, Baton Rouge, Louisiana
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - Skin Specialists PC, Omaha, Nebraska
  - Ohio Pediatric Research Association, Inc., Dayton, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Oklahoma State University - Center for Health Sciences, Tulsa, Oklahoma
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Innovate Research, LLC, Fort Worth, Texas
  - Austin Institute for Clinical Research, Houston, Texas
  - Austin Institute for Clinical Research, Inc., Pflugerville, Texas
  - Center for Clinical Studies, LTD. LLP, Webster, Texas
  - Jordan Valley Dermatology Center, South Jordan, Utah
  - PI-Coor Clinical Research LLC, Burke, Virginia
  - Dermatology Specialists of Spokane, Spokane, Washington
  - Principle Research Solutions, Spokane, Washington
- Australian Clinical Research Network, Maroubra, New South Wales, Australia
- Canada (5):
  - SimcoDerm Medical and Surgical Dermatology Center, Barrie, Ontario
  - Milestone Research , Inc, London, Ontario
  - North York Research Inc., North York, Ontario
  - Manna Research Toronto, Toronto, Ontario
  - Skinsense Medical Research, Saskatoon, Saskatchewan
- China (10):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Dermatology Hospital of Jiangxi Province, Nanchang, Jiangxi
  - Huashan Hospital Fudan University/Dermatology Department, Shanghai, Shanghai Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Hangzhou Third Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
- The Chaim Sheba Medical Center, Ramat Gan, Israel
- Turkey (Türkiye) (2):
  - Bezmialem Vakıf University Medical Faculty, Istanbul
  - Erciyes University Medical Faculty, Kayseri

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Eichenfield LF, Stein Gold LF, Lynde C, Guenther L, Greenberger S, Chu CY, Ghodsi Z, Vlahos B, Sanders P, Cha A, Canosa JM. Maintenance of Investigator's Static Global Assessment Response with Once-Daily Crisaborole in Participants with Mild to Moderate Atopic Dermatitis. Dermatol Ther (Heidelb). 2024 Apr;14(4):875-892. doi: 10.1007/s13555-024-01129-9. Epub 2024 Mar 28. PMID 38546803
- [Derived] Eichenfield LF, Gower RG, Xu J, Alam MS, Su JC, Myers DE, Sanders P, Vlahos B, Zang C, Lan J, Werth J. Once-Daily Crisaborole Ointment, 2%, as a Long-Term Maintenance Treatment in Patients Aged >/= 3 Months with Mild-to-Moderate Atopic Dermatitis: A 52-Week Clinical Study. Am J Clin Dermatol. 2023 Jul;24(4):623-635. doi: 10.1007/s40257-023-00780-w. Epub 2023 May 15. PMID 37184828
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3291035

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 620 participants signed the informed consent form and were enrolled in the study. 78 participants were screen failures who did not meet eligibility criteria. 542 participants were not screen failures, of which only 497 were assigned to study treatment.
Groups:
- Crisaborole 2% Twice Daily (BID): Participants with mild to moderate atopic dermatitis (AD) were administered crisaborole 2% ointment applied topically BID for maximum duration of up to 8 weeks in open label (OL) run-in period.
- Vehicle Once Daily (QD): Participants identified as responders during the OL period were randomized to receive vehicle applied topically once daily (QD) for 52 weeks in the double-blind (DB) maintenance period. If any participant developed flares during the DB maintenance period, the participant was switched to receive flare rescue treatment with crisaborole 2% ointment BID in an open-label manner until resolution of flares following which DB treatment with vehicle was resumed.
- Crisaborole 2% QD: Participants identified as responders during the OL period were randomized to receive crisaborole 2% ointment applied topically QD for 52 weeks in the DB maintenance period. If any participant developed flares during the DB maintenance period, the participant was switched to receive flare rescue treatment with crisaborole 2% ointment BID in an open-label manner until resolution of flares following which DB treatment with crisaborole 2% QD was resumed.
Period: Open Label Run-in Period (up to 8 Weeks)
Arm/Group | Crisaborole 2% Twice Daily (BID) | Vehicle Once Daily (QD) | Crisaborole 2% QD
Started | 497 | 0 | 0
Completed | 270 (Participants were randomized to DB period.) | 0 | 0
Not Completed | 227 | 0 | 0
Not completed — Adverse Event | 18 | 0 | 0
Not completed — Lost to Follow-up | 14 | 0 | 0
Not completed — Physician Decision | 3 | 0 | 0
Not completed — Protocol Violation | 3 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 0 | 0
Not completed — Withdrawal by parent/guardian | 18 | 0 | 0
Not completed — Failure to meet randomization criteria | 152 | 0 | 0
Not completed — Other | 11 | 0 | 0
Period: Double Blind Period (up to 52 Weeks)
Arm/Group | Crisaborole 2% Twice Daily (BID) | Vehicle Once Daily (QD) | Crisaborole 2% QD
Started | 0 (In DB period, participants were randomized to receive Vehicle QD and Crisaborole 2% QD.) | 135 (Crisaborole responders in OL period were randomized to Vehicle QD arm.) | 135 (Crisaborole responders in OL period were randomized to Crisaborole 2% QD arm.)
Completed | 0 | 78 | 78
Not Completed | 0 | 57 | 57
Not completed — Adverse Event | 0 | 3 | 1
Not completed — Lost to Follow-up | 0 | 6 | 10
Not completed — Physician Decision | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 6 | 11
Not completed — Withdrawal by parent/guardian | 0 | 8 | 7
Not completed — Other | 0 | 29 | 18
Not completed — Pregnancy | 0 | 2 | 0
Not completed — Missing | 0 | 2 | 5

BASELINE CHARACTERISTICS:
Population: Evaluable OL population comprised of all participants who received at least 1 dose of study intervention in the OL period.
Groups:
- Crisaborole 2% BID: Participants with mild to moderate AD were administered crisaborole 2% ointment applied topically BID for maximum duration of up to 8 weeks in OL run-in period. Participants identified as responders during the OL period were randomized to receive vehicle or crisaborole 2% ointment applied topically QD for 52 weeks in the DB maintenance period.
Arm/Group | Crisaborole 2% BID
Number analyzed (Participants) | 497
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Here, number analyzed signifies number of participants evaluable for specified rows. i.e., Crisaborole 2% BID arm including all participants who were enrolled and received at least 1 dose of study intervention in OL run-in period and Vehicle QD and Crisaborole 2% QD arms including all participants who were randomized to the respective arms in DB period.
  Years
    Crisaborole 2% BID | 19.89 (18.443)
    Vehicle QD: number analyzed (Participants) | 135
    Vehicle QD | 21.76 (20.373)
    Crisaborole 2% QD: number analyzed (Participants) | 135
    Crisaborole 2% QD | 22.62 (20.175)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Here, number analyzed signifies number of participants evaluable for specified rows. i.e., Crisaborole 2% BID arm including all participants who were enrolled and received at least 1 dose of study intervention in OL run-in period and Vehicle QD and Crisaborole 2% QD arms including all participants who were randomized to the respective arms in DB period.
  Participants
    Crisaborole 2% BID: Female | 283
    Crisaborole 2% BID: Male | 214
    Vehicle QD: number analyzed (Participants) | 135
    Vehicle QD: Female | 76
    Vehicle QD: Male | 59
    Crisaborole 2% QD: number analyzed (Participants) | 135
    Crisaborole 2% QD: Female | 71
    Crisaborole 2% QD: Male | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Here, number analyzed signifies number of participants evaluable for specified rows. i.e., Crisaborole 2% BID arm including all participants who were enrolled and received at least 1 dose of study intervention in OL run-in period and Vehicle QD and Crisaborole 2% QD arms including all participants who were randomized to the respective arms in DB period.
  Participants
    Crisaborole 2% BID: Hispanic or Latino | 54
    Crisaborole 2% BID: Not Hispanic or Latino | 426
    Crisaborole 2% BID: Unknown or Not Reported | 17
    Vehicle QD: number analyzed (Participants) | 135
    Vehicle QD: Hispanic or Latino | 10
    Vehicle QD: Not Hispanic or Latino | 120
    Vehicle QD: Unknown or Not Reported | 5
    Crisaborole 2% QD: number analyzed (Participants) | 135
    Crisaborole 2% QD: Hispanic or Latino | 19
    Crisaborole 2% QD: Not Hispanic or Latino | 110
    Crisaborole 2% QD: Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Here, number analyzed signifies number of participants evaluable for specified rows. i.e., Crisaborole 2% BID arm including all participants who were enrolled and received at least 1 dose of study intervention in OL run-in period and Vehicle QD and Crisaborole 2% QD arms including all participants who were randomized to the respective arms in DB period.
  Participants
    Crisaborole 2% BID: American Indian or Alaska Native | 2
    Crisaborole 2% BID: Asian | 101
    Crisaborole 2% BID: Native Hawaiian or Other Pacific Islander | 1
    Crisaborole 2% BID: Black or African American | 161
    Crisaborole 2% BID: White | 204
    Crisaborole 2% BID: More than one race | 18
    Crisaborole 2% BID: Unknown or Not Reported | 10
    Vehicle QD: number analyzed (Participants) | 135
    Vehicle QD: American Indian or Alaska Native | 0
    Vehicle QD: Asian | 27
    Vehicle QD: Native Hawaiian or Other Pacific Islander | 0
    Vehicle QD: Black or African American | 47
    Vehicle QD: White | 54
    Vehicle QD: More than one race | 7
    Vehicle QD: Unknown or Not Reported | 0
    Crisaborole 2% QD: number analyzed (Participants) | 135
    Crisaborole 2% QD: American Indian or Alaska Native | 2
    Crisaborole 2% QD: Asian | 28
    Crisaborole 2% QD: Native Hawaiian or Other Pacific Islander | 1
    Crisaborole 2% QD: Black or African American | 42
    Crisaborole 2% QD: White | 55
    Crisaborole 2% QD: More than one race | 4
    Crisaborole 2% QD: Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Duration of Flare-Free Maintenance Until Onset of First-Flare During the Double Blind (DB) Period
Description: The duration of flare-free maintenance was the time from randomization to the last Investigator's Static Global Assessment (ISGA) and was right censored, if an intercurrent event (eg, death, dropout, loss to follow up, or end of study) occurred before the first flare. When a flare occurred first, the duration of flare free maintenance was the time from randomization to the first flare and was not censored. Duration of flare free maintenance was estimated using the Kaplan-Meier method.
Time Frame: From randomization to first flare or last ISGA assessment (up to 52 weeks)
Population: Evaluable-DB (Eval-DB) population included all randomized participants with success in ISGA (i.e., achieving a score of clear [0] or almost clear [1] with a >=2 grade improvement from the run-in baseline) and Eczema Area Severity Index score (EASI50) criteria as responders at randomization and received at least 1 dose of study intervention in the DB period.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Vehicle QD: Participants identified as responders during the OL period were randomized to receive vehicle applied topically QD for 52 weeks in the DB maintenance period. Participants who developed flares during the DB maintenance period were switched to receive crisaborole 2% ointment BID in an open-label manner until resumption of DB treatment with vehicle.
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 129 | 125
Days | 30 (28) [28 to 56] | 111 (56) [56 to 224]
Statistical Analysis 1: Comparison: Vehicle QD vs Crisaborole 2% QD; Test type: Other; p = 0.0034, Log Rank — p-value was estimated by the log-rank test, stratified by age group, duration of the BID treatment in OL period, and ISGA score at randomization

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE was considered a TEAE if the event started on or after the treatment period start date and before end of study (at least 28 days after last dose of study intervention).
Time Frame: Crisaborole 2% BID: From start of study intervention in OL period up to 8 weeks ; Vehicle QD and crisaborole 2% QD: From start of study intervention in DB period up to 28 days after last dose of study intervention (maximum of 56 weeks)
Population: Safety population comprised of all participants who received at least 1 dose of study intervention during the study.
Measure: Count of Participants; unit: Participants
Groups:
- Crisaborole 2% BID: Participants with mild to moderate AD were administered crisaborole 2% ointment applied topically BID for maximum duration of up to 8 weeks in OL run-in period.
Arm/Group | Crisaborole 2% BID | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 497 | 135 | 135
Participants | 109 | 49 | 36

3. Secondary Outcome: Number of Flare-Free Days During the DB Period
Description: Flare - free days was the sum of the duration of flare-free maintenance during the DB maintenance period for each participant.
Time Frame: Up to maximum of 52 weeks
Population: Eval-DB population included all randomized participants with success in ISGA and EASI50 criteria as responders at randomization and received at least 1 dose of study intervention in the DB period.
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 129 | 125
Days | 199.42 (11.824) [lower limit 11.824] | 234.01 (12.323) [lower limit 12.323]
Statistical Analysis 1: Comparison: Vehicle QD vs Crisaborole 2% QD; Test type: Other — Analysis of covariance (ANCOVA) model included fixed effects of treatment group, age group, duration of the BID treatment in OL period, and ISGA score at randomization; p = 0.0346, ANCOVA; Least square mean difference = 34.59, 95% CI 2-sided [2.53 to 66.64], Standard Error of Mean 16.274

4. Secondary Outcome: Number of Flares During the DB Period
Description: Flare was defined as an ISGA score of >=2. The ISGA is a 5-point scale (range 0 to 4), reflecting a global assessment of AD severity based on erythema, induration/papulation, and oozing/crusting. ISGA score of 2: mild (faint pink erythema with mild induration/papulation and no oozing/crusting) 3: moderate (pink-red erythema with moderate induration/papulation with or without oozing/crusting) and 4: severe (deep or bright red erythema with severe induration/papulation and with oozing/crusting).
Time Frame: Up to maximum of 52 weeks
Population: as for outcome 3
Measure: Median (Full Range); unit: Flares
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 129 | 125
Flares | 1.00 [0 to 6] | 1.00 [0 to 4]
Statistical Analysis 1: Comparison: Vehicle QD vs Crisaborole 2% QD; Test type: Other; p = 0.0042, Wilcoxon (Mann-Whitney) — p-value was estimated by Wilcoxon rank sum test stratified by age group, duration of the BID treatment in OL period, and ISGA score at randomization; Median Difference (Final Values) = -0.50, 95% CI 2-sided [-1.00 to 0.00] — Median difference and 95%CI were estimated using Hodges-Lehmann method

5. Secondary Outcome: Secondary: Duration of Pruritus Response Maintenance Until Onset of First Flare During the DB Period: Participants Aged >=12 Years With Baseline Peak Pruritus Numerical Rating Scale (PP NRS) >=3, >=4 and >=3, >=4 Points Reduction in PP NRS
Description: Duration of pruritus response maintenance=time from randomization to loss of pruritus response or first flare onset(ISGA>=2) during 52-week DB period evaluated among pruritus responders at randomization. Responders=participants with success in ISGA and EASI50 criteria. Pruritus response maintenance=maintenance of >=50% improvement in pruritus from baseline obtained at randomization. If event (e.g., death, first flare[ISGA >=2], lost to follow up or end of study) occurred before loss of pruritus response for first flare-free period, duration of pruritus response maintenance was time from randomization to last assessment and was censored. Here,pruritus response maintenance duration was presented for participants aged >=12 years with OL baseline PP NRS >=3, >=4 and >=3, >=4 points reduction from OL baseline to randomization in PP NRS. PP NRS: Participants were asked to rate their itch at worst moment during previous 24 hours on a scale of 0 to 10; 0=no itch and 10=worst itch imaginable".
Time Frame: From randomization up to loss of pruritus response or onset of first flare or the last assessment (maximum of 52 weeks)
Population: Eval-DB population included all randomized participants with success in ISGA and EASI50 criteria as responders at randomization and received at least 1 dose of study intervention in the DB period. Here, '"Overall Number of Participants Analyzed'' signifies number of participants evaluable for this outcome measure and "Number Analyzed'' signifies participants evaluable for specified rows.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 25 | 37
Days
  Baseline PP NRS >=3 and >=3 point reduction in PP NRS | NA [18 to NA] — Median and upper limit of 95 % CI could not be estimated due to less number of participants with events. | 164 [105 to NA] — Upper limit of 95 % CI could not be estimated due to less number of participants with events.
  Baseline PP NRS >=4 and >=4 point reduction in PP NRS: number analyzed (Participants) | 18 | 24
  Baseline PP NRS >=4 and >=4 point reduction in PP NRS | NA [16 to NA] — Median and upper limit of 95 % CI could not be estimated due to less number of participants with events. | 309 [141 to NA] — Upper limit of 95 % CI could not be estimated due to less number of participants with events.
Statistical Analysis 1: Comparison: Vehicle QD vs Crisaborole 2% QD; Baseline PP NRS >=3 and >=3 point reduction in PP NRS; Test type: Other; p = 0.6815, Log Rank — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Vehicle QD vs Crisaborole 2% QD; Baseline PP NRS >=4 and >=4 point reduction in PP NRS; Test type: Other; p = 0.1518, Log Rank — [p-value comment as in outcome 1, analysis 1]

6. Secondary Outcome: Secondary: Duration of Pruritus Response Maintenance Until Onset of First Flare During the DB Period: Participants Aged 6 to <12 Years With Baseline Patient Reported Itch Severity (PRIS) >=2 and >=2 Points Reduction in PRIS
Description: Duration of pruritus response maintenance=time from randomization to loss of pruritus response or first flare onset (ISGA>=2) during 52-week DB period. Evaluated among pruritus responders at randomization. Responders were defined as participants with success in ISGA and EASI50 criteria. Pruritus response maintenance=maintenance of >=50% improvement in pruritus from baseline that was obtained at randomization. If an event (e.g., death, first flare [ISGA >=2], lost to follow up, or end of study) occurred before loss of pruritus response for first flare-free period, duration of maintenance of pruritus response was time from randomization to last assessment and was censored. Here, pruritus response maintenance duration was presented for participants aged 6 to <12 years with baseline PRIS >=2 and >=2 points reduction from baseline to randomization in PRIS. PRIS: a 5-point scale (range: 0=no itch to 4=worst itch imaginable) and was completed by participants.
Time Frame: From randomization up to loss of pruritus response or onset of first flare or the last assessment (maximum of 52 weeks)
Population: Eval-DB population included all randomized participants with success in ISGA and EASI50 criteria as responders at randomization and received at least 1 dose of study intervention in the DB period. Here, ''Overall Number of Participants Analyzed'' signifies number of participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 10 | 2
Days | NA [2 to NA] — Median and upper limit of 95 % CI could not be estimated due to less number of participants with events. | 133 [28 to 238]
Statistical Analysis 1: Comparison: Vehicle QD vs Crisaborole 2% QD; Test type: Other; p = 0.1933, Log Rank — [p-value comment as in outcome 1, analysis 1]

7. Secondary Outcome: Duration of Pruritus Response Maintenance Until Onset of First Flare During the DB Period: Observer Reported Itch Severity Scale (ORIS) in Participants Aged 3 to <6 Months
Description: Duration of pruritus response maintenance=time from randomization to loss of pruritus response or first flare onset(ISGA>=2)during52-weekDB period. Evaluated among pruritus responders (success in ISGA, EASI 50) at randomization. Pruritus response maintenance=maintenance of >=50% improvement in pruritus from baseline obtained at randomization. If event(e.g., death, first flare[ISGA >=2], lost to follow up, or end of study) occurred before loss of pruritus response for first flare-free period, duration of maintenance of pruritus response was time from randomization to last assessment and was censored. Here, pruritus response maintenance duration was presented for participants aged 3 to <6 months with OL baseline ORIS>=3 or >=4 and >=3 or >=4 points reduction from OL baseline to randomization in ORIS. Caregivers were asked to rate observation of their child's itch(scratching, rubbing) at worst moment during previous 24 hours on a scale of 0 to 10;0=no itch,10=worst itch imaginable.
Time Frame: From randomization up to loss of pruritus response or onset of first flare or the last assessment (maximum of 52 weeks)
Population: Eval-DB population included all randomized participants with success in ISGA and EASI50 criteria as responders at randomization and received at least 1 dose of study intervention in the DB period. Here, ''Overall Number of Participants Analyzed'' signifies number of participants evaluable for this outcome measure and ''number of participants analyzed'' signifies participants evaluable at specified rows.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 20 | 10
Days
  Baseline ORIS Scale >=3 and >=3 point reduction | 7 [4 to NA] — Upper limit of 95 % CI could not be estimated due to insufficient number of participants with events. | NA [2 to NA] — Median and upper limit of 95 % CI could not be estimated due to insufficient number of participants with events.
  Baseline ORIS Scale >=4 and >=4 point reduction: number analyzed (Participants) | 12 | 8
  Baseline ORIS Scale >=4 and >=4 point reduction | 8 [4 to NA] — Upper limit of 95 % CI could not be estimated due to insufficient number of participants with events. | NA [2 to NA] — Median and upper limit of 95 % CI could not be estimated due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Vehicle QD vs Crisaborole 2% QD; Baseline ORIS Scale >=3 and >=3 point reduction; Test type: Other — p-value was estimated by the log-rank test, stratified by age group, duration of the BID treatment in OL period, and ISGA score at randomization; p = 0.3778, Log Rank
Statistical Analysis 2: Comparison: Vehicle QD vs Crisaborole 2% QD; Baseline ORIS Scale >=4 and >=4 point reduction; Test type: Other — [test comment as in outcome 7, analysis 1]; p = 0.4870, Log Rank

8. Secondary Outcome: Duration of Maintenance of >=50% Reduction in Eczema Area and Severity Index (EASI) Total Score Until Onset of First Flare During the DB Period
Description: EASI assessed severity of AD, based on severity of lesion clinical signs (erythema [E], induration/papulation [I], excoriation [Ex], lichenification [L]) and % body surface area (BSA) affected. Each of clinical signs scored separately for each of 4 body regions (head and neck [h], upper limbs [u], trunk [t] [including axillae and groin], lower limbs [l] [including buttocks]) on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score (A) according to %BSA with AD: 0 (0%), 1(>0 to <10%), 2(10 to <30%), 3(30 to <50%), 4(50 to <70%), 5(70 to <90%), 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh + Ih + Exh + Lh) + 0.2*Au*(Eu + Iu + ExU + Lu) + 0.3*At*(Et +It + Ext + Lt) + 0.4*Al*(El + Il + Exl + Ll). Total EASI score ranged from 0.0 to 72.0, higher score = greater severity of AD. EASI response maintenance = score that does not lose more than 50% of achieved reduction from Day1/Baseline run-in EASI score.
Time Frame: From randomization to loss of EASI response or onset of first flare or the last EASI assessment (up to maximum of 52 weeks)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 129 | 125
Days | 198 [84 to NA] — Upper limit of 95%CI could not be estimated due to insufficient number of participants with events. | NA [175 to NA] — Upper limit of 95%CI could not be estimated due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Vehicle QD vs Crisaborole 2% QD; Test type: Other; p = 0.1159, Log Rank — [p-value comment as in outcome 1, analysis 1]

9. Secondary Outcome: Duration of Maintenance of Dermatology Life Quality Index (DLQI) Response Until Onset of First Flare During the DB Period
Description: Duration of DLQI maintenance=time from randomization to loss of DLQI response during 52-week DB period for responders at randomization. If event(e.g., death, first flare[ISGA >=2], lost to follow up or end of study) occurred before loss of DLQI response, duration of maintenance of DLQI response=time from randomization to last assessment and censored. Responders=participants with success in ISGA,EASI50 criteria. DLQI response maintenance=response that does not lose more than minimal clinical important difference. DLQI =10-item questionnaire, measured impact of skin disease in participants aged >=16 years. Children's DLQI (CDLQI): participants aged 4 to15 years. Each question in DLQI and CDLQI evaluated on 4-point scale (range 0=not at all to 3=very much). Scores from10 items were added for DLQI/CDLQI total score, range:0 (not at all) to 30 (very much). Higher scores=more impact on quality of life of participants/children.
Time Frame: From randomization to loss of DLQI response or onset of first flare or the last assessment up to first flare (up to maximum of 52 weeks)
Population: Eval-DB population included all randomized participants with success in ISGA and EASI50 criteria as responders at randomization and received at least 1 dose of study intervention in the DB period. Here, ''Overall Number of Participants Analyzed'' signifies number of participants evaluable for this outcome measure and ''number of participants analyzed'' signifies participants evaluable for specified rows.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 105 | 105
Days
  DLQI for participants >=16 years of age: number analyzed (Participants) | 51 | 54
  DLQI for participants >=16 years of age | NA [111 to NA] — Median and upper limit of 95%CI could not be estimated due to insufficient number of participants with events. | NA [187 to NA] — Median and upper limit of 95%CI could not be estimated due to insufficient number of participants with events.
  Children's DLQI: participants 4-<16 yrs of age: number analyzed (Participants) | 54 | 51
  Children's DLQI: participants 4-<16 yrs of age | NA [360 to NA] — Median and upper limit of 95%CI could not be estimated due to insufficient number of participants with events. | NA [271 to NA] — Median and upper limit of 95%CI could not be estimated due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Vehicle QD vs Crisaborole 2% QD; DLQI for participants >=16 years of age; Test type: Other; p = 0.6973, Log Rank — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Vehicle QD vs Crisaborole 2% QD; Children's DLQI: participants 4-<16 yrs of age; Test type: Other; p = 0.7456, Log Rank — [p-value comment as in outcome 1, analysis 1]

10. Secondary Outcome: Duration of Maintenance of Patient Oriented Eczema Measure (POEM) Response Until Onset of First Flare During the DB Period
Description: POEM was a 7-item participant reported outcome measure used to assess the impact of AD (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) over the past week. Each item was scored as: no days=0, 1-2 days=1, 3-4 days=2, 5-6 days=3 and every day=4. The total score ranged from 0 to 28, where higher score indicated greater severity. POEM response maintenance was defined as the response that does not lose more than minimal clinical important difference. Duration of POEM maintenance was time from randomization to loss of POEM response during 52-week DB period for responders at randomization. Responders were defined as participants with success in ISGA and EASI50 criteria. If an event (e.g., death, first flare [ISGA >=2], lost to follow up, or end of study) occurred before loss of POEM response, duration of maintenance of POEM response was time from randomization to last assessment and was censored. Proxy POEM was used for participants aged 3 months to <12 years.
Time Frame: From randomization to loss POEM response or onset of first flare or the last assessment up to the first flare (up to maximum of 52 weeks)
Population: Eval-DB population included all randomized participants with success in ISGA and EASI50 criteria as responders at randomization and received at least 1 dose of study intervention in the DB period. Here, ''Overall Number of Participants Analyzed'' signifies number of participants evaluable for this outcome measure and ''Number Analyzed'' signifies participants evaluable for specified rows.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 125 | 122
Days
  POEM: number analyzed (Participants) | 67 | 76
  POEM | 55 [25 to 222] | 180 [69 to 322]
  Proxy POEM: number analyzed (Participants) | 58 | 46
  Proxy POEM | 20 [13 to 124] | 150 [33 to NA] — Upper limit of 95%CI could not be estimated due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Vehicle QD vs Crisaborole 2% QD; POEM; Test type: Other; p = 0.0513, Log Rank — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Vehicle QD vs Crisaborole 2% QD; Proxy POEM; Test type: Other; p = 0.0217, Log Rank — [p-value comment as in outcome 1, analysis 1]

11. Secondary Outcome: Investigator's Static Global Assessment (ISGA) Score for the First Flare Period
Description: ISGA:5- point global assessment scale of AD severity, used to characterize overall disease severity across all treatable AD lesions (excluding the scalp). Score ranged from 0 to 4: where 0= clear(minor residual hypo/hyperpigmentation; no erythema or induration/papulation; no oozing/crusting), 1= almost clear (trace faint pink erythema, with barely perceptible induration/papulation and no oozing/crusting), 2= mild (faint pink erythema with mild induration/papulation and no oozing/crusting), 3= moderate (pink-red erythema with moderate induration/papulation with or without oozing/crusting), 4= severe (deep or bright red erythema with severe induration/papulation and with oozing/crusting). Higher scores indicate greater severity of AD. First flare period was the time from the onset of flare (ISGA>=2) during DB maintenance period where the participant was switched to receive open-label crisaborole ointment 2%, BID for up to 12 weeks until resolution of flares.
Time Frame: Week 0 (Day 1), Week 4, Week 8 and Week 12
Population: Eval-DB population included all randomized participants with success in ISGA and EASI50 criteria as responders at randomization and received at least 1 dose of study intervention in the DB period. Here, ''Overall Number of Participants Analyzed'' signifies number of participants evaluable for this outcome measure and ''Number Analyzed'' signifies participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 96 | 81
Units on a scale
  Week 0 | 2.4 (0.51) | 2.3 (0.47)
  Week 4: number analyzed (Participants) | 53 | 47
  Week 4 | 2.2 (0.45) | 2.2 (0.41)
  Week 8: number analyzed (Participants) | 33 | 27
  Week 8 | 2.1 (0.33) | 2.4 (0.57)
  Week 12: number analyzed (Participants) | 10 | 11
  Week 12 | 2.3 (0.48) | 2.5 (0.52)

12. Secondary Outcome: EASI Score for the First Flare Period
Description: EASI assessed severity of AD, based on severity of lesion clinical signs (erythema[E], induration/papulation[I], excoriation[Ex], lichenification[L]) and % body surface area(BSA) affected.Each of clinical signs scored separately for each of 4 body regions (head and neck[h], upper limbs[u], trunk[t] [including axillae and groin], lower limbs[l] [including buttocks]) on 4-point scale: 0= absent; 1=mild; 2= moderate; 3= severe.EASI area score(A) according to %BSA with AD: 0 (0%), 1(>0 to <10%), 2(10 to <30%), 3(30 to <50%), 4(50 to <70%), 5(70 to <90%), 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh + Ih + Exh + Lh) + 0.2*Au*(Eu + Iu + ExU + Lu) + 0.3*At*(Et +It + Ext + Lt) + 0.4*Al*(El + Il + Exl + Ll). Total EASI score ranged from 0.0 to 72.0, higher score = greater severity of AD.First flare period=time from onset of flare(ISGA>=2) during DB maintenance period where participant was switched to receive open-label crisaborole ointment 2%,BID for up to 12 weeks until resolution of flares.
Time Frame: Week 0 (Day 1), Week 4, Week 8 and Week 12
Population: Eval-DB population included all randomized participants with success in ISGA and EASI50 criteria as responders at randomization and received at least 1 dose of study intervention in the DB period. Here, ''Overall Number of Participants Analyzed'' signifies number of participants evaluable for this outcome measure and ''Number of Participants Analyzed'' signifies participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 96 | 81
Units on a scale
  Week 0 | 6.53 (5.897) | 5.27 (3.933)
  Week 4: number analyzed (Participants) | 54 | 47
  Week 4 | 6.09 (5.471) | 5.02 (3.869)
  Week 8: number analyzed (Participants) | 33 | 27
  Week 8 | 4.84 (5.322) | 5.66 (4.459)
  Week 12: number analyzed (Participants) | 10 | 11
  Week 12 | 6.25 (4.546) | 6.56 (5.647)

13. Secondary Outcome: Duration (Days) of Flare Period
Description: Duration of flare period was average duration calculated from sum of durations divided by number of flares for each participant.
Time Frame: Up to 52 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 96 | 81
Days | 54.2 (28.77) [lower limit 28.77] | 55.3 (35.73) [lower limit 35.73]

14. Secondary Outcome: Percent Change From Baseline in EASI Scores at Weeks 2, 4, 6 and 8: OL Run-in Period
Description: EASI assessed severity of AD, based on severity of lesion clinical signs (erythema [E], induration/papulation [I], excoriation [Ex], lichenification [L]) and % body surface area (BSA) affected. Each of clinical signs scored separately for each of 4 body regions (head and neck [h], upper limbs [u], trunk [t] [including axillae and groin], lower limbs [l] [including buttocks]) on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score (A) according to %BSA with AD: 0 (0%), 1(>0 to <10%), 2(10 to <30%), 3(30 to <50%), 4(50 to <70%), 5(70 to <90%), 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh + Ih + Exh + Lh) + 0.2*Au*(Eu + Iu + ExU + Lu) + 0.3*At*(Et +It + Ext + Lt) + 0.4*Al*(El + Il + Exl + Ll). Total EASI score ranged from 0.0 to 72.0, higher score = greater severity of AD.
Time Frame: Baseline (last observation up to and including Day 1 of OL period), Weeks 2, 4, 6 and 8
Population: Evaluable-OL (Eval-OL) population included all participants that received at least 1 dose of study intervention in the OL period.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Crisaborole 2% BID
Number analyzed (Participants) | 497
Percent change
  Week 2 | -31.44 (37.151)
  Week 4 | -38.52 (44.448)
  Week 6 | -45.35 (49.453)
  Week 8 | -52.86 (51.209)

15. Secondary Outcome: Percent Change From Baseline in EASI Scores at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52: DB Period
Description: as for outcome 14
Time Frame: Baseline (last observation up to and including the randomization day), Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Crisaborole 2% BID: Flare Period: Participants with an onset of flare (ISGA>=2) during DB maintenance period were switched to receive open-label crisaborole ointment 2%, BID for up to 12 weeks until resolution of flares and resumption of DB maintenance treatment.
Arm/Group | Vehicle QD | Crisaborole 2% QD | Crisaborole 2% BID: Flare Period
Number analyzed (Participants) | 129 | 125 | 175
Percent change
  Week 4: number analyzed (Participants) | 38 | 57 | 78
  Week 4 | 2.87 (72.981) | -10.16 (61.161) | 407.52 (562.691)
  Week 8: number analyzed (Participants) | 42 | 53 | 69
  Week 8 | 1.04 (95.062) | 34.26 (224.615) | 239.90 (321.514)
  Week 12: number analyzed (Participants) | 44 | 50 | 54
  Week 12 | -0.11 (126.465) | -8.22 (93.118) | 401.37 (937.078)
  Week 16: number analyzed (Participants) | 53 | 57 | 36
  Week 16 | 26.30 (156.188) | 27.98 (282.035) | 272.90 (314.387)
  Week 20: number analyzed (Participants) | 8 | 6 | 21
  Week 20 | 26.38 (147.113) | -45.44 (54.768) | 264.70 (341.948)
  Week 24: number analyzed (Participants) | 46 | 50 | 32
  Week 24 | -20.62 (78.665) | 6.94 (162.911) | 270.22 (314.301)
  Week 28: number analyzed (Participants) | 9 | 5 | 22
  Week 28 | 19.17 (112.841) | -33.04 (31.617) | 453.99 (848.739)
  Week 32: number analyzed (Participants) | 44 | 45 | 27
  Week 32 | 13.57 (131.633) | -19.33 (81.663) | 341.18 (500.843)
  Week 36: number analyzed (Participants) | 3 | 4 | 20
  Week 36 | -55.95 (51.052) | 211.13 (155.547) | 184.26 (195.695)
  Week 40: number analyzed (Participants) | 40 | 40 | 26
  Week 40 | 10.00 (142.168) | -12.94 (148.586) | 330.78 (447.039)
  Week 44: number analyzed (Participants) | 10 | 3 | 17
  Week 44 | -59.74 (34.119) | 127.56 (322.953) | 444.00 (505.329)
  Week 48: number analyzed (Participants) | 38 | 39 | 22
  Week 48 | -22.23 (87.761) | -30.01 (72.497) | 390.33 (502.931)
  Week 52: number analyzed (Participants) | 42 | 38 | 23
  Week 52 | -39.27 (72.619) | -49.81 (56.391) | 250.13 (497.782)

16. Secondary Outcome: Percent Change From Baseline in EASI Scores at Weeks 0, 4, 8 and 12: First Flare Treatment Period
Description: EASI assessed severity of AD, based on severity of lesion clinical signs (erythema [E], induration/papulation [I], excoriation [Ex], lichenification [L]) and % body surface area (BSA) affected. Each of clinical signs scored separately for each of 4 body regions (head and neck [h], upper limbs [u], trunk [t] [including axillae and groin], lower limbs [l] [including buttocks]) on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score (A) according to % BSA with AD: 0 (0%), 1(>0 to <10%), 2(10 to <30%), 3(30 to <50%), 4(50 to <70%), 5(70 to <90%), 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh + Ih + Exh + Lh) + 0.2*Au*(Eu + Iu + ExU + Lu) + 0.3*At*(Et +It + Ext + Lt) + 0.4*Al*(El + Il + Exl + Ll). Total EASI score ranged from 0.0 to 72.0, higher score = greater severity of AD.
Time Frame: Baseline (last observation up to and including the randomization day of DB period),Weeks 0, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 73 | 57
Percent change
  Week 0 | 484.69 (672.923) | 324.54 (484.380)
  Week 4: number analyzed (Participants) | 48 | 35
  Week 4 | 294.83 (350.182) | 293.63 (461.044)
  Week 8: number analyzed (Participants) | 32 | 22
  Week 8 | 245.70 (411.541) | 275.66 (447.181)
  Week 12: number analyzed (Participants) | 9 | 11
  Week 12 | 196.69 (272.911) | 408.94 (665.204)

17. Secondary Outcome: Percent Change From Baseline in EASI Scores at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52: First Flare Free Period
Description: as for outcome 14
Time Frame: Baseline (last observation up to and including the randomization day of DB period), Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: Eval-DB population included all randomized participants with success in ISGA and EASI50 criteria as responders at randomization and received at least 1 dose of study intervention in the DB period. Here, ''Number Analyzed'' signifies participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 129 | 125
Percent change
  Week 4: number analyzed (Participants) | 35 | 56
  Week 4 | -0.46 (67.355) | -10.34 (61.699)
  Week 8: number analyzed (Participants) | 26 | 48
  Week 8 | -21.34 (59.257) | 10.36 (144.770)
  Week 12: number analyzed (Participants) | 24 | 42
  Week 12 | 2.24 (143.094) | -9.44 (100.314)
  Week 16: number analyzed (Participants) | 19 | 37
  Week 16 | -14.82 (50.412) | -0.47 (109.386)
  Week 20: number analyzed (Participants) | 1 | 4
  Week 20 | 200.00 (NA) — Standard deviation could not be estimated as a single participant was analyzed. | -74.29 (40.808)
  Week 24: number analyzed (Participants) | 16 | 32
  Week 24 | -35.57 (55.674) | -10.82 (109.364)
  Week 28: number analyzed (Participants) | 1 | 2
  Week 28 | 0.00 (NA) — Standard deviation could not be estimated as a single participant was analyzed. | -34.52 (48.824)
  Week 32: number analyzed (Participants) | 15 | 26
  Week 32 | -28.39 (62.657) | -27.82 (94.806)
  Week 36: number analyzed (Participants) | 1 | 0
  Week 36 | -67.86 (NA) — Standard deviation could not be estimated as a single participant was analyzed. |
  Week 40: number analyzed (Participants) | 14 | 22
  Week 40 | 2.19 (83.621) | -47.60 (64.625)
  Week 44: number analyzed (Participants) | 1 | 0
  Week 44 | -36.84 (NA) — Standard deviation could not be estimated as a single participant was analyzed. |
  Week 48: number analyzed (Participants) | 14 | 20
  Week 48 | -27.27 (61.689) | -39.13 (82.669)
  Week 52: number analyzed (Participants) | 12 | 18
  Week 52 | -54.33 (45.072) | -59.87 (58.964)

18. Secondary Outcome: Change From Baseline in ISGA Scores at Weeks 2, 4, 6 and 8 for OL run-in Period
Description: ISGA is a 5- point global assessment scale, used to characterize overall disease severity across all treatable AD lesions (excluding the scalp). Score ranged from 0 to 4: where 0= clear(minor residual hypo/hyperpigmentation; no erythema or induration/papulation; no oozing/crusting), 1= almost clear (trace faint pink erythema, with barely perceptible induration/papulation and no oozing/crusting), 2= mild (faint pink erythema with mild induration/papulation and no oozing/crusting), 3= moderate (pink-red erythema with moderate induration/papulation with or without oozing/crusting), 4= severe (deep or bright red erythema with severe induration/papulation and with oozing/crusting). Higher scores indicate greater severity of AD.
Time Frame: Baseline (last observation up to and including Day 1 of OL period), Weeks 2, 4, 6 and 8
Population: Eval-OL population included all participants that received at least 1 dose of study intervention in the OL period.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crisaborole 2% BID
Number analyzed (Participants) | 497
Units on a scale
  Baseline | 2.7 (0.48)
  Change at Week 2 | -0.5 (0.69)
  Change at Week 4 | -0.7 (0.84)
  Change at Week 6 | -0.9 (0.93)
  Change at Week 8 | -1.2 (1.04)

19. Secondary Outcome: Change From Baseline in ISGA Scores at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52 for DB Period
Description: as for outcome 18
Time Frame: as for outcome 15
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD | Crisaborole 2% BID: Flare Period
Number analyzed (Participants) | 129 | 125 | 175
Units on a scale
  Baseline: number analyzed (Participants) | 129 | 125 | 0
  Baseline | 0.6 (0.50) | 0.6 (0.49) |
  Change at Week 4: number analyzed (Participants) | 60 | 81 | 105
  Change at Week 4 | 0.2 (0.52) | 0.1 (0.49) | 1.7 (0.53)
  Change at Week 8: number analyzed (Participants) | 71 | 80 | 84
  Change at Week 8 | 0.2 (0.50) | 0.1 (0.58) | 1.5 (0.55)
  Change at Week 12: number analyzed (Participants) | 65 | 76 | 73
  Change at Week 12 | 0.1 (0.52) | 0.0 (0.54) | 1.5 (0.58)
  Change at Week 16: number analyzed (Participants) | 75 | 83 | 50
  Change at Week 16 | 0.2 (0.46) | -0.0 (0.53) | 1.6 (0.60)
  Change at Week 20: number analyzed (Participants) | 13 | 13 | 32
  Change at Week 20 | 0.3 (0.75) | 0.2 (0.69) | 1.8 (0.68)
  Change at Week 24: number analyzed (Participants) | 70 | 78 | 35
  Change at Week 24 | 0.0 (0.67) | -0.1 (0.56) | 1.5 (0.61)
  Change at Week 28: number analyzed (Participants) | 12 | 6 | 26
  Change at Week 28 | 0.3 (0.45) | 0.2 (0.41) | 1.6 (0.64)
  Change at Week 32: number analyzed (Participants) | 62 | 72 | 36
  Change at Week 32 | -0.0 (0.60) | -0.1 (0.53) | 1.7 (0.53)
  Change at Week 36: number analyzed (Participants) | 8 | 5 | 23
  Change at Week 36 | 0.4 (0.74) | 0.0 (0.00) | 1.5 (0.51)
  Change at Week 40: number analyzed (Participants) | 59 | 64 | 32
  Change at Week 40 | 0.0 (0.57) | 0.0 (0.59) | 1.6 (0.67)
  Change at Week 44: number analyzed (Participants) | 13 | 8 | 21
  Change at Week 44 | -0.1 (0.64) | 0.3 (0.71) | 1.8 (0.68)
  Change at Week 48: number analyzed (Participants) | 58 | 64 | 28
  Change at Week 48 | 0.1 (0.65) | -0.0 (0.63) | 1.6 (0.68)
  Change at Week 52: number analyzed (Participants) | 63 | 63 | 28
  Change at Week 52 | 0.0 (0.66) | -0.0 (0.57) | 1.6 (0.57)

20. Secondary Outcome: Change From Baseline in ISGA Scores at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52 for First Flare Free Period
Description: as for outcome 18
Time Frame: as for outcome 15
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 129 | 125
Units on a scale
  Baseline | 0.6 (0.50) | 0.6 (0.49)
  Change at Week 4: number analyzed (Participants) | 55 | 80
  Change at Week 4 | 0.2 (0.54) | 0.1 (0.49)
  Change at Week 8: number analyzed (Participants) | 43 | 67
  Change at Week 8 | 0.2 (0.50) | 0.1 (0.60)
  Change at Week 12: number analyzed (Participants) | 37 | 59
  Change at Week 12 | 0.1 (0.55) | -0.1 (0.54)
  Change at Week 16: number analyzed (Participants) | 31 | 52
  Change at Week 16 | 0.2 (0.43) | 0.0 (0.52)
  Change at Week 20: number analyzed (Participants) | 1 | 5
  Change at Week 20 | 0.0 (NA) — Standard deviation could not be estimated as a single participant was analyzed. | -0.4 (0.55)
  Change at Week 24: number analyzed (Participants) | 26 | 46
  Change at Week 24 | 0.0 (0.63) | -0.1 (0.55)
  Change at Week 28: number analyzed (Participants) | 2 | 2
  Change at Week 28 | 0.5 (0.71) | 0.0 (0.00)
  Change at Week 32: number analyzed (Participants) | 25 | 39
  Change at Week 32 | -0.1 (0.64) | -0.1 (0.53)
  Change at Week 36: number analyzed (Participants) | 1 | 1
  Change at Week 36 | 0.0 (NA) — Standard deviation could not be estimated as a single participant was analyzed. | 0.0 (NA) — Standard deviation could not be estimated as a single participant was analyzed.
  Change at Week 40: number analyzed (Participants) | 23 | 33
  Change at Week 40 | 0.0 (0.60) | -0.1 (0.66)
  Change at Week 44: number analyzed (Participants) | 2 | 3
  Change at Week 44 | 0.0 (0.00) | 0.7 (0.58)
  Change at Week 48: number analyzed (Participants) | 24 | 32
  Change at Week 48 | 0.0 (0.66) | -0.1 (0.64)
  Change at Week 52: number analyzed (Participants) | 22 | 30
  Change at Week 52 | 0.0 (0.62) | -0.0 (0.61)

21. Secondary Outcome: Change From Baseline in ISGA Scores at Weeks 0, 4, 8 and 12 for First Flare Treatment Period
Description: ISGA:5-point global assessment scale, used to characterize overall disease severity across all treatable AD lesions (excluding scalp). Score ranged:0 to 4,where 0=clear(minor residual hypo/hyperpigmentation; no erythema or induration/papulation; no oozing/crusting), 1=almost clear(trace faint pink erythema, with barely perceptible induration/papulation and no oozing/crusting), 2=mild(faint pink erythema with mild induration/papulation and no oozing/crusting), 3=moderate(pink-red erythema with moderate induration/papulation with or without oozing/crusting), 4=severe(deep or bright red erythema with severe induration/papulation and with oozing/crusting). Higher scores indicate greater severity of AD. The period for which OL crisaborole 2% ointment BID was initiated for treatment of flare developed during DB maintenance until resumption of DB treatment was defined as flare treatment period.
Time Frame: Baseline (last observation up to and including the randomization day), Weeks 0, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 96 | 81
Units on a scale
  Change at Week 0 | 1.8 (0.57) | 1.7 (0.49)
  Change at Week 4: number analyzed (Participants) | 53 | 47
  Change at Week 4 | 1.5 (0.54) | 1.5 (0.55)
  Change at Week 8: number analyzed (Participants) | 33 | 27
  Change at Week 8 | 1.3 (0.47) | 1.6 (0.74)
  Change at Week 12: number analyzed (Participants) | 10 | 11
  Change at Week 12 | 1.5 (0.53) | 1.6 (0.67)

22. Secondary Outcome: Change From Baseline in Treatable Percent Body Surface Area (% BSA): OL Run-in Period
Description: The extent (%) to which a body region was involved with AD was determined using handprint method. Four body regions evaluated: head and neck (hn), upper limbs (ul), trunk (tr) (including axillae) and lower limbs (ll) (including buttocks). Total number of handprints=10 for hn, 20 for ul, 30 for tr, 40 for ll in participants aged >=8 years; 20 for hn, 20 for ul, 30 for tr, 30 for ll in participants aged 3 months to 7 years. Surface area of body region equivalent to 1 handprint: 10% for hn, 5% for ul, 3.33% for tr, 2.5% for ll in participants aged >=8 years; 5% for hn, 5% for ul, 3.33% for tr, 3.33% for ll in participants aged 3 months to 7 years. % BSA for a body region= total number of handprints in a body region * % surface area equivalent to 1 handprint. Overall % BSA for an individual=sum of % BSA across all 4 body regions and ranged from 0 to 100%, with higher values representing greater extent of BSA involvement with AD.
Time Frame: Baseline (last observation up to and including the randomization day) Weeks 2, 4, 6 and 8
Population: Eval-OL population included all participants that received at least 1 dose of study intervention in the OL period.
Measure: Mean (Standard Deviation); unit: Percentage BSA
Arm/Group | Crisaborole 2% BID
Number analyzed (Participants) | 497
Percentage BSA
  Baseline | 19.61 (16.807) [lower limit 16.807]
  Change at Week 2 | -3.86 (8.313) [lower limit 8.313]
  Change at Week 4 | -5.09 (10.061) [lower limit 10.061]
  Change at Week 6 | -6.42 (11.398) [lower limit 11.398]
  Change at Week 8 | -7.35 (12.301) [lower limit 12.301]

23. Secondary Outcome: Change From Baseline in Treatable %BSA: DB Period
Description: as for outcome 22
Time Frame: as for outcome 15
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Percentage BSA
Arm/Group | Vehicle QD | Crisaborole 2% QD | Crisaborole 2% BID: Flare Period
Number analyzed (Participants) | 129 | 125 | 175
Percentage BSA
  Baseline: number analyzed (Participants) | 129 | 125 | 0
  Baseline | 5.25 (9.588) | 5.22 (7.170) |
  Change at Week 4: number analyzed (Participants) | 60 | 81 | 175
  Change at Week 4 | 1.16 (4.391) | 0.52 (5.164) | 6.25 (8.208)
  Change at Week 8: number analyzed (Participants) | 71 | 80 | 84
  Change at Week 8 | 0.59 (6.202) | -0.19 (6.659) | 4.65 (8.568)
  Change at Week 12: number analyzed (Participants) | 65 | 76 | 72
  Change at Week 12 | 1.20 (6.821) | 0.26 (6.093) | 6.17 (9.801)
  Change at Week 16: number analyzed (Participants) | 75 | 83 | 50
  Change at Week 16 | 1.25 (5.623) | 0.58 (5.848) | 5.33 (9.369)
  Change at Week 20: number analyzed (Participants) | 13 | 12 | 32
  Change at Week 20 | -1.29 (5.363) | 1.38 (6.846) | 7.45 (13.678)
  Change at Week 24: number analyzed (Participants) | 70 | 78 | 35
  Change at Week 24 | 2.42 (9.213) | 2.15 (11.217) | 4.79 (7.483)
  Change at Week 28: number analyzed (Participants) | 12 | 6 | 26
  Change at Week 28 | -0.30 (6.323) | -1.25 (5.906) | 7.22 (9.389)
  Change at Week 32: number analyzed (Participants) | 62 | 72 | 36
  Change at Week 32 | 0.33 (7.623) | 0.84 (5.971) | 6.36 (11.286)
  Change at Week 36: number analyzed (Participants) | 8 | 5 | 24
  Change at Week 36 | 0.44 (1.917) | 2.50 (3.623) | 3.36 (6.603)
  Change at Week 40: number analyzed (Participants) | 59 | 64 | 32
  Change at Week 40 | 0.02 (6.752) | 0.89 (6.097) | 3.50 (8.292)
  Change at Week 44: number analyzed (Participants) | 13 | 7 | 21
  Change at Week 44 | -2.56 (4.889) | 0.57 (2.524) | 5.71 (7.559)
  Change at Week 48: number analyzed (Participants) | 58 | 64 | 28
  Change at Week 48 | -0.37 (7.134) | 0.48 (6.295) | 4.05 (8.689)
  Change at Week 52: number analyzed (Participants) | 63 | 63 | 28
  Change at Week 52 | -1.23 (5.531) | -1.91 (5.411) | 4.20 (8.835)

24. Secondary Outcome: Change From Baseline in Treatable %BSA: First Flare Free Period
Description: as for outcome 22
Time Frame: as for outcome 15
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Percentage BSA
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 129 | 125
Percentage BSA
  Baseline | 5.25 (9.588) | 5.22 (7.170)
  Change at Week 4: number analyzed (Participants) | 55 | 80
  Change at Week 4 | 1.20 (4.487) | 0.53 (5.196)
  Change at Week 8: number analyzed (Participants) | 43 | 67
  Change at Week 8 | 0.21 (7.661) | -0.10 (6.954)
  Change at Week 12: number analyzed (Participants) | 37 | 59
  Change at Week 12 | 0.96 (6.161) | 0.05 (6.309)
  Change at Week 16: number analyzed (Participants) | 31 | 52
  Change at Week 16 | 1.05 (5.929) | 0.28 (5.891)
  Change at Week 20: number analyzed (Participants) | 1 | 5
  Change at Week 20 | 5.00 (NA) — Standard deviation could not be estimated as a single participant was analyzed. | -0.60 (9.659)
  Change at Week 24: number analyzed (Participants) | 26 | 46
  Change at Week 24 | 2.46 (8.669) | 3.09 (13.575)
  Change at Week 28: number analyzed (Participants) | 2 | 2
  Change at Week 28 | -1.50 (2.121) | -3.00 (12.728)
  Change at Week 32: number analyzed (Participants) | 25 | 39
  Change at Week 32 | 0.40 (8.581) | 0.91 (5.669)
  Change at Week 36: number analyzed (Participants) | 1 | 1
  Change at Week 36 | -2.00 (NA) — Standard deviation could not be estimated as a single participant was analyzed. | 0.00 (NA) — Standard deviation could not be estimated as a single participant was analyzed.
  Change at Week 40: number analyzed (Participants) | 23 | 33
  Change at Week 40 | -0.46 (7.881) | 1.17 (6.153)
  Change at Week 44: number analyzed (Participants) | 2 | 3
  Change at Week 44 | -3.25 (4.596) | 2.33 (3.215)
  Change at Week 48: number analyzed (Participants) | 24 | 32
  Change at Week 48 | -0.85 (7.724) | 1.14 (6.959)
  Change at Week 52: number analyzed (Participants) | 22 | 30
  Change at Week 52 | -1.50 (7.365) | -1.47 (5.232)

25. Secondary Outcome: Change From Baseline in Treatable %BSA: First Flare Period
Description: as for outcome 22
Time Frame: Baseline (last observation up to and including the randomization day), Weeks 0, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percentage BSA
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 96 | 81
Percentage BSA
  Change at Week 0 | 8.27 (12.154) | 4.68 (6.304)
  Change at Week 4: number analyzed (Participants) | 54 | 47
  Change at Week 4 | 6.92 (9.704) | 4.17 (6.884)
  Change at Week 8: number analyzed (Participants) | 33 | 27
  Change at Week 8 | 4.95 (11.642) | 3.56 (6.646)
  Change at Week 12: number analyzed (Participants) | 10 | 11
  Change at Week 12 | 5.75 (10.499) | 3.39 (5.328)

26. Secondary Outcome: Change From Baseline in Most Commonly Affected Atopic Dermatitis (AD) % BSA: DB Period
Description: The investigators were required to draw the skin areas affected by AD for each participant in a body map and the most commonly affected BSA was documented.
Time Frame: Baseline (last observation up to and including the randomization day), Weeks 24 and 52
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percentage BSA affected
Arm/Group | Vehicle QD | Crisaborole 2% QD | Crisaborole 2% BID: Flare Period
Number analyzed (Participants) | 129 | 125 | 68
Percentage BSA affected
  Baseline: number analyzed (Participants) | 129 | 125 | 0
  Baseline | 14.28 (13.957) | 10.77 (9.834) |
  Change at Week 24: number analyzed (Participants) | 72 | 76 | 4
  Change at Week 24 | 2.29 (11.579) | -0.20 (3.919) | 1.75 (3.304)
  Change at Week 52: number analyzed (Participants) | 73 | 75 | 68
  Change at Week 52 | -3.46 (10.536) | -4.95 (7.731) | 0.71 (16.649)

27. Secondary Outcome: Night Time Itch Score for Participants >=12 Years of Age: OL Run-in Period
Description: The severity and frequency of itch (pruritus) during the night due to AD was assessed using a horizontal scale. Participants 12 years of age or older were asked to assess their worst itching and frequency of itching due to AD during their most recent night's sleep on a scale of 0 to 10, where 0= no itch and 10= worst itch imaginable. Higher scores indicated worse itch. Scale range of Frequency of night time itch was 0 to 10, where 0=no and 10=the most frequency imaginable. Higher score indicated higher frequency.
Time Frame: Baseline (last observation up to and including Day 1 of OL period), Weeks 2, 4, 6 and 8
Population: Eval-OL population included all participants that received at least 1 dose of study intervention in the OL period. Here, ''Overall Number of Participants Analyzed'' signifies number of participants evaluable for this outcome measure and ''Number Analyzed'' signifies participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crisaborole 2% BID
Number analyzed (Participants) | 275
Units on a scale
  Severity of night time itch: Baseline: number analyzed (Participants) | 248
  Severity of night time itch: Baseline | 4.6 (3.02)
  Severity of night time itch: Week 2: number analyzed (Participants) | 264
  Severity of night time itch: Week 2 | 2.9 (2.21)
  Severity of night time itch: Week 4: number analyzed (Participants) | 266
  Severity of night time itch: Week 4 | 2.7 (2.25)
  Severity of night time itch: Week 6: number analyzed (Participants) | 266
  Severity of night time itch: Week 6 | 2.5 (2.16)
  Severity of night time itch: Week 8: number analyzed (Participants) | 266
  Severity of night time itch: Week 8 | 2.5 (2.19)
  Frequency of night time itch: Baseline: number analyzed (Participants) | 248
  Frequency of night time itch: Baseline | 4.4 (2.80)
  Frequency of night time itch: Week 2: number analyzed (Participants) | 264
  Frequency of night time itch: Week 2 | 2.8 (2.20)
  Frequency of night time itch: Week 4: number analyzed (Participants) | 266
  Frequency of night time itch: Week 4 | 2.7 (2.23)
  Frequency of night time itch: Week 6: number analyzed (Participants) | 266
  Frequency of night time itch: Week 6 | 2.4 (2.15)
  Frequency of night time itch: Week 8: number analyzed (Participants) | 266
  Frequency of night time itch: Week 8 | 2.4 (2.16)

28. Secondary Outcome: Night Time Itch Score for Participants >=12 Years of Age: DB Period
Description: as for outcome 27
Time Frame: as for outcome 15
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD | Crisaborole 2% BID: Flare Period
Number analyzed (Participants) | 68 | 76 | 77
Units on a scale
  Severity of night time itch: Baseline: number analyzed (Participants) | 68 | 76 | 0
  Severity of night time itch: Baseline | 1.9 (1.71) | 1.8 (1.79) |
  Severity of night time itch: Week 4: number analyzed (Participants) | 40 | 58 | 39
  Severity of night time itch: Week 4 | 2.0 (1.83) | 1.2 (1.49) | 2.2 (1.87)
  Severity of night time itch: Week 8: number analyzed (Participants) | 34 | 52 | 77
  Severity of night time itch: Week 8 | 1.6 (1.61) | 1.1 (1.59) | 2.0 (2.08)
  Severity of night time itch: Week 12: number analyzed (Participants) | 32 | 52 | 36
  Severity of night time itch: Week 12 | 1.6 (1.74) | 1.1 (1.64) | 2.2 (2.18)
  Severity of night time itch: Week 16: number analyzed (Participants) | 44 | 51 | 22
  Severity of night time itch: Week 16 | 1.7 (1.85) | 1.2 (1.70) | 1.9 (1.77)
  Severity of night time itch: Week 20: number analyzed (Participants) | 44 | 49 | 15
  Severity of night time itch: Week 20 | 1.6 (1.86) | 1.3 (1.86) | 2.2 (1.57)
  Severity of night time itch: Week 24: number analyzed (Participants) | 39 | 48 | 16
  Severity of night time itch: Week 24 | 1.6 (1.71) | 1.2 (1.79) | 1.7 (1.72)
  Severity of night time itch: Week 28: number analyzed (Participants) | 41 | 48 | 13
  Severity of night time itch: Week 28 | 1.6 (1.69) | 1.2 (1.73) | 1.9 (1.84)
  Severity of night time itch: Week 32: number analyzed (Participants) | 37 | 46 | 13
  Severity of night time itch: Week 32 | 1.4 (1.57) | 1.1 (1.74) | 2.2 (2.02)
  Severity of night time itch: Week 36: number analyzed (Participants) | 35 | 46 | 12
  Severity of night time itch: Week 36 | 1.4 (1.56) | 1.1 (1.85) | 1.8 (1.94)
  Severity of night time itch: Week 40: number analyzed (Participants) | 36 | 45 | 9
  Severity of night time itch: Week 40 | 1.4 (1.46) | 1.2 (1.95) | 2.2 (1.68)
  Severity of night time itch: Week 44: number analyzed (Participants) | 30 | 45 | 10
  Severity of night time itch: Week 44 | 1.6 (1.69) | 1.2 (1.98) | 1.6 (1.52)
  Severity of night time itch: Week 48: number analyzed (Participants) | 29 | 43 | 12
  Severity of night time itch: Week 48 | 1.6 (1.76) | 1.1 (1.93) | 1.7 (1.72)
  Severity of night time itch: Week 52: number analyzed (Participants) | 32 | 40 | 8
  Severity of night time itch: Week 52 | 1.4 (1.69) | 1.2 (1.96) | 1.3 (1.12)
  Frequency of night time itch: Baseline: number analyzed (Participants) | 68 | 76 | 0
  Frequency of night time itch: Baseline | 1.9 (1.66) | 1.8 (1.79) |
  Frequency of night time itch: Week 4: number analyzed (Participants) | 40 | 58 | 39
  Frequency of night time itch: Week 4 | 1.9 (1.89) | 1.1 (1.43) | 2.2 (1.83)
  Frequency of night time itch: Week 8: number analyzed (Participants) | 34 | 52 | 77
  Frequency of night time itch: Week 8 | 1.6 (1.71) | 1.1 (1.55) | 2.0 (2.10)
  Frequency of night time itch: Week 12: number analyzed (Participants) | 32 | 52 | 36
  Frequency of night time itch: Week 12 | 1.5 (1.76) | 1.1 (1.64) | 2.1 (2.25)
  Frequency of night time itch: Week 16: number analyzed (Participants) | 44 | 51 | 22
  Frequency of night time itch: Week 16 | 1.6 (1.87) | 1.2 (1.64) | 1.8 (1.97)
  Frequency of night time itch: Week 20: number analyzed (Participants) | 44 | 49 | 15
  Frequency of night time itch: Week 20 | 1.6 (1.82) | 1.3 (1.82) | 2.0 (1.54)
  Frequency of night time itch: Week 24: number analyzed (Participants) | 39 | 48 | 16
  Frequency of night time itch: Week 24 | 1.5 (1.71) | 1.2 (1.77) | 1.7 (1.69)
  Frequency of night time itch: Week 28: number analyzed (Participants) | 41 | 48 | 13
  Frequency of night time itch: Week 28 | 1.5 (1.71) | 1.2 (1.70) | 1.7 (1.81)
  Frequency of night time itch: Week 32: number analyzed (Participants) | 37 | 46 | 13
  Frequency of night time itch: Week 32 | 1.3 (1.56) | 1.0 (1.72) | 2.1 (1.84)
  Frequency of night time itch: Week 36: number analyzed (Participants) | 35 | 46 | 12
  Frequency of night time itch: Week 36 | 1.3 (1.57) | 1.1 (1.82) | 1.8 (1.87)
  Frequency of night time itch: Week 40: number analyzed (Participants) | 36 | 45 | 9
  Frequency of night time itch: Week 40 | 1.4 (1.53) | 1.2 (1.91) | 2.1 (1.81)
  Frequency of night time itch: Week 44: number analyzed (Participants) | 30 | 45 | 10
  Frequency of night time itch: Week 44 | 1.5 (1.71) | 1.2 (1.95) | 1.5 (1.63)
  Frequency of night time itch: Week 48: number analyzed (Participants) | 29 | 43 | 12
  Frequency of night time itch: Week 48 | 1.6 (1.78) | 1.1 (1.87) | 1.5 (1.66)
  Frequency of night time itch: Week 52: number analyzed (Participants) | 32 | 40 | 8
  Frequency of night time itch: Week 52 | 1.3 (1.70) | 1.2 (1.98) | 1.3 (1.21)

29. Secondary Outcome: Night Time Itch Score for Participants >=12 Years of Age: First Flare Period
Description: as for outcome 27
Time Frame: Weeks 0, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 41 | 39
Units on a scale
  Severity of night time itch: Week 0: number analyzed (Participants) | 15 | 17
  Severity of night time itch: Week 0 | 2.0 (1.12) | 2.0 (2.32)
  Severity of night time itch: Week 4 | 2.0 (1.95) | 2.2 (2.18)
  Severity of night time itch: Week 8: number analyzed (Participants) | 19 | 15
  Severity of night time itch: Week 8 | 2.2 (1.73) | 2.8 (2.60)
  Severity of night time itch: Week 12: number analyzed (Participants) | 9 | 16
  Severity of night time itch: Week 12 | 1.8 (1.32) | 2.8 (2.03)
  Frequency of night time itch: Week 0: number analyzed (Participants) | 15 | 17
  Frequency of night time itch: Week 0 | 2.0 (1.13) | 2.0 (2.32)
  Frequency of night time itch: Week 4 | 2.0 (2.13) | 2.1 (2.11)
  Frequency of night time itch: Week 8: number analyzed (Participants) | 19 | 15
  Frequency of night time itch: Week 8 | 2.1 (1.96) | 2.6 (2.54)
  Frequency of night time itch: Week 12: number analyzed (Participants) | 9 | 16
  Frequency of night time itch: Week 12 | 1.3 (1.26) | 2.7 (2.09)

30. Secondary Outcome: Night Time Itch Score for Participants >=12 Years of Age: First Flare Free Period
Description: as for outcome 27
Time Frame: as for outcome 15
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 68 | 76
Units on a scale
  Severity of night time itch: Baseline | 1.9 (1.71) | 1.8 (1.79)
  Severity of night time itch: Week 4: number analyzed (Participants) | 38 | 55
  Severity of night time itch: Week 4 | 2.0 (1.87) | 1.2 (1.49)
  Severity of night time itch: Week 8: number analyzed (Participants) | 27 | 46
  Severity of night time itch: Week 8 | 1.8 (1.68) | 1.2 (1.64)
  Severity of night time itch: Week 12: number analyzed (Participants) | 22 | 41
  Severity of night time itch: Week 12 | 1.5 (1.27) | 1.1 (1.72)
  Severity of night time itch: Week 16: number analyzed (Participants) | 19 | 38
  Severity of night time itch: Week 16 | 1.7 (1.30) | 1.2 (1.84)
  Severity of night time itch: Week 20: number analyzed (Participants) | 18 | 34
  Severity of night time itch: Week 20 | 1.6 (1.26) | 1.4 (1.99)
  Severity of night time itch: Week 24: number analyzed (Participants) | 18 | 33
  Severity of night time itch: Week 24 | 1.6 (1.23) | 1.2 (1.92)
  Severity of night time itch: Week 28: number analyzed (Participants) | 17 | 29
  Severity of night time itch: Week 28 | 1.6 (1.21) | 1.2 (1.86)
  Severity of night time itch: Week 32: number analyzed (Participants) | 17 | 27
  Severity of night time itch: Week 32 | 1.5 (1.27) | 1.2 (1.99)
  Severity of night time itch: Week 36: number analyzed (Participants) | 17 | 28
  Severity of night time itch: Week 36 | 1.5 (1.24) | 1.1 (2.02)
  Severity of night time itch: Week 40: number analyzed (Participants) | 17 | 25
  Severity of night time itch: Week 40 | 1.6 (1.24) | 1.1 (2.08)
  Severity of night time itch: Week 44: number analyzed (Participants) | 16 | 24
  Severity of night time itch: Week 44 | 1.9 (1.20) | 1.1 (2.26)
  Severity of night time itch: Week 48: number analyzed (Participants) | 16 | 24
  Severity of night time itch: Week 48 | 1.5 (1.27) | 1.2 (2.24)
  Severity of night time itch: Week 52: number analyzed (Participants) | 12 | 20
  Severity of night time itch: Week 52 | 1.6 (1.35) | 1.2 (2.29)
  Frequency of night time itch: Baseline | 1.9 (1.66) | 1.8 (1.79)
  Frequency of night time itch: Week 4: number analyzed (Participants) | 38 | 55
  Frequency of night time itch: Week 4 | 1.9 (1.93) | 1.1 (1.43)
  Frequency of night time itch: Week 8: number analyzed (Participants) | 27 | 46
  Frequency of night time itch: Week 8 | 1.8 (1.80) | 1.1 (1.60)
  Frequency of night time itch: Week 12: number analyzed (Participants) | 22 | 41
  Frequency of night time itch: Week 12 | 1.4 (1.31) | 1.1 (1.73)
  Frequency of night time itch: Week 16: number analyzed (Participants) | 19 | 38
  Frequency of night time itch: Week 16 | 1.6 (1.29) | 1.2 (1.79)
  Frequency of night time itch: Week 20: number analyzed (Participants) | 18 | 34
  Frequency of night time itch: Week 20 | 1.5 (1.16) | 1.3 (1.92)
  Frequency of night time itch: Week 24: number analyzed (Participants) | 18 | 33
  Frequency of night time itch: Week 24 | 1.4 (1.21) | 1.2 (1.91)
  Frequency of night time itch: Week 28: number analyzed (Participants) | 17 | 29
  Frequency of night time itch: Week 28 | 1.3 (1.19) | 1.2 (1.89)
  Frequency of night time itch: Week 32: number analyzed (Participants) | 17 | 27
  Frequency of night time itch: Week 32 | 1.3 (1.24) | 1.1 (2.04)
  Frequency of night time itch: Week 36: number analyzed (Participants) | 17 | 28
  Frequency of night time itch: Week 36 | 1.3 (1.22) | 1.1 (2.05)
  Frequency of night time itch: Week 40: number analyzed (Participants) | 17 | 25
  Frequency of night time itch: Week 40 | 1.6 (1.37) | 1.1 (2.06)
  Frequency of night time itch: Week 44: number analyzed (Participants) | 16 | 24
  Frequency of night time itch: Week 44 | 1.8 (1.22) | 1.2 (2.25)
  Frequency of night time itch: Week 48: number analyzed (Participants) | 16 | 24
  Frequency of night time itch: Week 48 | 1.5 (1.32) | 1.3 (2.18)
  Frequency of night time itch: Week 52: number analyzed (Participants) | 12 | 20
  Frequency of night time itch: Week 52 | 1.3 (1.38) | 1.2 (2.30)

31. Secondary Outcome: AD Skin Pain Scores for Participants >=12 Years of Age: OL Run-in Period
Description: Participants 12 years of age or older were asked to assess their worst skin pain due to AD at the analysis time, with the question: 'AD skin pain right now' using the skin pain numerical rating scale (NRS). Skin pain NRS was a 11-point horizontal scale anchored at 0 and 10, with 0 representing "no pain" and 10 representing "worst pain imaginable." Higher scores indicated worse pain.
Time Frame: Baseline (the last observation up to and including Day 1 of OL period), Weeks 2, 4, 6 and 8
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crisaborole 2% BID
Number analyzed (Participants) | 266
Units on a scale
  Baseline: number analyzed (Participants) | 248
  Baseline | 2.6 (2.60)
  Week 2: number analyzed (Participants) | 264
  Week 2 | 2.0 (1.96)
  Week 4 | 1.9 (2.03)
  Week 6 | 1.8 (2.08)
  Week 8 | 1.7 (2.06)

32. Secondary Outcome: AD Skin Pain Scores for Participants >=12 Years of Age: DB Period
Description: as for outcome 31
Time Frame: Baseline (the last observation up to and including Day 1 of DB period), Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD | Crisaborole 2% BID: Flare Period
Number analyzed (Participants) | 68 | 76 | 77
Units on a scale
  Baseline: number analyzed (Participants) | 68 | 76 | 0
  Baseline | 1.1 (1.34) | 1.2 (1.74) |
  Week 4: number analyzed (Participants) | 40 | 58 | 39
  Week 4 | 1.1 (1.55) | 0.7 (1.27) | 1.6 (1.68)
  Week 8: number analyzed (Participants) | 34 | 52 | 44
  Week 8 | 1.0 (1.09) | 1.0 (1.59) | 1.5 (2.00)
  Week 12: number analyzed (Participants) | 32 | 52 | 36
  Week 12 | 1.1 (1.69) | 0.9 (1.62) | 1.5 (1.80)
  Week 16: number analyzed (Participants) | 44 | 51 | 22
  Week 16 | 1.3 (1.90) | 1.1 (1.67) | 1.2 (1.30)
  Week 20: number analyzed (Participants) | 44 | 49 | 15
  Week 20 | 1.0 (1.49) | 1.1 (1.81) | 1.8 (1.65)
  Week 24: number analyzed (Participants) | 39 | 48 | 16
  Week 24 | 1.1 (1.52) | 1.0 (1.82) | 1.1 (1.53)
  Week 28: number analyzed (Participants) | 41 | 48 | 13
  Week 28 | 1.0 (1.54) | 1.0 (1.78) | 1.8 (1.97)
  Week 32: number analyzed (Participants) | 37 | 46 | 13
  Week 32 | 1.0 (1.53) | 0.8 (1.71) | 1.6 (1.76)
  Week 36: number analyzed (Participants) | 35 | 46 | 12
  Week 36 | 1.1 (1.61) | 0.9 (1.78) | 1.2 (1.66)
  Week 40: number analyzed (Participants) | 36 | 45 | 9
  Week 40 | 1.1 (1.49) | 1.1 (1.95) | 1.5 (1.85)
  Week 44: number analyzed (Participants) | 30 | 45 | 10
  Week 44 | 1.1 (1.67) | 1.1 (1.99) | 1.2 (1.82)
  Week 48: number analyzed (Participants) | 29 | 43 | 12
  Week 48 | 1.3 (1.64) | 0.9 (1.88) | 1.6 (2.00)
  Week 52: number analyzed (Participants) | 32 | 40 | 8
  Week 52 | 1.0 (1.62) | 1.0 (1.99) | 1.1 (1.45)

33. Secondary Outcome: AD Skin Pain Scores for Participants >=12 Years of Age: First Flare Period
Description: as for outcome 31
Time Frame: Weeks 0, 4, 8, 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 41 | 39
Units on a scale
  Week 0: number analyzed (Participants) | 15 | 17
  Week 0 | 1.2 (1.26) | 2.2 (2.01)
  Week 4 | 1.4 (1.75) | 1.7 (1.94)
  Week 8: number analyzed (Participants) | 19 | 15
  Week 8 | 1.3 (1.53) | 2.3 (2.15)
  Week 12: number analyzed (Participants) | 9 | 16
  Week 12 | 2.0 (1.66) | 2.3 (2.05)

34. Secondary Outcome: AD Skin Pain Scores: for Participants >=12 Years of Age First Flare Free Period
Description: Participants 12 years of age or older were asked to assess their worst skin pain due to AD at the analysis time, with the question: 'AD skin pain right now' using the skin pain NRS. Skin pain NRS was a 11-point horizontal scale anchored at 0 and 10, with 0 representing "no pain" and 10 representing "worst pain imaginable." Higher scores indicated worse pain.
Time Frame: as for outcome 32
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 68 | 76
Units on a scale
  Baseline | 1.1 (1.34) | 1.2 (1.74)
  Week 4: number analyzed (Participants) | 38 | 55
  Week 4 | 1.2 (1.58) | 0.7 (1.30)
  Week 8: number analyzed (Participants) | 27 | 46
  Week 8 | 1.0 (1.16) | 1.0 (1.65)
  Week 12: number analyzed (Participants) | 22 | 41
  Week 12 | 0.9 (1.17) | 1.0 (1.75)
  Week 16: number analyzed (Participants) | 19 | 38
  Week 16 | 1.1 (1.28) | 1.1 (1.83)
  Week 20: number analyzed (Participants) | 18 | 34
  Week 20 | 1.1 (1.18) | 1.1 (2.02)
  Week 24: number analyzed (Participants) | 18 | 33
  Week 24 | 1.2 (1.36) | 1.0 (1.97)
  Week 28: number analyzed (Participants) | 17 | 29
  Week 28 | 1.0 (1.35) | 1.0 (2.04)
  Week 32: number analyzed (Participants) | 17 | 27
  Week 32 | 1.1 (1.41) | 1.0 (2.06)
  Week 36: number analyzed (Participants) | 17 | 28
  Week 36 | 1.2 (1.44) | 1.0 (2.08)
  Week 40: number analyzed (Participants) | 17 | 25
  Week 40 | 1.2 (1.43) | 1.1 (2.21)
  Week 44: number analyzed (Participants) | 16 | 24
  Week 44 | 1.2 (1.48) | 1.1 (2.37)
  Week 48: number analyzed (Participants) | 16 | 24
  Week 48 | 1.3 (1.43) | 1.0 (2.28)
  Week 52: number analyzed (Participants) | 12 | 20
  Week 52 | 1.1 (1.46) | 1.0 (2.32)

35. Secondary Outcome: Patient/Observer Global Impression of Severity Score: OL Run-in Period
Description: Patient/Observer Global Impression of Severity (PGIS/OGIS) is a single item participant or observer rated measure of the participant's AD condition severity at a given point in time using a 7-point rating scale, which ranges from 1 to 7, where 1=not present to 7=extremely severe. The PGIS was completed by all participants >=12 years of age and OGIS was completed by the observer for participants 3 months-<12 years of age.
Time Frame: Baseline (the last observation up to and including Day 1 of OL period), Weeks 2, 4, 6 and 8
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crisaborole 2% BID
Number analyzed (Participants) | 491
Units on a scale
  >= 12 years of age: Baseline: number analyzed (Participants) | 247
  >= 12 years of age: Baseline | 3.8 (1.30)
  >= 12 years of age: Week 2: number analyzed (Participants) | 268
  >= 12 years of age: Week 2 | 3.2 (1.08)
  >= 12 years of age: Week 4: number analyzed (Participants) | 269
  >= 12 years of age: Week 4 | 3.1 (1.12)
  >= 12 years of age: Week 6: number analyzed (Participants) | 269
  >= 12 years of age: Week 6 | 3.0 (1.16)
  >= 12 years of age: Week 8: number analyzed (Participants) | 269
  >= 12 years of age: Week 8 | 3.0 (1.19)
  3 months to <12 years of age: Baseline: number analyzed (Participants) | 207
  3 months to <12 years of age: Baseline | 4.4 (1.20)
  3 months to <12 years of age: Week 2: number analyzed (Participants) | 222
  3 months to <12 years of age: Week 2 | 3.3 (1.13)
  3 months to <12 years of age: Week 4: number analyzed (Participants) | 222
  3 months to <12 years of age: Week 4 | 3.3 (1.15)
  3 months to <12 years of age: Week 6: number analyzed (Participants) | 222
  3 months to <12 years of age: Week 6 | 3.2 (1.21)
  3 months to <12 years of age: Week 8: number analyzed (Participants) | 222
  3 months to <12 years of age: Week 8 | 3.1 (1.19)

36. Secondary Outcome: Patient/Observer Global Impression of Severity Score: DB Period
Description: PGIS/OGIS is a single item participant or observer rated measure of the participant's AD condition severity at a given point in time using a 7-point rating scale, which ranges from 1 to 7, where 1=not present to 7=extremely severe. The PGIS was completed by all participants >=12 years of age and OGIS was completed by the observer for participants 3 months-<12 years of age.
Time Frame: as for outcome 32
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD | Crisaborole 2% BID: Flare Period
Number analyzed (Participants) | 126 | 122 | 89
Units on a scale
  >= 12 years of age: Baseline: number analyzed (Participants) | 68 | 76 | 0
  >= 12 years of age: Baseline | 2.6 (1.03) | 2.5 (0.90) |
  >= 12 years of age: Week 4: number analyzed (Participants) | 40 | 58 | 39
  >= 12 years of age: Week 4 | 2.7 (1.14) | 2.3 (0.97) | 3.0 (0.88)
  >= 12 years of age: Week 8: number analyzed (Participants) | 34 | 52 | 44
  >= 12 years of age: Week 8 | 2.6 (0.93) | 2.2 (1.02) | 2.9 (1.10)
  >= 12 years of age: Week 12: number analyzed (Participants) | 32 | 52 | 36
  >= 12 years of age: Week 12 | 2.7 (1.05) | 2.2 (0.98) | 3.1 (1.05)
  >= 12 years of age: Week 16: number analyzed (Participants) | 44 | 51 | 22
  >= 12 years of age: Week 16 | 2.7 (1.15) | 2.3 (1.06) | 2.9 (1.21)
  >= 12 years of age: Week 20: number analyzed (Participants) | 44 | 49 | 15
  >= 12 years of age: Week 20 | 2.7 (0.98) | 2.4 (1.23) | 3.0 (1.19)
  >= 12 years of age: Week 24: number analyzed (Participants) | 39 | 48 | 16
  >= 12 years of age: Week 24 | 2.6 (1.06) | 2.4 (1.29) | 2.7 (1.16)
  >= 12 years of age: Week 28: number analyzed (Participants) | 41 | 48 | 13
  >= 12 years of age: Week 28 | 2.7 (1.04) | 2.4 (1.21) | 3.1 (1.31)
  >= 12 years of age: Week 32: number analyzed (Participants) | 37 | 46 | 13
  >= 12 years of age: Week 32 | 2.6 (1.07) | 2.4 (1.19) | 2.7 (1.30)
  >= 12 years of age: Week 36: number analyzed (Participants) | 35 | 46 | 12
  >= 12 years of age: Week 36 | 2.7 (1.15) | 2.4 (1.29) | 2.6 (1.25)
  >= 12 years of age: Week 40: number analyzed (Participants) | 36 | 45 | 9
  >= 12 years of age: Week 40 | 2.6 (1.12) | 2.4 (1.34) | 2.6 (1.00)
  >= 12 years of age: Week 44: number analyzed (Participants) | 30 | 45 | 10
  >= 12 years of age: Week 44 | 2.6 (1.18) | 2.5 (1.21) | 2.4 (0.74)
  >= 12 years of age: Week 48: number analyzed (Participants) | 29 | 43 | 12
  >= 12 years of age: Week 48 | 2.7 (1.27) | 2.4 (1.19) | 2.5 (1.10)
  >= 12 years of age: Week 52: number analyzed (Participants) | 32 | 40 | 8
  >= 12 years of age: Week 52 | 2.4 (1.19) | 2.3 (1.26) | 2.8 (0.35)
  3 months to <12 years of age: Baseline: number analyzed (Participants) | 58 | 46 | 0
  3 months to <12 years of age: Baseline | 2.6 (0.99) | 2.6 (0.83) |
  3 months to <12 years of age: Week 4: number analyzed (Participants) | 26 | 28 | 45
  3 months to <12 years of age: Week 4 | 2.6 (1.14) | 2.4 (0.93) | 3.0 (1.08)
  3 months to <12 years of age: Week 8: number analyzed (Participants) | 29 | 27 | 45
  3 months to <12 years of age: Week 8 | 2.3 (1.13) | 2.4 (1.03) | 2.8 (1.10)
  3 months to <12 years of age: Week 12: number analyzed (Participants) | 32 | 23 | 42
  3 months to <12 years of age: Week 12 | 2.3 (0.99) | 2.2 (0.73) | 2.9 (1.16)
  3 months to <12 years of age: Week 16: number analyzed (Participants) | 32 | 28 | 30
  3 months to <12 years of age: Week 16 | 2.4 (1.14) | 2.1 (0.77) | 2.8 (1.13)
  3 months to <12 years of age: Week 20: number analyzed (Participants) | 31 | 32 | 21
  3 months to <12 years of age: Week 20 | 2.4 (1.03) | 2.2 (0.88) | 2.7 (1.07)
  3 months to <12 years of age: Week 24: number analyzed (Participants) | 32 | 32 | 18
  3 months to <12 years of age: Week 24 | 2.4 (1.04) | 2.3 (1.02) | 2.7 (0.76)
  3 months to <12 years of age: Week 28: number analyzed (Participants) | 31 | 29 | 19
  3 months to <12 years of age: Week 28 | 2.4 (1.08) | 2.0 (0.66) | 2.5 (0.65)
  3 months to <12 years of age: Week 32: number analyzed (Participants) | 27 | 25 | 21
  3 months to <12 years of age: Week 32 | 2.1 (0.80) | 2.1 (0.64) | 2.7 (0.79)
  3 months to <12 years of age: Week 36: number analyzed (Participants) | 25 | 22 | 19
  3 months to <12 years of age: Week 36 | 2.4 (1.18) | 2.0 (0.58) | 2.9 (1.06)
  3 months to <12 years of age: Week 40: number analyzed (Participants) | 25 | 17 | 21
  3 months to <12 years of age: Week 40 | 2.2 (0.74) | 2.1 (0.67) | 2.8 (1.18)
  3 months to <12 years of age: Week 44: number analyzed (Participants) | 26 | 21 | 17
  3 months to <12 years of age: Week 44 | 2.3 (1.05) | 2.0 (0.64) | 3.0 (1.25)
  3 months to <12 years of age: Week 48: number analyzed (Participants) | 26 | 18 | 17
  3 months to <12 years of age: Week 48 | 2.2 (0.80) | 1.8 (0.53) | 2.8 (0.95)
  3 months to <12 years of age: Week 52: number analyzed (Participants) | 26 | 16 | 14
  3 months to <12 years of age: Week 52 | 2.1 (1.00) | 1.7 (0.62) | 2.6 (1.04)

37. Secondary Outcome: Patient/Observer Global Impression of Severity Score: First Flare Period
Description: as for outcome 36
Time Frame: Weeks 0, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 93 | 75
Units on a scale
  >= 12 years of age: Week 0: number analyzed (Participants) | 15 | 17
  >= 12 years of age: Week 0 | 2.8 (0.93) | 3.1 (1.10)
  >= 12 years of age: Week 4: number analyzed (Participants) | 41 | 39
  >= 12 years of age: Week 4 | 2.9 (0.98) | 2.9 (1.14)
  >= 12 years of age: Week 8: number analyzed (Participants) | 19 | 15
  >= 12 years of age: Week 8 | 3.1 (1.02) | 3.6 (1.17)
  >= 12 years of age: Week 12: number analyzed (Participants) | 9 | 16
  >= 12 years of age: Week 12 | 3.3 (1.56) | 3.1 (1.50)
  3 months to <12 years of age: Week 0: number analyzed (Participants) | 15 | 11
  3 months to <12 years of age: Week 0 | 2.8 (0.94) | 3.0 (0.79)
  3 months to <12 years of age: Week 4: number analyzed (Participants) | 52 | 36
  3 months to <12 years of age: Week 4 | 3.0 (1.19) | 2.8 (0.90)
  3 months to <12 years of age: Week 8: number analyzed (Participants) | 23 | 17
  3 months to <12 years of age: Week 8 | 2.9 (1.16) | 3.1 (1.03)
  3 months to <12 years of age: Week 12: number analyzed (Participants) | 9 | 6
  3 months to <12 years of age: Week 12 | 2.8 (0.95) | 3.4 (0.79)

38. Secondary Outcome: Patient/Observer Global Impression of Severity Score: First Flare Free Period
Description: as for outcome 36
Time Frame: as for outcome 32
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 126 | 122
Units on a scale
  >= 12 years of age: Baseline: number analyzed (Participants) | 68 | 76
  >= 12 years of age: Baseline | 2.6 (1.03) | 2.5 (0.90)
  >= 12 years of age: Week 4: number analyzed (Participants) | 40 | 57
  >= 12 years of age: Week 4 | 2.7 (1.14) | 2.3 (0.98)
  >= 12 years of age: Week 8: number analyzed (Participants) | 29 | 47
  >= 12 years of age: Week 8 | 2.6 (1.00) | 2.3 (1.05)
  >= 12 years of age: Week 12: number analyzed (Participants) | 22 | 42
  >= 12 years of age: Week 12 | 2.6 (1.03) | 2.2 (1.03)
  >= 12 years of age: Week 16: number analyzed (Participants) | 20 | 38
  >= 12 years of age: Week 16 | 2.6 (1.04) | 2.1 (1.00)
  >= 12 years of age: Week 20: number analyzed (Participants) | 18 | 35
  >= 12 years of age: Week 20 | 2.7 (0.96) | 2.2 (1.10)
  >= 12 years of age: Week 24: number analyzed (Participants) | 18 | 33
  >= 12 years of age: Week 24 | 2.7 (1.06) | 2.2 (1.11)
  >= 12 years of age: Week 28: number analyzed (Participants) | 17 | 30
  >= 12 years of age: Week 28 | 2.7 (1.05) | 2.2 (1.07)
  >= 12 years of age: Week 32: number analyzed (Participants) | 17 | 27
  >= 12 years of age: Week 32 | 2.6 (1.05) | 2.1 (1.02)
  >= 12 years of age: Week 36: number analyzed (Participants) | 17 | 28
  >= 12 years of age: Week 36 | 2.7 (1.05) | 2.1 (1.08)
  >= 12 years of age: Week 40: number analyzed (Participants) | 17 | 25
  >= 12 years of age: Week 40 | 2.7 (1.10) | 2.1 (1.10)
  >= 12 years of age: Week 44: number analyzed (Participants) | 16 | 24
  >= 12 years of age: Week 44 | 2.7 (1.10) | 2.3 (1.24)
  >= 12 years of age: Week 48: number analyzed (Participants) | 16 | 24
  >= 12 years of age: Week 48 | 2.6 (1.14) | 2.3 (1.28)
  >= 12 years of age: Week 52: number analyzed (Participants) | 14 | 21
  >= 12 years of age: Week 52 | 2.6 (1.15) | 2.0 (1.25)
  3 months to <12 years of age: Baseline: number analyzed (Participants) | 58 | 46
  3 months to <12 years of age: Baseline | 2.6 (0.99) | 2.6 (0.83)
  3 months to <12 years of age: Week 4: number analyzed (Participants) | 26 | 28
  3 months to <12 years of age: Week 4 | 2.6 (1.14) | 2.4 (0.93)
  3 months to <12 years of age: Week 8: number analyzed (Participants) | 19 | 22
  3 months to <12 years of age: Week 8 | 2.5 (1.28) | 2.3 (0.98)
  3 months to <12 years of age: Week 12: number analyzed (Participants) | 18 | 17
  3 months to <12 years of age: Week 12 | 2.3 (1.12) | 2.3 (0.78)
  3 months to <12 years of age: Week 16: number analyzed (Participants) | 16 | 16
  3 months to <12 years of age: Week 16 | 2.4 (1.14) | 2.0 (0.84)
  3 months to <12 years of age: Week 20: number analyzed (Participants) | 11 | 15
  3 months to <12 years of age: Week 20 | 2.3 (1.24) | 2.1 (0.83)
  3 months to <12 years of age: Week 24: number analyzed (Participants) | 10 | 14
  3 months to <12 years of age: Week 24 | 2.3 (1.47) | 1.9 (0.59)
  3 months to <12 years of age: Week 28: number analyzed (Participants) | 9 | 13
  3 months to <12 years of age: Week 28 | 2.4 (1.59) | 2.0 (0.57)
  3 months to <12 years of age: Week 32: number analyzed (Participants) | 8 | 13
  3 months to <12 years of age: Week 32 | 1.8 (0.75) | 2.1 (0.58)
  3 months to <12 years of age: Week 36: number analyzed (Participants) | 8 | 9
  3 months to <12 years of age: Week 36 | 2.6 (1.77) | 1.7 (0.56)
  3 months to <12 years of age: Week 40: number analyzed (Participants) | 8 | 7
  3 months to <12 years of age: Week 40 | 2.0 (0.99) | 1.8 (0.60)
  3 months to <12 years of age: Week 44: number analyzed (Participants) | 8 | 9
  3 months to <12 years of age: Week 44 | 2.7 (1.66) | 1.7 (0.56)
  3 months to <12 years of age: Week 48: number analyzed (Participants) | 7 | 7
  3 months to <12 years of age: Week 48 | 2.1 (0.92) | 1.7 (0.41)
  3 months to <12 years of age: Week 52: number analyzed (Participants) | 7 | 6
  3 months to <12 years of age: Week 52 | 1.5 (0.50) | 1.6 (0.65)

39. Secondary Outcome: Patient/Observer Global Impression of Change Score: OL Run-in Period
Description: Patient/Observer Global Impression of Change (PGIC/OGIC) is a single item instrument using 7-point rating scale and was used to determine global improvement at a given point in time since the start of study drug. The scores ranged from 1=very much improved to 7=very much worse. The PGIC was completed by all participants >=12 years of age and OGIC was completed by the observer for participants 3 months-<12 years of age.
Time Frame: Weeks 2, 4, 6 and 8
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crisaborole 2% BID
Number analyzed (Participants) | 495
Units on a scale
  >= 12 years of age: Week 2: number analyzed (Participants) | 271
  >= 12 years of age: Week 2 | 2.8 (1.17)
  >= 12 years of age: Week 4: number analyzed (Participants) | 273
  >= 12 years of age: Week 4 | 2.7 (1.32)
  >= 12 years of age: Week 6: number analyzed (Participants) | 273
  >= 12 years of age: Week 6 | 2.6 (1.36)
  >= 12 years of age: Week 8: number analyzed (Participants) | 273
  >= 12 years of age: Week 8 | 2.6 (1.46)
  3 months to <12 years: Week 2: number analyzed (Participants) | 222
  3 months to <12 years: Week 2 | 2.6 (1.21)
  3 months to <12 years: Week 4: number analyzed (Participants) | 222
  3 months to <12 years: Week 4 | 2.6 (1.36)
  3 months to <12 years: Week 6: number analyzed (Participants) | 222
  3 months to <12 years: Week 6 | 2.5 (1.50)
  3 months to <12 years: Week 8: number analyzed (Participants) | 222
  3 months to <12 years: Week 8 | 2.5 (1.57)

40. Secondary Outcome: Patient/Observer Global Impression of Change Score: DB Period
Description: PGIC/OGIC is a single item instrument using 7-point rating scale and was used to determine global improvement at a given point in time since the start of study drug. The scores ranged from 1=very much improved to 7=very much worse. The PGIC was completed by all participants >=12 years of age and OGIC was completed by the observer for participants 3 months-<12 years of age.
Time Frame: as for outcome 32
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD | Crisaborole 2% BID: Flare Period
Number analyzed (Participants) | 129 | 125 | 101
Units on a scale
  >= 12 years of age: Baseline: number analyzed (Participants) | 69 | 78 | 0
  >= 12 years of age: Baseline | 1.8 (0.68) | 1.8 (0.75) |
  >= 12 years of age: Week 4: number analyzed (Participants) | 32 | 51 | 51
  >= 12 years of age: Week 4 | 1.9 (0.84) | 1.8 (0.76) | 3.7 (1.53)
  >= 12 years of age: Week 8: number analyzed (Participants) | 36 | 50 | 38
  >= 12 years of age: Week 8 | 2.0 (0.74) | 1.9 (0.88) | 2.9 (1.38)
  >= 12 years of age: Week 12: number analyzed (Participants) | 32 | 49 | 32
  >= 12 years of age: Week 12 | 2.0 (0.76) | 1.9 (1.00) | 3.1 (1.41)
  >= 12 years of age: Week 16: number analyzed (Participants) | 42 | 52 | 21
  >= 12 years of age: Week 16 | 2.1 (1.00) | 1.8 (0.79) | 3.0 (1.32)
  >= 12 years of age: Week 20: number analyzed (Participants) | 21 | 21 | 11
  >= 12 years of age: Week 20 | 2.3 (1.10) | 1.6 (0.80) | 2.4 (1.03)
  >= 12 years of age: Week 24: number analyzed (Participants) | 37 | 47 | 14
  >= 12 years of age: Week 24 | 1.7 (0.70) | 1.8 (1.10) | 2.9 (1.23)
  >= 12 years of age: Week 28: number analyzed (Participants) | 18 | 17 | 14
  >= 12 years of age: Week 28 | 2.2 (1.06) | 1.6 (0.80) | 3.4 (1.34)
  >= 12 years of age: Week 32: number analyzed (Participants) | 34 | 45 | 13
  >= 12 years of age: Week 32 | 1.7 (0.72) | 1.8 (1.26) | 2.4 (1.19)
  >= 12 years of age: Week 36: number analyzed (Participants) | 17 | 17 | 7
  >= 12 years of age: Week 36 | 1.9 (0.93) | 1.8 (0.66) | 2.4 (1.13)
  >= 12 years of age: Week 40: number analyzed (Participants) | 34 | 47 | 8
  >= 12 years of age: Week 40 | 1.8 (0.91) | 1.8 (1.10) | 3.3 (1.58)
  >= 12 years of age: Week 44: number analyzed (Participants) | 18 | 17 | 11
  >= 12 years of age: Week 44 | 1.8 (0.79) | 1.8 (0.75) | 3.2 (1.33)
  >= 12 years of age: Week 48: number analyzed (Participants) | 30 | 43 | 12
  >= 12 years of age: Week 48 | 1.5 (0.63) | 1.9 (1.34) | 2.8 (1.42)
  >= 12 years of age: Week 52: number analyzed (Participants) | 32 | 43 | 15
  >= 12 years of age: Week 52 | 1.8 (0.76) | 1.6 (1.01) | 1.8 (0.86)
  3 months to <12 years of age: Baseline: number analyzed (Participants) | 60 | 47 | 0
  3 months to <12 years of age: Baseline | 1.5 (0.60) | 1.6 (0.61) |
  3 months to <12 years of age: Week 4: number analyzed (Participants) | 24 | 24 | 50
  3 months to <12 years of age: Week 4 | 1.7 (0.95) | 2.0 (1.23) | 3.4 (1.62)
  3 months to <12 years of age: Week 8: number analyzed (Participants) | 30 | 24 | 38
  3 months to <12 years of age: Week 8 | 1.5 (0.57) | 1.8 (0.98) | 2.8 (1.37)
  3 months to <12 years of age: Week 12: number analyzed (Participants) | 29 | 26 | 34
  3 months to <12 years of age: Week 12 | 1.6 (0.68) | 1.5 (0.65) | 2.8 (1.15)
  3 months to <12 years of age: Week 16: number analyzed (Participants) | 26 | 28 | 27
  3 months to <12 years of age: Week 16 | 1.8 (0.97) | 1.5 (0.58) | 2.6 (1.31)
  3 months to <12 years of age: Week 20: number analyzed (Participants) | 16 | 17 | 17
  3 months to <12 years of age: Week 20 | 1.9 (0.72) | 1.4 (0.62) | 2.4 (0.80)
  3 months to <12 years of age: Week 24: number analyzed (Participants) | 27 | 29 | 20
  3 months to <12 years of age: Week 24 | 1.7 (0.90) | 1.7 (0.77) | 2.3 (1.21)
  3 months to <12 years of age: Week 28: number analyzed (Participants) | 16 | 19 | 14
  3 months to <12 years of age: Week 28 | 1.6 (0.73) | 1.4 (0.68) | 2.1 (1.03)
  3 months to <12 years of age: Week 32: number analyzed (Participants) | 25 | 24 | 20
  3 months to <12 years of age: Week 32 | 1.9 (1.24) | 1.8 (1.09) | 2.7 (1.26)
  3 months to <12 years of age: Week 36: number analyzed (Participants) | 13 | 15 | 15
  3 months to <12 years of age: Week 36 | 1.6 (0.51) | 1.5 (0.64) | 2.7 (1.28)
  3 months to <12 years of age: Week 40: number analyzed (Participants) | 21 | 16 | 23
  3 months to <12 years of age: Week 40 | 1.9 (0.85) | 1.7 (0.87) | 2.8 (1.56)
  3 months to <12 years of age: Week 44: number analyzed (Participants) | 13 | 12 | 9
  3 months to <12 years of age: Week 44 | 1.6 (0.51) | 1.8 (1.14) | 2.4 (0.73)
  3 months to <12 years of age: Week 48: number analyzed (Participants) | 22 | 20 | 16
  3 months to <12 years of age: Week 48 | 1.6 (0.67) | 1.6 (0.89) | 2.6 (1.41)
  3 months to <12 years of age: Week 52: number analyzed (Participants) | 29 | 20 | 13
  3 months to <12 years of age: Week 52 | 1.6 (0.78) | 1.5 (0.60) | 2.3 (0.75)

41. Secondary Outcome: Patient/Observer Global Impression of Change Score: First Flare Period
Description: as for outcome 40
Time Frame: Weeks 0, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 89 | 77
Units on a scale
  >= 12 years of age: Week 0: number analyzed (Participants) | 43 | 44
  >= 12 years of age: Week 0 | 3.8 (1.56) | 3.1 (1.51)
  >= 12 years of age: Week 4: number analyzed (Participants) | 21 | 24
  >= 12 years of age: Week 4 | 2.7 (1.42) | 2.9 (1.30)
  >= 12 years of age: Week 8: number analyzed (Participants) | 13 | 15
  >= 12 years of age: Week 8 | 2.4 (0.51) | 3.2 (1.26)
  >= 12 years of age: Week 12: number analyzed (Participants) | 3 | 7
  >= 12 years of age: Week 12 | 2.7 (0.58) | 3.7 (1.11)
  3 months to <12 years of age: Week 0: number analyzed (Participants) | 46 | 33
  3 months to <12 years of age: Week 0 | 3.8 (1.84) | 3.3 (1.53)
  3 months to <12 years of age: Week 4: number analyzed (Participants) | 28 | 21
  3 months to <12 years of age: Week 4 | 2.4 (0.95) | 2.6 (0.97)
  3 months to <12 years of age: Week 8: number analyzed (Participants) | 18 | 11
  3 months to <12 years of age: Week 8 | 2.3 (0.97) | 3.0 (1.41)
  3 months to <12 years of age: Week 12: number analyzed (Participants) | 5 | 2
  3 months to <12 years of age: Week 12 | 2.4 (0.55) | 4.5 (0.71)

42. Secondary Outcome: Patient/Observer Global Impression of Change Score: First Flare Free Period
Description: as for outcome 40
Time Frame: as for outcome 32
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 129 | 125
Units on a scale
  >= 12 years of age: Baseline: number analyzed (Participants) | 69 | 78
  >= 12 years of age: Baseline | 1.8 (0.68) | 1.8 (0.75)
  >= 12 years of age: Week 4: number analyzed (Participants) | 30 | 51
  >= 12 years of age: Week 4 | 2.0 (0.83) | 1.8 (0.76)
  >= 12 years of age: Week 8: number analyzed (Participants) | 25 | 44
  >= 12 years of age: Week 8 | 2.1 (0.73) | 1.9 (0.90)
  >= 12 years of age: Week 12: number analyzed (Participants) | 20 | 40
  >= 12 years of age: Week 12 | 2.0 (0.86) | 2.0 (1.04)
  >= 12 years of age: Week 16: number analyzed (Participants) | 19 | 37
  >= 12 years of age: Week 16 | 2.3 (1.29) | 1.8 (0.76)
  >= 12 years of age: Week 20: number analyzed (Participants) | 8 | 13
  >= 12 years of age: Week 20 | 1.9 (0.64) | 1.5 (0.52)
  >= 12 years of age: Week 24: number analyzed (Participants) | 17 | 31
  >= 12 years of age: Week 24 | 1.8 (0.83) | 1.6 (0.80)
  >= 12 years of age: Week 28: number analyzed (Participants) | 7 | 9
  >= 12 years of age: Week 28 | 1.9 (0.69) | 1.4 (0.53)
  >= 12 years of age: Week 32: number analyzed (Participants) | 16 | 27
  >= 12 years of age: Week 32 | 1.7 (0.60) | 1.6 (0.97)
  >= 12 years of age: Week 36: number analyzed (Participants) | 6 | 7
  >= 12 years of age: Week 36 | 2.0 (1.26) | 1.4 (0.53)
  >= 12 years of age: Week 40: number analyzed (Participants) | 17 | 26
  >= 12 years of age: Week 40 | 1.7 (0.85) | 1.5 (0.58)
  >= 12 years of age: Week 44: number analyzed (Participants) | 7 | 9
  >= 12 years of age: Week 44 | 2.1 (1.07) | 1.6 (0.73)
  >= 12 years of age: Week 48: number analyzed (Participants) | 17 | 24
  >= 12 years of age: Week 48 | 1.5 (0.62) | 1.6 (1.10)
  >= 12 years of age: Week 52: number analyzed (Participants) | 15 | 23
  >= 12 years of age: Week 52 | 1.7 (0.88) | 1.4 (0.50)
  3 months to <12 years of age: Baseline: number analyzed (Participants) | 60 | 47
  3 months to <12 years of age: Baseline | 1.5 (0.60) | 1.6 (0.61)
  3 months to <12 years of age: Week 4: number analyzed (Participants) | 22 | 24
  3 months to <12 years of age: Week 4 | 1.8 (0.97) | 2.0 (1.23)
  3 months to <12 years of age: Week 8: number analyzed (Participants) | 15 | 18
  3 months to <12 years of age: Week 8 | 1.7 (0.62) | 1.8 (1.00)
  3 months to <12 years of age: Week 12: number analyzed (Participants) | 15 | 18
  3 months to <12 years of age: Week 12 | 1.7 (0.80) | 1.6 (0.62)
  3 months to <12 years of age: Week 16: number analyzed (Participants) | 10 | 14
  3 months to <12 years of age: Week 16 | 1.6 (0.97) | 1.6 (0.63)
  3 months to <12 years of age: Week 20: number analyzed (Participants) | 3 | 9
  3 months to <12 years of age: Week 20 | 1.7 (0.58) | 1.4 (0.73)
  3 months to <12 years of age: Week 24: number analyzed (Participants) | 7 | 14
  3 months to <12 years of age: Week 24 | 1.6 (0.53) | 1.6 (0.84)
  3 months to <12 years of age: Week 28: number analyzed (Participants) | 3 | 9
  3 months to <12 years of age: Week 28 | 1.0 (0.00) | 1.3 (0.71)
  3 months to <12 years of age: Week 32: number analyzed (Participants) | 8 | 11
  3 months to <12 years of age: Week 32 | 1.6 (0.52) | 1.7 (0.90)
  3 months to <12 years of age: Week 36: number analyzed (Participants) | 1 | 8
  3 months to <12 years of age: Week 36 | 1.0 (NA) — Standard deviation could not be estimated as a single participant was analyzed. | 1.5 (0.53)
  3 months to <12 years of age: Week 40: number analyzed (Participants) | 7 | 8
  3 months to <12 years of age: Week 40 | 1.7 (0.76) | 1.3 (0.46)
  3 months to <12 years of age: Week 44: number analyzed (Participants) | 1 | 5
  3 months to <12 years of age: Week 44 | 1.0 (NA) — Standard deviation could not be estimated as a single participant was analyzed. | 1.4 (0.55)
  3 months to <12 years of age: Week 48: number analyzed (Participants) | 6 | 7
  3 months to <12 years of age: Week 48 | 1.5 (0.55) | 1.3 (0.49)
  3 months to <12 years of age: Week 52: number analyzed (Participants) | 7 | 7
  3 months to <12 years of age: Week 52 | 1.1 (0.38) | 1.3 (0.49)

43. Secondary Outcome: Medical Outcome Study Sleep Scale Score in Participants >=12 Years of Age: OL Run-in Period
Description: The Medical Outcomes Study (MOS) Sleep Scale is a 12-item measure that is segregated into subscales addressing seven sleep domains (i.e. sleep disturbance, snoring, short of breath or headache, adequacy of sleep, somnolence, sleep problems index I and sleep problems index II) and a single item assessing quantity of sleep. Quantity of sleep scores ranged from 0 to 24 (number of hours slept) and Optimal Sleep score ranged from 0 (no) to 1(yes) based on whether the participant slept for 7-8 hours per night, All other subscales including sleep problems index 1 and 2:were scored on a range of 0 to 100 where, higher scores=greater impairment. Observed scores for each individual sleep domain and quantity of sleep are reported in this outcome measure.
Time Frame: Baseline (the last observation up to and including Day 1 of OL period), Weeks 2, 4, 6 and 8
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crisaborole 2% BID
Number analyzed (Participants) | 273
Units on a scale
  Quantity Hours Slept Score: Baseline: number analyzed (Participants) | 268
  Quantity Hours Slept Score: Baseline | 7.4 (3.27)
  Quantity Hours Slept Score: Week 2: number analyzed (Participants) | 271
  Quantity Hours Slept Score: Week 2 | 7.6 (3.06)
  Quantity Hours Slept Score: Week 4 | 7.6 (3.24)
  Quantity Hours Slept Score: Week 6 | 7.9 (3.43)
  Quantity Hours Slept Score: Week 8 | 7.8 (3.41)
  Optimal Hours Slept Score: Baseline: number analyzed (Participants) | 268
  Optimal Hours Slept Score: Baseline | 0.4 (0.50)
  Optimal Hours Slept Score: Week 2: number analyzed (Participants) | 271
  Optimal Hours Slept Score: Week 2 | 0.5 (0.50)
  Optimal Hours Slept Score: Week 4 | 0.5 (0.50)
  Optimal Hours Slept Score: Week 6 | 0.5 (0.50)
  Optimal Hours Slept Score: Week 8 | 0.5 (0.50)
  Short of Breath or Headache score: Baseline: number analyzed (Participants) | 268
  Short of Breath or Headache score: Baseline | 27.8 (15.18)
  Short of Breath or Headache score: Week 2: number analyzed (Participants) | 271
  Short of Breath or Headache score: Week 2 | 27.6 (13.98)
  Short of Breath or Headache score: Week 4 | 27.0 (14.56)
  Short of Breath or Headache score: Week 6 | 27.0 (13.95)
  Short of Breath or Headache score: Week 8 | 26.4 (14.00)
  Snoring Score: Baseline: number analyzed (Participants) | 268
  Snoring Score: Baseline | 43.3 (27.34)
  Snoring Score: Week 2: number analyzed (Participants) | 271
  Snoring Score: Week 2 | 41.1 (26.73)
  Snoring Score: Week 4 | 41.0 (26.02)
  Snoring Score: Week 6 | 40.9 (26.44)
  Snoring Score: Week 8 | 40.5 (26.09)
  Sleep Disturbance Score: Baseline: number analyzed (Participants) | 268
  Sleep Disturbance Score: Baseline | 45.0 (21.27)
  Sleep Disturbance Score: Week 2: number analyzed (Participants) | 271
  Sleep Disturbance Score: Week 2 | 40.0 (20.21)
  Sleep Disturbance Score: Week 4 | 40.3 (21.20)
  Sleep Disturbance Score: Week 6 | 38.5 (20.25)
  Sleep Disturbance Score: Week 8 | 38.6 (20.93)
  Sleep Adequacy Score: Baseline: number analyzed (Participants) | 268
  Sleep Adequacy Score: Baseline | 63.0 (19.99)
  Sleep Adequacy Score: Week 2: number analyzed (Participants) | 271
  Sleep Adequacy Score: Week 2 | 66.1 (20.64)
  Sleep Adequacy Score: Week 4 | 65.5 (20.67)
  Sleep Adequacy Score: Week 6 | 66.8 (20.12)
  Sleep Adequacy Score: Week 8 | 67.3 (20.33)
  Sleep Somnolence Score: Baseline: number analyzed (Participants) | 268
  Sleep Somnolence Score: Baseline | 44.9 (18.01)
  Sleep Somnolence Score: Week 2: number analyzed (Participants) | 271
  Sleep Somnolence Score: Week 2 | 42.5 (17.19)
  Sleep Somnolence Score: Week 4 | 42.5 (18.12)
  Sleep Somnolence Score: Week 6 | 42.5 (17.93)
  Sleep Somnolence Score: Week 8 | 42.5 (19.08)
  Sleep Problems Index I Score: Baseline: number analyzed (Participants) | 268
  Sleep Problems Index I Score: Baseline | 38.3 (14.74)
  Sleep Problems Index I Score: Week 2: number analyzed (Participants) | 271
  Sleep Problems Index I Score: Week 2 | 35.3 (13.83)
  Sleep Problems Index I Score: Week 4 | 36.1 (14.97)
  Sleep Problems Index I Score: Week 6 | 34.9 (14.08)
  Sleep Problems Index I Score: Week 8 | 34.7 (14.03)
  Sleep Problems Index II Score: Baseline: number analyzed (Participants) | 268
  Sleep Problems Index II Score: Baseline | 41.5 (15.39)
  Sleep Problems Index II Score: Week 2: number analyzed (Participants) | 271
  Sleep Problems Index II Score: Week 2 | 37.7 (14.67)
  Sleep Problems Index II Score: Week 4 | 38.1 (15.73)
  Sleep Problems Index II Score: Week 6 | 36.9 (14.82)
  Sleep Problems Index II Score: Week 8 | 36.6 (15.13)

44. Secondary Outcome: Medical Outcome Study Sleep Scale Score in Participants >=12 Years of Age: DB Period
Description: MOS Sleep Scale is a 12-item measure that is segregated into subscales addressing seven sleep domains (i.e. sleep disturbance, snoring, short of breath or headache, adequacy of sleep, somnolence, sleep problems index I and sleep problems index II) and a single item assessing quantity of sleep. Quantity of sleep scores ranged from 0 to 24 (number of hours slept) and Optimal Sleep score ranged from 0 (no) to 1(yes) based on whether the participant slept for 7-8 hours per night, All other subscales including sleep problems index 1 and 2:were scored on a range of 0 to 100 where, higher scores=greater impairment. Observed scores for each individual sleep domain and quantity of sleep are reported in this outcome measure.
Time Frame: Baseline (the last observation up to and including Day 1 of DB period),Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD | Crisaborole 2% BID: Flare Period
Number analyzed (Participants) | 69 | 78 | 88
Units on a scale
  Quantity Hours Slept Score: Baseline: number analyzed (Participants) | 69 | 78 | 0
  Quantity Hours Slept Score: Baseline | 8.3 (3.79) | 7.5 (2.42) |
  Quantity Hours Slept Score: Week 4: number analyzed (Participants) | 31 | 51 | 51
  Quantity Hours Slept Score: Week 4 | 8.9 (4.55) | 8.1 (3.32) | 6.9 (1.92)
  Quantity Hours Slept Score: Week 8: number analyzed (Participants) | 36 | 50 | 37
  Quantity Hours Slept Score: Week 8 | 8.1 (3.31) | 7.8 (3.72) | 7.9 (3.19)
  Quantity Hours Slept Score: Week 12: number analyzed (Participants) | 32 | 49 | 32
  Quantity Hours Slept Score: Week 12 | 8.8 (4.46) | 7.5 (3.18) | 7.7 (2.89)
  Quantity Hours Slept Score: Week 16: number analyzed (Participants) | 42 | 52 | 21
  Quantity Hours Slept Score: Week 16 | 8.2 (3.89) | 8.1 (4.35) | 8.4 (3.80)
  Quantity Hours Slept Score: Week 20: number analyzed (Participants) | 21 | 21 | 11
  Quantity Hours Slept Score: Week 20 | 6.9 (1.28) | 7.3 (1.49) | 8.9 (3.83)
  Quantity Hours Slept Score: Week 24: number analyzed (Participants) | 37 | 47 | 14
  Quantity Hours Slept Score: Week 24 | 8.0 (4.21) | 8.0 (4.33) | 8.3 (2.13)
  Quantity Hours Slept Score: Week 28: number analyzed (Participants) | 18 | 17 | 14
  Quantity Hours Slept Score: Week 28 | 8.4 (5.20) | 7.2 (1.38) | 7.9 (2.98)
  Quantity Hours Slept Score: Week 32: number analyzed (Participants) | 34 | 45 | 13
  Quantity Hours Slept Score: Week 32 | 9.2 (5.64) | 8.3 (3.70) | 7.8 (4.25)
  Quantity Hours Slept Score: Week 36: number analyzed (Participants) | 17 | 17 | 7
  Quantity Hours Slept Score: Week 36 | 6.9 (1.58) | 7.2 (1.48) | 7.4 (0.98)
  Quantity Hours Slept Score: Week 40: number analyzed (Participants) | 34 | 47 | 8
  Quantity Hours Slept Score: Week 40 | 8.1 (4.39) | 8.1 (3.92) | 10.0 (6.23)
  Quantity Hours Slept Score: Week 44: number analyzed (Participants) | 18 | 17 | 11
  Quantity Hours Slept Score: Week 44 | 7.1 (2.04) | 6.7 (0.99) | 8.7 (5.44)
  Quantity Hours Slept Score: Week 48: number analyzed (Participants) | 30 | 43 | 12
  Quantity Hours Slept Score: Week 48 | 7.6 (3.88) | 7.7 (3.06) | 8.2 (5.29)
  Quantity Hours Slept Score: Week 52: number analyzed (Participants) | 32 | 43 | 15
  Quantity Hours Slept Score: Week 52 | 7.7 (4.30) | 7.7 (3.12) | 7.5 (4.93)
  Optimal Hours Slept Score: Baseline: number analyzed (Participants) | 69 | 78 | 0
  Optimal Hours Slept Score: Baseline | 0.5 (0.50) | 0.6 (0.50) |
  Optimal Hours Slept Score: Week 4: number analyzed (Participants) | 31 | 51 | 51
  Optimal Hours Slept Score: Week 4 | 0.6 (0.50) | 0.6 (0.50) | 0.5 (0.50)
  Optimal Hours Slept Score: Week 8: number analyzed (Participants) | 36 | 50 | 37
  Optimal Hours Slept Score: Week 8 | 0.7 (0.47) | 0.6 (0.49) | 0.5 (0.51)
  Optimal Hours Slept Score: Week 12: number analyzed (Participants) | 32 | 49 | 32
  Optimal Hours Slept Score: Week 12 | 0.4 (0.50) | 0.6 (0.50) | 0.6 (0.50)
  Optimal Hours Slept Score: Week 16: number analyzed (Participants) | 42 | 52 | 21
  Optimal Hours Slept Score: Week 16 | 0.5 (0.50) | 0.6 (0.50) | 0.6 (0.51)
  Optimal Hours Slept Score: Week 20: number analyzed (Participants) | 21 | 21 | 11
  Optimal Hours Slept Score: Week 20 | 0.7 (0.46) | 0.5 (0.51) | 0.6 (0.50)
  Optimal Hours Slept Score: Week 24: number analyzed (Participants) | 37 | 47 | 14
  Optimal Hours Slept Score: Week 24 | 0.4 (0.50) | 0.5 (0.51) | 0.5 (0.52)
  Optimal Hours Slept Score: Week 28: number analyzed (Participants) | 18 | 17 | 14
  Optimal Hours Slept Score: Week 28 | 0.4 (0.51) | 0.5 (0.51) | 0.6 (0.51)
  Optimal Hours Slept Score: Week 32: number analyzed (Participants) | 34 | 45 | 13
  Optimal Hours Slept Score: Week 32 | 0.5 (0.51) | 0.6 (0.50) | 0.3 (0.48)
  Optimal Hours Slept Score: Week 36: number analyzed (Participants) | 17 | 17 | 7
  Optimal Hours Slept Score: Week 36 | 0.5 (0.51) | 0.6 (0.51) | 0.7 (0.49)
  Optimal Hours Slept Score: Week 40: number analyzed (Participants) | 34 | 47 | 8
  Optimal Hours Slept Score: Week 40 | 0.5 (0.51) | 0.4 (0.49) | 0.1 (0.35)
  Optimal Hours Slept Score: Week 44: number analyzed (Participants) | 18 | 17 | 11
  Optimal Hours Slept Score: Week 44 | 0.6 (0.51) | 0.7 (0.47) | 0.2 (0.40)
  Optimal Hours Slept Score: Week 48: number analyzed (Participants) | 30 | 43 | 12
  Optimal Hours Slept Score: Week 48 | 0.6 (0.50) | 0.4 (0.50) | 0.3 (0.49)
  Optimal Hours Slept Score: Week 52: number analyzed (Participants) | 32 | 43 | 15
  Optimal Hours Slept Score: Week 52 | 0.4 (0.49) | 0.5 (0.51) | 0.4 (0.51)
  Short of Breath or Headache score: Baseline: number analyzed (Participants) | 69 | 78 | 0
  Short of Breath or Headache score: Baseline | 24.1 (9.44) | 27.2 (15.45) |
  Short of Breath or Headache score: Week 4: number analyzed (Participants) | 32 | 51 | 51
  Short of Breath or Headache score: Week 4 | 23.8 (11.85) | 23.9 (9.81) | 27.1 (13.16)
  Short of Breath or Headache score: Week 8: number analyzed (Participants) | 36 | 50 | 38
  Short of Breath or Headache score: Week 8 | 24.4 (10.81) | 25.2 (12.66) | 27.4 (17.03)
  Short of Breath or Headache score: Week 12: number analyzed (Participants) | 32 | 49 | 32
  Short of Breath or Headache score: Week 12 | 25.0 (10.16) | 26.5 (13.16) | 28.1 (15.95)
  Short of Breath or Headache score: Week 16: number analyzed (Participants) | 42 | 52 | 21
  Short of Breath or Headache score: Week 16 | 26.2 (12.87) | 25.0 (11.11) | 22.9 (9.56)
  Short of Breath or Headache score: Week 20: number analyzed (Participants) | 21 | 21 | 11
  Short of Breath or Headache score: Week 20 | 24.8 (10.78) | 29.5 (18.57) | 23.6 (12.06)
  Short of Breath or Headache score: Week 24: number analyzed (Participants) | 37 | 47 | 14
  Short of Breath or Headache score: Week 24 | 27.6 (15.88) | 27.7 (13.55) | 25.7 (12.22)
  Short of Breath or Headache score: Week 28: number analyzed (Participants) | 18 | 17 | 14
  Short of Breath or Headache score: Week 28 | 27.8 (19.57) | 29.4 (18.86) | 30.0 (15.19)
  Short of Breath or Headache score: Week 32: number analyzed (Participants) | 34 | 45 | 13
  Short of Breath or Headache score: Week 32 | 26.5 (12.76) | 23.1 (10.41) | 29.2 (15.53)
  Short of Breath or Headache score: Week 36: number analyzed (Participants) | 17 | 17 | 7
  Short of Breath or Headache score: Week 36 | 25.9 (11.76) | 23.5 (14.55) | 22.9 (7.56)
  Short of Breath or Headache score: Week 40: number analyzed (Participants) | 34 | 47 | 8
  Short of Breath or Headache score: Week 40 | 25.3 (12.37) | 26.0 (13.13) | 30.0 (21.38)
  Short of Breath or Headache score: Week 44: number analyzed (Participants) | 18 | 17 | 11
  Short of Breath or Headache score: Week 44 | 28.9 (17.11) | 27.1 (14.04) | 25.5 (12.93)
  Short of Breath or Headache score: Week 48: number analyzed (Participants) | 30 | 43 | 12
  Short of Breath or Headache score: Week 48 | 25.3 (11.67) | 26.5 (14.29) | 26.7 (13.03)
  Short of Breath or Headache score: Week 52: number analyzed (Participants) | 32 | 43 | 15
  Short of Breath or Headache score: Week 52 | 26.3 (12.89) | 27.0 (12.25) | 25.3 (11.87)
  Snoring Score: Baseline: number analyzed (Participants) | 69 | 78 | 0
  Snoring Score: Baseline | 42.9 (26.41) | 37.2 (23.40) |
  Snoring Score: Week 4: number analyzed (Participants) | 32 | 51 | 51
  Snoring Score: Week 4 | 46.9 (27.17) | 36.5 (21.43) | 41.2 (25.74)
  Snoring Score: Week 8: number analyzed (Participants) | 36 | 50 | 38
  Snoring Score: Week 8 | 47.2 (26.25) | 36.8 (22.99) | 46.8 (28.77)
  Snoring Score: Week 12: number analyzed (Participants) | 32 | 49 | 32
  Snoring Score: Week 12 | 45.6 (27.93) | 34.7 (21.12) | 40.0 (23.83)
  Snoring Score: Week 16: number analyzed (Participants) | 42 | 52 | 21
  Snoring Score: Week 16 | 43.3 (24.96) | 35.0 (20.15) | 44.8 (28.22)
  Snoring Score: Week 20: number analyzed (Participants) | 21 | 21 | 11
  Snoring Score: Week 20 | 41.9 (27.50) | 30.5 (17.46) | 38.2 (26.01)
  Snoring Score: Week 24: number analyzed (Participants) | 37 | 47 | 14
  Snoring Score: Week 24 | 50.3 (27.74) | 39.6 (24.13) | 32.9 (20.16)
  Snoring Score: Week 28: number analyzed (Participants) | 18 | 17 | 14
  Snoring Score: Week 28 | 45.6 (28.95) | 31.8 (21.28) | 32.9 (21.64)
  Snoring Score: Week 32: number analyzed (Participants) | 34 | 45 | 13
  Snoring Score: Week 32 | 42.4 (24.50) | 39.1 (22.55) | 24.6 (16.64)
  Snoring Score: Week 36: number analyzed (Participants) | 17 | 17 | 7
  Snoring Score: Week 36 | 37.6 (21.07) | 31.8 (18.79) | 40.0 (25.82)
  Snoring Score: Week 40: number analyzed (Participants) | 34 | 47 | 8
  Snoring Score: Week 40 | 44.1 (26.87) | 37.4 (21.52) | 32.5 (14.88)
  Snoring Score: Week 44: number analyzed (Participants) | 18 | 17 | 11
  Snoring Score: Week 44 | 36.7 (24.97) | 34.1 (19.70) | 34.5 (20.18)
  Snoring Score: Week 48: number analyzed (Participants) | 30 | 43 | 12
  Snoring Score: Week 48 | 44.0 (22.53) | 37.2 (23.74) | 38.3 (21.67)
  Snoring Score: Week 52: number analyzed (Participants) | 32 | 43 | 15
  Snoring Score: Week 52 | 45.6 (23.41) | 37.2 (22.07) | 37.3 (19.81)
  Sleep Disturbance Score: Baseline: number analyzed (Participants) | 69 | 78 | 0
  Sleep Disturbance Score: Baseline | 38.3 (18.74) | 34.8 (17.51) |
  Sleep Disturbance Score: Week 4: number analyzed (Participants) | 32 | 51 | 51
  Sleep Disturbance Score: Week 4 | 33.7 (15.01) | 32.2 (14.92) | 41.6 (19.69)
  Sleep Disturbance Score: Week 8: number analyzed (Participants) | 36 | 50 | 38
  Sleep Disturbance Score: Week 8 | 32.9 (13.80) | 35.3 (15.70) | 39.8 (20.46)
  Sleep Disturbance Score: Week 12: number analyzed (Participants) | 32 | 49 | 32
  Sleep Disturbance Score: Week 12 | 35.1 (16.20) | 32.8 (16.90) | 38.8 (15.51)
  Sleep Disturbance Score: Week 16: number analyzed (Participants) | 42 | 52 | 21
  Sleep Disturbance Score: Week 16 | 38.6 (19.44) | 30.8 (15.43) | 40.8 (16.03)
  Sleep Disturbance Score: Week 20: number analyzed (Participants) | 21 | 21 | 11
  Sleep Disturbance Score: Week 20 | 38.7 (22.89) | 32.1 (13.85) | 36.0 (11.92)
  Sleep Disturbance Score: Week 24: number analyzed (Participants) | 37 | 47 | 14
  Sleep Disturbance Score: Week 24 | 32.2 (19.95) | 36.3 (18.02) | 35.8 (13.29)
  Sleep Disturbance Score: Week 28: number analyzed (Participants) | 18 | 17 | 14
  Sleep Disturbance Score: Week 28 | 39.3 (22.69) | 37.2 (16.40) | 38.5 (13.20)
  Sleep Disturbance Score: Week 32: number analyzed (Participants) | 34 | 45 | 13
  Sleep Disturbance Score: Week 32 | 34.2 (20.09) | 32.0 (14.20) | 33.6 (10.53)
  Sleep Disturbance Score: Week 36: number analyzed (Participants) | 17 | 17 | 7
  Sleep Disturbance Score: Week 36 | 38.2 (23.61) | 32.2 (16.82) | 45.9 (21.67)
  Sleep Disturbance Score: Week 40: number analyzed (Participants) | 34 | 47 | 8
  Sleep Disturbance Score: Week 40 | 34.7 (18.96) | 33.0 (16.83) | 33.9 (16.91)
  Sleep Disturbance Score: Week 44: number analyzed (Participants) | 18 | 17 | 11
  Sleep Disturbance Score: Week 44 | 32.9 (23.13) | 38.9 (16.87) | 43.3 (19.70)
  Sleep Disturbance Score: Week 48: number analyzed (Participants) | 30 | 43 | 12
  Sleep Disturbance Score: Week 48 | 36.3 (18.59) | 32.1 (16.29) | 34.9 (18.61)
  Sleep Disturbance Score: Week 52: number analyzed (Participants) | 32 | 43 | 15
  Sleep Disturbance Score: Week 52 | 35.9 (19.59) | 32.9 (17.59) | 28.1 (9.24)
  Sleep Adequacy Score: Baseline: number analyzed (Participants) | 69 | 78 | 0
  Sleep Adequacy Score: Baseline | 68.6 (18.25) | 69.1 (21.69) |
  Sleep Adequacy Score: Week 4: number analyzed (Participants) | 32 | 51 | 51
  Sleep Adequacy Score: Week 4 | 70.6 (20.15) | 71.6 (18.80) | 68.4 (19.53)
  Sleep Adequacy Score: Week 8: number analyzed (Participants) | 36 | 50 | 38
  Sleep Adequacy Score: Week 8 | 72.5 (16.45) | 72.6 (20.58) | 66.1 (24.11)
  Sleep Adequacy Score: Week 12: number analyzed (Participants) | 32 | 49 | 32
  Sleep Adequacy Score: Week 12 | 71.9 (22.92) | 68.2 (21.47) | 70.9 (20.69)
  Sleep Adequacy Score: Week 16: number analyzed (Participants) | 42 | 52 | 21
  Sleep Adequacy Score: Week 16 | 73.3 (20.20) | 69.0 (18.71) | 71.4 (16.52)
  Sleep Adequacy Score: Week 20: number analyzed (Participants) | 21 | 21 | 11
  Sleep Adequacy Score: Week 20 | 70.5 (21.56) | 67.6 (17.86) | 75.5 (16.35)
  Sleep Adequacy Score: Week 24: number analyzed (Participants) | 37 | 47 | 14
  Sleep Adequacy Score: Week 24 | 71.6 (21.02) | 67.4 (20.59) | 70.7 (18.17)
  Sleep Adequacy Score: Week 28: number analyzed (Participants) | 18 | 17 | 14
  Sleep Adequacy Score: Week 28 | 71.7 (22.03) | 71.2 (21.47) | 64.3 (19.89)
  Sleep Adequacy Score: Week 32: number analyzed (Participants) | 34 | 45 | 13
  Sleep Adequacy Score: Week 32 | 74.7 (21.21) | 72.4 (19.67) | 64.6 (23.67)
  Sleep Adequacy Score: Week 36: number analyzed (Participants) | 17 | 17 | 7
  Sleep Adequacy Score: Week 36 | 74.1 (22.38) | 68.8 (15.76) | 62.9 (25.63)
  Sleep Adequacy Score: Week 40: number analyzed (Participants) | 34 | 47 | 8
  Sleep Adequacy Score: Week 40 | 68.5 (21.34) | 69.1 (18.51) | 67.5 (23.15)
  Sleep Adequacy Score: Week 44: number analyzed (Participants) | 18 | 17 | 11
  Sleep Adequacy Score: Week 44 | 72.2 (22.90) | 70.0 (21.79) | 60.9 (21.19)
  Sleep Adequacy Score: Week 48: number analyzed (Participants) | 30 | 43 | 12
  Sleep Adequacy Score: Week 48 | 73.0 (18.96) | 70.2 (19.70) | 65.8 (19.75)
  Sleep Adequacy Score: Week 52: number analyzed (Participants) | 32 | 43 | 15
  Sleep Adequacy Score: Week 52 | 70.0 (20.48) | 68.6 (22.74) | 68.0 (18.97)
  Sleep Somnolence Score: Baseline: number analyzed (Participants) | 69 | 78 | 0
  Sleep Somnolence Score: Baseline | 40.3 (17.05) | 41.8 (18.51) |
  Sleep Somnolence Score: Week 4: number analyzed (Participants) | 32 | 51 | 51
  Sleep Somnolence Score: Week 4 | 39.6 (15.23) | 42.4 (18.13) | 44.8 (20.87)
  Sleep Somnolence Score: Week 8: number analyzed (Participants) | 36 | 50 | 38
  Sleep Somnolence Score: Week 8 | 36.5 (10.75) | 40.1 (18.78) | 46.7 (21.81)
  Sleep Somnolence Score: Week 12: number analyzed (Participants) | 32 | 49 | 32
  Sleep Somnolence Score: Week 12 | 41.7 (18.86) | 40.4 (18.48) | 43.8 (21.15)
  Sleep Somnolence Score: Week 16: number analyzed (Participants) | 42 | 52 | 21
  Sleep Somnolence Score: Week 16 | 37.1 (16.00) | 39.1 (17.06) | 47.0 (18.07)
  Sleep Somnolence Score: Week 20: number analyzed (Participants) | 21 | 21 | 11
  Sleep Somnolence Score: Week 20 | 41.3 (19.62) | 37.5 (17.82) | 40.0 (18.14)
  Sleep Somnolence Score: Week 24: number analyzed (Participants) | 37 | 47 | 14
  Sleep Somnolence Score: Week 24 | 39.5 (17.02) | 43.4 (18.06) | 39.0 (16.71)
  Sleep Somnolence Score: Week 28: number analyzed (Participants) | 18 | 17 | 14
  Sleep Somnolence Score: Week 28 | 44.4 (21.57) | 41.2 (19.33) | 46.7 (17.15)
  Sleep Somnolence Score: Week 32: number analyzed (Participants) | 34 | 45 | 13
  Sleep Somnolence Score: Week 32 | 43.7 (21.16) | 41.5 (15.63) | 48.2 (17.46)
  Sleep Somnolence Score: Week 36: number analyzed (Participants) | 17 | 17 | 7
  Sleep Somnolence Score: Week 36 | 34.9 (17.41) | 39.2 (14.70) | 45.7 (24.77)
  Sleep Somnolence Score: Week 40: number analyzed (Participants) | 34 | 47 | 8
  Sleep Somnolence Score: Week 40 | 38.6 (17.96) | 43.3 (14.70) | 41.7 (25.88)
  Sleep Somnolence Score: Week 44: number analyzed (Participants) | 18 | 17 | 11
  Sleep Somnolence Score: Week 44 | 39.3 (17.84) | 44.3 (16.99) | 50.3 (26.89)
  Sleep Somnolence Score: Week 48: number analyzed (Participants) | 30 | 43 | 12
  Sleep Somnolence Score: Week 48 | 41.3 (15.40) | 42.3 (13.48) | 46.1 (23.52)
  Sleep Somnolence Score: Week 52: number analyzed (Participants) | 32 | 43 | 15
  Sleep Somnolence Score: Week 52 | 39.0 (16.60) | 40.0 (14.47) | 44.4 (20.57)
  Sleep Problems Index I Score: Baseline: number analyzed (Participants) | 69 | 78 | 0
  Sleep Problems Index I Score: Baseline | 33.4 (12.63) | 33.2 (14.19) |
  Sleep Problems Index I Score: Week 4: number analyzed (Participants) | 32 | 51 | 51
  Sleep Problems Index I Score: Week 4 | 31.4 (13.22) | 31.6 (11.53) | 35.6 (13.51)
  Sleep Problems Index I Score: Week 8: number analyzed (Participants) | 36 | 50 | 38
  Sleep Problems Index I Score: Week 8 | 29.6 (10.77) | 31.5 (13.98) | 36.1 (16.52)
  Sleep Problems Index I Score: Week 12: number analyzed (Participants) | 32 | 49 | 32
  Sleep Problems Index I Score: Week 12 | 32.2 (14.36) | 33.3 (12.89) | 34.1 (13.03)
  Sleep Problems Index I Score: Week 16: number analyzed (Participants) | 42 | 52 | 21
  Sleep Problems Index I Score: Week 16 | 32.1 (14.44) | 31.8 (12.14) | 34.0 (9.92)
  Sleep Problems Index I Score: Week 20: number analyzed (Participants) | 21 | 21 | 11
  Sleep Problems Index I Score: Week 20 | 34.0 (16.21) | 32.9 (13.01) | 29.7 (7.67)
  Sleep Problems Index I Score: Week 24: number analyzed (Participants) | 37 | 47 | 14
  Sleep Problems Index I Score: Week 24 | 30.9 (14.92) | 34.6 (13.63) | 30.7 (9.71)
  Sleep Problems Index I Score: Week 28: number analyzed (Participants) | 18 | 17 | 14
  Sleep Problems Index I Score: Week 28 | 34.4 (18.22) | 32.9 (13.74) | 37.9 (13.18)
  Sleep Problems Index I Score: Week 32: number analyzed (Participants) | 34 | 45 | 13
  Sleep Problems Index I Score: Week 32 | 31.7 (14.10) | 30.5 (11.72) | 35.1 (13.92)
  Sleep Problems Index I Score: Week 36: number analyzed (Participants) | 17 | 17 | 7
  Sleep Problems Index I Score: Week 36 | 31.4 (18.11) | 31.6 (12.86) | 35.2 (12.00)
  Sleep Problems Index I Score: Week 40: number analyzed (Participants) | 34 | 47 | 8
  Sleep Problems Index I Score: Week 40 | 33.0 (15.07) | 33.7 (13.55) | 34.6 (17.27)
  Sleep Problems Index I Score: Week 44: number analyzed (Participants) | 18 | 17 | 11
  Sleep Problems Index I Score: Week 44 | 32.4 (18.32) | 33.5 (13.25) | 38.5 (14.86)
  Sleep Problems Index I Score: Week 48: number analyzed (Participants) | 30 | 43 | 12
  Sleep Problems Index I Score: Week 48 | 33.3 (15.06) | 32.0 (12.20) | 34.4 (11.66)
  Sleep Problems Index I Score: Week 52: number analyzed (Participants) | 32 | 43 | 15
  Sleep Problems Index I Score: Week 52 | 32.4 (13.92) | 32.6 (14.08) | 31.6 (9.91)
  Sleep Problems Index II Score: Baseline: number analyzed (Participants) | 69 | 78 | 0
  Sleep Problems Index II Score: Baseline | 35.5 (13.20) | 34.4 (14.17) |
  Sleep Problems Index II Score: Week 4: number analyzed (Participants) | 32 | 51 | 51
  Sleep Problems Index II Score: Week 4 | 32.6 (11.70) | 32.1 (11.57) | 38.2 (14.53)
  Sleep Problems Index II Score: Week 8: number analyzed (Participants) | 36 | 50 | 38
  Sleep Problems Index II Score: Week 8 | 31.4 (10.70) | 33.1 (13.16) | 38.5 (17.14)
  Sleep Problems Index II Score: Week 12: number analyzed (Participants) | 32 | 49 | 32
  Sleep Problems Index II Score: Week 12 | 33.2 (14.40) | 33.2 (13.21) | 36.4 (13.26)
  Sleep Problems Index II Score: Week 16: number analyzed (Participants) | 42 | 52 | 21
  Sleep Problems Index II Score: Week 16 | 33.9 (15.58) | 32.0 (11.95) | 36.8 (11.34)
  Sleep Problems Index II Score: Week 20: number analyzed (Participants) | 21 | 21 | 11
  Sleep Problems Index II Score: Week 20 | 35.9 (17.75) | 33.1 (11.87) | 32.0 (8.63)
  Sleep Problems Index II Score: Week 24: number analyzed (Participants) | 37 | 47 | 14
  Sleep Problems Index II Score: Week 24 | 32.1 (15.49) | 35.9 (13.54) | 33.8 (11.25)
  Sleep Problems Index II Score: Week 28: number analyzed (Participants) | 18 | 17 | 14
  Sleep Problems Index II Score: Week 28 | 36.7 (18.79) | 35.0 (13.07) | 38.8 (11.64)
  Sleep Problems Index II Score: Week 32: number analyzed (Participants) | 34 | 45 | 13
  Sleep Problems Index II Score: Week 32 | 33.5 (14.89) | 31.6 (11.07) | 36.3 (12.86)
  Sleep Problems Index II Score: Week 36: number analyzed (Participants) | 17 | 17 | 7
  Sleep Problems Index II Score: Week 36 | 33.5 (19.04) | 32.2 (12.20) | 40.7 (14.56)
  Sleep Problems Index II Score: Week 40: number analyzed (Participants) | 34 | 47 | 8
  Sleep Problems Index II Score: Week 40 | 33.7 (15.62) | 33.9 (12.86) | 34.8 (16.31)
  Sleep Problems Index II Score: Week 44: number analyzed (Participants) | 18 | 17 | 11
  Sleep Problems Index II Score: Week 44 | 33.0 (18.97) | 36.9 (13.73) | 41.7 (15.83)
  Sleep Problems Index II Score: Week 48: number analyzed (Participants) | 30 | 43 | 12
  Sleep Problems Index II Score: Week 48 | 33.7 (15.44) | 32.9 (12.13) | 36.8 (13.82)
  Sleep Problems Index II Score: Week 52: number analyzed (Participants) | 32 | 43 | 15
  Sleep Problems Index II Score: Week 52 | 33.8 (14.86) | 33.0 (13.66) | 32.2 (10.53)

45. Secondary Outcome: Medical Outcome Study Sleep Scale Score in Participants >=12 Years of Age: First Flare Period
Description: as for outcome 44
Time Frame: Weeks 0, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 43 | 44
Units on a scale
  Quantity Hours Slept Score: Week 0: number analyzed (Participants) | 42 | 44
  Quantity Hours Slept Score: Week 0 | 7.3 (2.28) | 7.6 (3.56)
  Quantity Hours Slept Score: Week 4: number analyzed (Participants) | 21 | 24
  Quantity Hours Slept Score: Week 4 | 8.2 (3.88) | 7.3 (1.55)
  Quantity Hours Slept Score: Week 8: number analyzed (Participants) | 13 | 15
  Quantity Hours Slept Score: Week 8 | 8.3 (3.45) | 6.9 (1.68)
  Quantity Hours Slept Score: Week 12: number analyzed (Participants) | 3 | 7
  Quantity Hours Slept Score: Week 12 | 8.0 (1.00) | 7.3 (1.70)
  Optimal Hours Slept Score: Week 0: number analyzed (Participants) | 42 | 44
  Optimal Hours Slept Score: Week 0 | 0.6 (0.49) | 0.4 (0.50)
  Optimal Hours Slept Score: Week 4: number analyzed (Participants) | 21 | 24
  Optimal Hours Slept Score: Week 4 | 0.5 (0.51) | 0.6 (0.50)
  Optimal Hours Slept Score: Week 8: number analyzed (Participants) | 13 | 15
  Optimal Hours Slept Score: Week 8 | 0.5 (0.52) | 0.5 (0.52)
  Optimal Hours Slept Score: Week 12: number analyzed (Participants) | 3 | 7
  Optimal Hours Slept Score: Week 12 | 0.7 (0.58) | 0.4 (0.53)
  Short of Breath or Headache score: Week 0 | 27.9 (16.98) | 28.6 (17.47)
  Short of Breath or Headache score: Week 4: number analyzed (Participants) | 21 | 24
  Short of Breath or Headache score: Week 4 | 26.7 (13.17) | 27.5 (14.22)
  Short of Breath or Headache score: Week 8: number analyzed (Participants) | 13 | 15
  Short of Breath or Headache score: Week 8 | 27.7 (15.36) | 33.3 (19.52)
  Short of Breath or Headache score: Week 12: number analyzed (Participants) | 3 | 7
  Short of Breath or Headache score: Week 12 | 20.0 (0.00) | 22.9 (7.56)
  Snoring Score: Week 0 | 43.3 (28.26) | 37.7 (24.86)
  Snoring Score: Week 4: number analyzed (Participants) | 21 | 24
  Snoring Score: Week 4 | 45.7 (28.39) | 39.2 (27.96)
  Snoring Score: Week 8: number analyzed (Participants) | 13 | 15
  Snoring Score: Week 8 | 44.6 (24.70) | 38.7 (23.26)
  Snoring Score: Week 12: number analyzed (Participants) | 3 | 7
  Snoring Score: Week 12 | 53.3 (23.09) | 34.3 (19.02)
  Sleep Disturbance Score: Week 0 | 41.0 (19.08) | 40.9 (19.39)
  Sleep Disturbance Score: Week 4: number analyzed (Participants) | 21 | 24
  Sleep Disturbance Score: Week 4 | 38.3 (18.36) | 38.6 (18.61)
  Sleep Disturbance Score: Week 8: number analyzed (Participants) | 13 | 15
  Sleep Disturbance Score: Week 8 | 33.6 (12.81) | 41.4 (16.77)
  Sleep Disturbance Score: Week 12: number analyzed (Participants) | 3 | 7
  Sleep Disturbance Score: Week 12 | 43.3 (16.65) | 43.6 (13.02)
  Sleep Adequacy Score: Week 0 | 67.0 (20.99) | 66.1 (20.71)
  Sleep Adequacy Score: Week 4: number analyzed (Participants) | 21 | 24
  Sleep Adequacy Score: Week 4 | 71.0 (23.00) | 67.1 (24.22)
  Sleep Adequacy Score: Week 8: number analyzed (Participants) | 13 | 15
  Sleep Adequacy Score: Week 8 | 70.0 (22.36) | 66.0 (19.20)
  Sleep Adequacy Score: Week 12: number analyzed (Participants) | 3 | 7
  Sleep Adequacy Score: Week 12 | 76.7 (15.28) | 64.3 (17.18)
  Sleep Somnolence Score: Week 0 | 44.8 (20.74) | 45.9 (19.30)
  Sleep Somnolence Score: Week 4: number analyzed (Participants) | 21 | 24
  Sleep Somnolence Score: Week 4 | 42.9 (22.76) | 48.3 (19.49)
  Sleep Somnolence Score: Week 8: number analyzed (Participants) | 13 | 15
  Sleep Somnolence Score: Week 8 | 45.6 (22.91) | 54.2 (19.17)
  Sleep Somnolence Score: Week 12: number analyzed (Participants) | 3 | 7
  Sleep Somnolence Score: Week 12 | 33.3 (13.33) | 50.5 (19.57)
  Sleep Problems Index I Score: Week 0 | 36.3 (13.53) | 37.3 (15.29)
  Sleep Problems Index I Score: Week 4: number analyzed (Participants) | 21 | 24
  Sleep Problems Index I Score: Week 4 | 32.9 (16.27) | 36.7 (16.33)
  Sleep Problems Index I Score: Week 8: number analyzed (Participants) | 13 | 15
  Sleep Problems Index I Score: Week 8 | 32.8 (9.51) | 38.9 (13.07)
  Sleep Problems Index I Score: Week 12: number analyzed (Participants) | 3 | 7
  Sleep Problems Index I Score: Week 12 | 31.1 (11.71) | 39.0 (5.35)
  Sleep Problems Index II Score: Week 0 | 38.4 (14.19) | 38.6 (15.55)
  Sleep Problems Index II Score: Week 4: number analyzed (Participants) | 21 | 24
  Sleep Problems Index II Score: Week 4 | 35.8 (16.81) | 38.0 (16.06)
  Sleep Problems Index II Score: Week 8: number analyzed (Participants) | 13 | 15
  Sleep Problems Index II Score: Week 8 | 34.6 (10.26) | 41.4 (13.30)
  Sleep Problems Index II Score: Week 12: number analyzed (Participants) | 3 | 7
  Sleep Problems Index II Score: Week 12 | 34.1 (12.97) | 40.3 (6.13)

46. Secondary Outcome: Medical Outcome Study Sleep Scale Score in Participants >=12 Years of Age: First Flare Free Period
Description: as for outcome 44
Time Frame: as for outcome 32
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 69 | 78
Units on a scale
  Quantity Hours Slept Score: Baseline | 8.3 (3.79) | 7.5 (2.42)
  Quantity Hours Slept Score: Week 4: number analyzed (Participants) | 29 | 51
  Quantity Hours Slept Score: Week 4 | 9.0 (4.68) | 8.1 (3.32)
  Quantity Hours Slept Score: Week 8: number analyzed (Participants) | 25 | 44
  Quantity Hours Slept Score: Week 8 | 8.5 (3.77) | 7.9 (3.92)
  Quantity Hours Slept Score: Week 12: number analyzed (Participants) | 20 | 40
  Quantity Hours Slept Score: Week 12 | 8.6 (4.15) | 7.6 (3.22)
  Quantity Hours Slept Score: Week 16: number analyzed (Participants) | 19 | 37
  Quantity Hours Slept Score: Week 16 | 8.5 (4.11) | 8.5 (4.90)
  Quantity Hours Slept Score: Week 20: number analyzed (Participants) | 8 | 13
  Quantity Hours Slept Score: Week 20 | 7.0 (1.20) | 7.7 (1.55)
  Quantity Hours Slept Score: Week 24: number analyzed (Participants) | 17 | 31
  Quantity Hours Slept Score: Week 24 | 7.2 (1.99) | 7.4 (3.45)
  Quantity Hours Slept Score: Week 28: number analyzed (Participants) | 7 | 9
  Quantity Hours Slept Score: Week 28 | 6.9 (1.07) | 7.4 (1.51)
  Quantity Hours Slept Score: Week 32: number analyzed (Participants) | 16 | 27
  Quantity Hours Slept Score: Week 32 | 8.5 (4.24) | 7.6 (1.22)
  Quantity Hours Slept Score: Week 36: number analyzed (Participants) | 6 | 7
  Quantity Hours Slept Score: Week 36 | 7.0 (0.89) | 8.0 (1.41)
  Quantity Hours Slept Score: Week 40: number analyzed (Participants) | 17 | 26
  Quantity Hours Slept Score: Week 40 | 8.3 (4.57) | 7.5 (2.97)
  Quantity Hours Slept Score: Week 44: number analyzed (Participants) | 7 | 9
  Quantity Hours Slept Score: Week 44 | 6.7 (1.11) | 7.1 (0.60)
  Quantity Hours Slept Score: Week 48: number analyzed (Participants) | 17 | 24
  Quantity Hours Slept Score: Week 48 | 7.2 (1.63) | 7.2 (1.46)
  Quantity Hours Slept Score: Week 52: number analyzed (Participants) | 15 | 23
  Quantity Hours Slept Score: Week 52 | 8.0 (4.57) | 7.0 (1.24)
  Optimal Hours Slept Score: Baseline | 0.5 (0.50) | 0.6 (0.50)
  Optimal Hours Slept Score: Week 4: number analyzed (Participants) | 29 | 51
  Optimal Hours Slept Score: Week 4 | 0.6 (0.50) | 0.6 (0.50)
  Optimal Hours Slept Score: Week 8: number analyzed (Participants) | 25 | 44
  Optimal Hours Slept Score: Week 8 | 0.7 (0.46) | 0.6 (0.49)
  Optimal Hours Slept Score: Week 12: number analyzed (Participants) | 20 | 40
  Optimal Hours Slept Score: Week 12 | 0.4 (0.50) | 0.6 (0.50)
  Optimal Hours Slept Score: Week 16: number analyzed (Participants) | 19 | 37
  Optimal Hours Slept Score: Week 16 | 0.5 (0.51) | 0.6 (0.50)
  Optimal Hours Slept Score: Week 20: number analyzed (Participants) | 8 | 13
  Optimal Hours Slept Score: Week 20 | 0.6 (0.52) | 0.5 (0.52)
  Optimal Hours Slept Score: Week 24: number analyzed (Participants) | 17 | 31
  Optimal Hours Slept Score: Week 24 | 0.5 (0.51) | 0.6 (0.50)
  Optimal Hours Slept Score: Week 28: number analyzed (Participants) | 7 | 9
  Optimal Hours Slept Score: Week 28 | 0.7 (0.49) | 0.6 (0.53)
  Optimal Hours Slept Score: Week 32: number analyzed (Participants) | 16 | 27
  Optimal Hours Slept Score: Week 32 | 0.6 (0.50) | 0.7 (0.45)
  Optimal Hours Slept Score: Week 36: number analyzed (Participants) | 6 | 7
  Optimal Hours Slept Score: Week 36 | 0.7 (0.52) | 0.9 (0.38)
  Optimal Hours Slept Score: Week 40: number analyzed (Participants) | 17 | 26
  Optimal Hours Slept Score: Week 40 | 0.5 (0.51) | 0.5 (0.51)
  Optimal Hours Slept Score: Week 44: number analyzed (Participants) | 7 | 9
  Optimal Hours Slept Score: Week 44 | 0.6 (0.53) | 0.9 (0.33)
  Optimal Hours Slept Score: Week 48: number analyzed (Participants) | 17 | 24
  Optimal Hours Slept Score: Week 48 | 0.6 (0.51) | 0.4 (0.50)
  Optimal Hours Slept Score: Week 52: number analyzed (Participants) | 15 | 23
  Optimal Hours Slept Score: Week 52 | 0.4 (0.51) | 0.5 (0.51)
  Short of Breath or Headache score: Baseline | 24.1 (9.44) | 27.2 (15.45)
  Short of Breath or Headache score: Week 4: number analyzed (Participants) | 30 | 51
  Short of Breath or Headache score: Week 4 | 24.0 (12.21) | 23.9 (9.81)
  Short of Breath or Headache score: Week 8: number analyzed (Participants) | 25 | 44
  Short of Breath or Headache score: Week 8 | 24.8 (10.46) | 23.6 (9.90)
  Short of Breath or Headache score: Week 12: number analyzed (Participants) | 20 | 40
  Short of Breath or Headache score: Week 12 | 23.0 (7.33) | 26.0 (12.97)
  Short of Breath or Headache score: Week 16: number analyzed (Participants) | 19 | 37
  Short of Breath or Headache score: Week 16 | 24.2 (8.38) | 24.9 (10.96)
  Short of Breath or Headache score: Week 20: number analyzed (Participants) | 8 | 13
  Short of Breath or Headache score: Week 20 | 22.5 (7.07) | 29.2 (17.54)
  Short of Breath or Headache score: Week 24: number analyzed (Participants) | 17 | 31
  Short of Breath or Headache score: Week 24 | 24.7 (11.25) | 26.5 (11.99)
  Short of Breath or Headache score: Week 28: number analyzed (Participants) | 7 | 9
  Short of Breath or Headache score: Week 28 | 31.4 (22.68) | 26.7 (14.14)
  Short of Breath or Headache score: Week 32: number analyzed (Participants) | 16 | 27
  Short of Breath or Headache score: Week 32 | 25.0 (8.94) | 22.2 (8.47)
  Short of Breath or Headache score: Week 36: number analyzed (Participants) | 6 | 7
  Short of Breath or Headache score: Week 36 | 20.0 (0.00) | 20.0 (0.00)
  Short of Breath or Headache score: Week 40: number analyzed (Participants) | 17 | 26
  Short of Breath or Headache score: Week 40 | 22.4 (6.64) | 25.4 (12.08)
  Short of Breath or Headache score: Week 44: number analyzed (Participants) | 7 | 9
  Short of Breath or Headache score: Week 44 | 22.9 (7.56) | 28.9 (14.53)
  Short of Breath or Headache score: Week 48: number analyzed (Participants) | 17 | 24
  Short of Breath or Headache score: Week 48 | 22.4 (6.64) | 25.0 (12.16)
  Short of Breath or Headache score: Week 52: number analyzed (Participants) | 15 | 23
  Short of Breath or Headache score: Week 52 | 22.7 (7.04) | 27.8 (11.66)
  Snoring Score: Baseline | 42.9 (26.41) | 37.2 (23.40)
  Snoring Score: Week 4: number analyzed (Participants) | 30 | 51
  Snoring Score: Week 4 | 47.3 (27.53) | 36.5 (21.43)
  Snoring Score: Week 8: number analyzed (Participants) | 25 | 44
  Snoring Score: Week 8 | 49.6 (26.53) | 35.5 (22.77)
  Snoring Score: Week 12: number analyzed (Participants) | 20 | 40
  Snoring Score: Week 12 | 49.0 (28.64) | 33.5 (20.95)
  Snoring Score: Week 16: number analyzed (Participants) | 19 | 37
  Snoring Score: Week 16 | 45.3 (27.36) | 34.6 (19.80)
  Snoring Score: Week 20: number analyzed (Participants) | 8 | 13
  Snoring Score: Week 20 | 42.5 (27.12) | 23.1 (7.51)
  Snoring Score: Week 24: number analyzed (Participants) | 17 | 31
  Snoring Score: Week 24 | 54.1 (26.23) | 38.1 (22.72)
  Snoring Score: Week 28: number analyzed (Participants) | 7 | 9
  Snoring Score: Week 28 | 48.6 (30.24) | 22.2 (6.67)
  Snoring Score: Week 32: number analyzed (Participants) | 16 | 27
  Snoring Score: Week 32 | 40.0 (19.32) | 37.8 (21.72)
  Snoring Score: Week 36: number analyzed (Participants) | 6 | 7
  Snoring Score: Week 36 | 36.7 (15.06) | 25.7 (9.76)
  Snoring Score: Week 40: number analyzed (Participants) | 17 | 26
  Snoring Score: Week 40 | 44.7 (26.01) | 38.5 (21.85)
  Snoring Score: Week 44: number analyzed (Participants) | 7 | 9
  Snoring Score: Week 44 | 28.6 (10.69) | 28.9 (14.53)
  Snoring Score: Week 48: number analyzed (Participants) | 17 | 24
  Snoring Score: Week 48 | 44.7 (16.63) | 40.0 (24.32)
  Snoring Score: Week 52: number analyzed (Participants) | 15 | 23
  Snoring Score: Week 52 | 46.7 (20.93) | 41.7 (21.67)
  Sleep Disturbance Score: Baseline | 38.3 (18.74) | 34.8 (17.51)
  Sleep Disturbance Score: Week 4: number analyzed (Participants) | 30 | 51
  Sleep Disturbance Score: Week 4 | 34.3 (15.11) | 32.2 (14.92)
  Sleep Disturbance Score: Week 8: number analyzed (Participants) | 25 | 44
  Sleep Disturbance Score: Week 8 | 31.7 (12.00) | 35.1 (16.27)
  Sleep Disturbance Score: Week 12: number analyzed (Participants) | 20 | 40
  Sleep Disturbance Score: Week 12 | 33.3 (14.51) | 32.3 (17.12)
  Sleep Disturbance Score: Week 16: number analyzed (Participants) | 19 | 37
  Sleep Disturbance Score: Week 16 | 35.9 (17.17) | 30.6 (14.57)
  Sleep Disturbance Score: Week 20: number analyzed (Participants) | 8 | 13
  Sleep Disturbance Score: Week 20 | 32.8 (12.22) | 28.0 (9.31)
  Sleep Disturbance Score: Week 24: number analyzed (Participants) | 17 | 31
  Sleep Disturbance Score: Week 24 | 30.7 (15.90) | 35.9 (18.34)
  Sleep Disturbance Score: Week 28: number analyzed (Participants) | 7 | 9
  Sleep Disturbance Score: Week 28 | 37.3 (11.78) | 31.1 (12.43)
  Sleep Disturbance Score: Week 32: number analyzed (Participants) | 16 | 27
  Sleep Disturbance Score: Week 32 | 31.4 (14.75) | 32.3 (12.28)
  Sleep Disturbance Score: Week 36: number analyzed (Participants) | 6 | 7
  Sleep Disturbance Score: Week 36 | 27.7 (9.43) | 27.7 (10.93)
  Sleep Disturbance Score: Week 40: number analyzed (Participants) | 17 | 26
  Sleep Disturbance Score: Week 40 | 34.3 (14.80) | 33.2 (18.06)
  Sleep Disturbance Score: Week 44: number analyzed (Participants) | 7 | 9
  Sleep Disturbance Score: Week 44 | 23.9 (10.47) | 34.3 (16.25)
  Sleep Disturbance Score: Week 48: number analyzed (Participants) | 17 | 24
  Sleep Disturbance Score: Week 48 | 33.9 (11.81) | 30.2 (16.76)
  Sleep Disturbance Score: Week 52: number analyzed (Participants) | 15 | 23
  Sleep Disturbance Score: Week 52 | 32.4 (16.27) | 31.6 (15.29)
  Sleep Adequacy Score: Baseline | 68.6 (18.25) | 69.1 (21.69)
  Sleep Adequacy Score: Week 4: number analyzed (Participants) | 30 | 51
  Sleep Adequacy Score: Week 4 | 71.0 (20.74) | 71.6 (18.80)
  Sleep Adequacy Score: Week 8: number analyzed (Participants) | 25 | 44
  Sleep Adequacy Score: Week 8 | 72.8 (17.20) | 73.2 (21.43)
  Sleep Adequacy Score: Week 12: number analyzed (Participants) | 20 | 40
  Sleep Adequacy Score: Week 12 | 75.0 (20.90) | 68.0 (21.74)
  Sleep Adequacy Score: Week 16: number analyzed (Participants) | 19 | 37
  Sleep Adequacy Score: Week 16 | 74.7 (20.65) | 66.5 (17.98)
  Sleep Adequacy Score: Week 20: number analyzed (Participants) | 8 | 13
  Sleep Adequacy Score: Week 20 | 70.0 (22.68) | 66.9 (21.36)
  Sleep Adequacy Score: Week 24: number analyzed (Participants) | 17 | 31
  Sleep Adequacy Score: Week 24 | 76.5 (16.18) | 68.1 (20.88)
  Sleep Adequacy Score: Week 28: number analyzed (Participants) | 7 | 9
  Sleep Adequacy Score: Week 28 | 70.0 (19.15) | 72.2 (28.19)
  Sleep Adequacy Score: Week 32: number analyzed (Participants) | 16 | 27
  Sleep Adequacy Score: Week 32 | 78.8 (14.55) | 74.4 (19.87)
  Sleep Adequacy Score: Week 36: number analyzed (Participants) | 6 | 7
  Sleep Adequacy Score: Week 36 | 75.0 (15.17) | 72.9 (17.99)
  Sleep Adequacy Score: Week 40: number analyzed (Participants) | 17 | 26
  Sleep Adequacy Score: Week 40 | 72.9 (16.11) | 68.1 (18.33)
  Sleep Adequacy Score: Week 44: number analyzed (Participants) | 7 | 9
  Sleep Adequacy Score: Week 44 | 67.1 (26.28) | 73.3 (26.46)
  Sleep Adequacy Score: Week 48: number analyzed (Participants) | 17 | 24
  Sleep Adequacy Score: Week 48 | 75.3 (14.63) | 72.9 (18.99)
  Sleep Adequacy Score: Week 52: number analyzed (Participants) | 15 | 23
  Sleep Adequacy Score: Week 52 | 74.7 (13.56) | 67.8 (23.35)
  Sleep Somnolence Score: Baseline | 40.3 (17.05) | 41.8 (18.51)
  Sleep Somnolence Score: Week 4: number analyzed (Participants) | 30 | 51
  Sleep Somnolence Score: Week 4 | 40.0 (15.56) | 42.4 (18.13)
  Sleep Somnolence Score: Week 8: number analyzed (Participants) | 25 | 44
  Sleep Somnolence Score: Week 8 | 36.3 (10.55) | 39.1 (18.89)
  Sleep Somnolence Score: Week 12: number analyzed (Participants) | 20 | 40
  Sleep Somnolence Score: Week 12 | 38.0 (14.03) | 41.3 (18.81)
  Sleep Somnolence Score: Week 16: number analyzed (Participants) | 19 | 37
  Sleep Somnolence Score: Week 16 | 34.4 (10.00) | 40.5 (17.38)
  Sleep Somnolence Score: Week 20: number analyzed (Participants) | 8 | 13
  Sleep Somnolence Score: Week 20 | 42.5 (24.67) | 36.9 (20.66)
  Sleep Somnolence Score: Week 24: number analyzed (Participants) | 17 | 31
  Sleep Somnolence Score: Week 24 | 39.6 (16.07) | 42.8 (19.98)
  Sleep Somnolence Score: Week 28: number analyzed (Participants) | 7 | 9
  Sleep Somnolence Score: Week 28 | 48.6 (24.26) | 37.0 (20.03)
  Sleep Somnolence Score: Week 32: number analyzed (Participants) | 16 | 27
  Sleep Somnolence Score: Week 32 | 44.6 (20.76) | 42.5 (15.04)
  Sleep Somnolence Score: Week 36: number analyzed (Participants) | 6 | 7
  Sleep Somnolence Score: Week 36 | 35.6 (19.63) | 31.4 (9.20)
  Sleep Somnolence Score: Week 40: number analyzed (Participants) | 17 | 26
  Sleep Somnolence Score: Week 40 | 36.1 (16.51) | 43.1 (15.35)
  Sleep Somnolence Score: Week 44: number analyzed (Participants) | 7 | 9
  Sleep Somnolence Score: Week 44 | 37.1 (16.71) | 40.7 (18.99)
  Sleep Somnolence Score: Week 48: number analyzed (Participants) | 17 | 24
  Sleep Somnolence Score: Week 48 | 39.6 (14.62) | 43.1 (13.04)
  Sleep Somnolence Score: Week 52: number analyzed (Participants) | 15 | 23
  Sleep Somnolence Score: Week 52 | 38.7 (13.14) | 39.1 (14.11)
  Sleep Problems Index I Score: Baseline | 33.4 (12.63) | 33.2 (14.19)
  Sleep Problems Index I Score: Week 4: number analyzed (Participants) | 30 | 51
  Sleep Problems Index I Score: Week 4 | 31.4 (13.64) | 31.6 (11.53)
  Sleep Problems Index I Score: Week 8: number analyzed (Participants) | 25 | 44
  Sleep Problems Index I Score: Week 8 | 28.9 (10.79) | 30.7 (13.99)
  Sleep Problems Index I Score: Week 12: number analyzed (Participants) | 20 | 40
  Sleep Problems Index I Score: Week 12 | 29.3 (13.27) | 33.2 (13.22)
  Sleep Problems Index I Score: Week 16: number analyzed (Participants) | 19 | 37
  Sleep Problems Index I Score: Week 16 | 30.2 (11.78) | 32.6 (12.10)
  Sleep Problems Index I Score: Week 20: number analyzed (Participants) | 8 | 13
  Sleep Problems Index I Score: Week 20 | 32.5 (12.05) | 31.8 (14.12)
  Sleep Problems Index I Score: Week 24: number analyzed (Participants) | 17 | 31
  Sleep Problems Index I Score: Week 24 | 28.0 (12.25) | 34.4 (14.87)
  Sleep Problems Index I Score: Week 28: number analyzed (Participants) | 7 | 9
  Sleep Problems Index I Score: Week 28 | 35.7 (13.97) | 28.5 (13.34)
  Sleep Problems Index I Score: Week 32: number analyzed (Participants) | 16 | 27
  Sleep Problems Index I Score: Week 32 | 29.2 (8.39) | 30.5 (12.63)
  Sleep Problems Index I Score: Week 36: number analyzed (Participants) | 6 | 7
  Sleep Problems Index I Score: Week 36 | 28.3 (9.83) | 26.2 (11.45)
  Sleep Problems Index I Score: Week 40: number analyzed (Participants) | 17 | 26
  Sleep Problems Index I Score: Week 40 | 30.8 (11.15) | 34.4 (14.78)
  Sleep Problems Index I Score: Week 44: number analyzed (Participants) | 7 | 9
  Sleep Problems Index I Score: Week 44 | 29.5 (11.93) | 30.7 (14.32)
  Sleep Problems Index I Score: Week 48: number analyzed (Participants) | 17 | 24
  Sleep Problems Index I Score: Week 48 | 31.6 (10.74) | 31.0 (12.83)
  Sleep Problems Index I Score: Week 52: number analyzed (Participants) | 15 | 23
  Sleep Problems Index I Score: Week 52 | 30.2 (9.13) | 32.0 (13.62)
  Sleep Problems Index II Score: Baseline | 35.5 (13.20) | 34.4 (14.17)
  Sleep Problems Index II Score: Week 4: number analyzed (Participants) | 30 | 51
  Sleep Problems Index II Score: Week 4 | 32.8 (12.00) | 32.1 (11.57)
  Sleep Problems Index II Score: Week 8: number analyzed (Participants) | 25 | 44
  Sleep Problems Index II Score: Week 8 | 30.3 (10.27) | 32.4 (13.36)
  Sleep Problems Index II Score: Week 12: number analyzed (Participants) | 20 | 40
  Sleep Problems Index II Score: Week 12 | 30.5 (12.70) | 32.8 (13.47)
  Sleep Problems Index II Score: Week 16: number analyzed (Participants) | 19 | 37
  Sleep Problems Index II Score: Week 16 | 31.2 (12.90) | 32.7 (11.83)
  Sleep Problems Index II Score: Week 20: number analyzed (Participants) | 8 | 13
  Sleep Problems Index II Score: Week 20 | 33.2 (12.21) | 31.1 (11.85)
  Sleep Problems Index II Score: Week 24: number analyzed (Participants) | 17 | 31
  Sleep Problems Index II Score: Week 24 | 29.6 (11.67) | 35.4 (14.29)
  Sleep Problems Index II Score: Week 28: number analyzed (Participants) | 7 | 9
  Sleep Problems Index II Score: Week 28 | 36.9 (12.41) | 30.9 (11.08)
  Sleep Problems Index II Score: Week 32: number analyzed (Participants) | 16 | 27
  Sleep Problems Index II Score: Week 32 | 30.9 (8.47) | 31.5 (11.36)
  Sleep Problems Index II Score: Week 36: number analyzed (Participants) | 6 | 7
  Sleep Problems Index II Score: Week 36 | 27.9 (8.99) | 27.5 (8.80)
  Sleep Problems Index II Score: Week 40: number analyzed (Participants) | 17 | 26
  Sleep Problems Index II Score: Week 40 | 31.3 (10.00) | 34.3 (14.03)
  Sleep Problems Index II Score: Week 44: number analyzed (Participants) | 7 | 9
  Sleep Problems Index II Score: Week 44 | 28.1 (9.82) | 33.8 (14.04)
  Sleep Problems Index II Score: Week 48: number analyzed (Participants) | 17 | 24
  Sleep Problems Index II Score: Week 48 | 31.4 (9.57) | 31.6 (12.65)
  Sleep Problems Index II Score: Week 52: number analyzed (Participants) | 15 | 23
  Sleep Problems Index II Score: Week 52 | 30.6 (8.85) | 32.4 (12.20)

47. Secondary Outcome: European Quality of Life-5 Dimension 5-Level (EQ-5D-5L) Index Score in Participants Greater Than or Equal to (>=) 18 Years of Age: OL Run-in Period
Description: EQ-5D-5L: standardized participant completed questionnaire consisted of 2 components: a health state profile/a single utility index value and an optional VAS. EQ-5D health state profile/a single utility index value had 5 dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3= moderate problems, 4= severe problems and 5= extreme problems. Responses to 5 dimensions comprised a health state/a single utility index value. E.g. if a participant responded "no problems" for each 5 dimensions, then health state was coded as "11111" with a predefined index value to it. Every health state (coded as combination of responses on each of 5 dimensions) had a unique predefined utility index value assigned to it, by EuroQol. US value sets (with all possible health states) was used for adults in the study and total scores ranged from 1 to -0.109. Higher (positive) scores = better health state.
Time Frame: Baseline (the last observation up to and including Day 1 of OL period), Weeks 2, 4, 6 and 8
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crisaborole 2% BID
Number analyzed (Participants) | 169
Units on a scale
  Baseline: number analyzed (Participants) | 166
  Baseline | 0.9 (0.12)
  Week 2: number analyzed (Participants) | 168
  Week 2 | 0.9 (0.13)
  Week 4 | 0.9 (0.11)
  Week 6 | 0.9 (0.12)
  Week 8 | 0.9 (0.11)

48. Secondary Outcome: European Quality of Life-5 Dimension Youth (EuroQoL EQ-5D Y) Index Score in Participants Between 8-17 Years of Age: OL Run-in Period
Description: EQ-5D-Y: child-friendly version of EQ-5D questionnaire related to health status. Health state profile assessed health in 5 dimensions (mobility; looking after myself; doing usual activities; having pain or discomfort; feeling worried, sad or unhappy) used to obtain an index score, each of which had three levels of response (no problems/no pain/not worried, some problems/some pain/a bit worried, a lot of problems/a lot of pain/very worried). Participants indicated their health state by choosing the appropriate level from each dimension. The 5 digit health states thus obtained for each dimension were then converted into a single median index value. A health state index score was calculated from individual health profiles using a USA scoring algorithm. Health state index scores generally ranged from -0.109 to 1, where,-0.109= the worst health status, 1= full health. Higher the score the better the health status. A positive change from baseline indicated improvement in health status.
Time Frame: Baseline (the last observation up to and including Day 1 of OL period), Weeks 2, 4, 6 and 8
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crisaborole 2% BID
Number analyzed (Participants) | 169
Units on a scale
  Baseline: number analyzed (Participants) | 164
  Baseline | 0.9 (0.13)
  Week 2: number analyzed (Participants) | 168
  Week 2 | 0.9 (0.11)
  Week 4 | 0.9 (0.12)
  Week 6 | 0.9 (0.11)
  Week 8 | 0.9 (0.15)

49. Secondary Outcome: EuroQoL EQ-5D Y Proxy Index Scores in Participants Between 2-7 Years of Age: OL Run-in Period
Description: EQ-5D-Y:child-friendly version of EQ-5D questionnaire related to health status.Health state profile assessed health in 5 dimensions(Mobility;Looking After Myself;Doing Usual Activities;Having Pain or Discomfort;Feeling Worried,Sad or Unhappy)used to obtain index score,each of which had three levels of response(no problems/no pain/not worried,some problems/some pain/a bit worried,a lot of problems/a lot of pain/very worried).Participants indicated health state by choosing appropriate level from each dimension.5-digit health states obtained for each dimension were converted into single median index value using index value calculator,recommended by EuroQoL group.Health state index score calculated from individual health profiles using USA scoring algorithm. Scores ranged from -0.109 to 1,where, -0.109=worst health status, 1=full health. Higher score=better health status.Positive change from baseline indicated improvement in health status.Proxy version filled by care-giver of participant
Time Frame: Baseline (the last observation up to and including Day 1 of OL period), Weeks 2, 4, 6 and 8
Population: Eval-OL population included all participants that received at least 1 dose of study intervention in the OL period. Here, ''Overall Number of Participants Analyzed'' signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crisaborole 2% BID
Number analyzed (Participants) | 136
Units on a scale
  Baseline | 0.8 (0.17) [lower limit 0.17]
  Week 2 | 0.9 (0.16) [lower limit 0.16]
  Week 4 | 0.9 (0.17) [lower limit 0.17]
  Week 6 | 0.9 (0.17) [lower limit 0.17]
  Week 8 | 0.9 (0.18) [lower limit 0.18]

50. Secondary Outcome: EuroQoL EQ-5D-5L Visual Analog Scale (VAS) Score in Participants >= 18 Years of Age: OL Run-in Period
Description: EQ-5D-5L VAS was used to record participant's rating for current health-related quality of life state on vertical VAS (0-100);0=worst imaginable health state;100=best imaginable health state.
Time Frame: Baseline (the last observation up to and including Day 1 of OL period), Weeks 2, 4, 6 and 8
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crisaborole 2% BID
Number analyzed (Participants) | 169
Units on a scale
  Baseline: number analyzed (Participants) | 166
  Baseline | 81.2 (15.81)
  Week 2: number analyzed (Participants) | 168
  Week 2 | 82.2 (16.14)
  Week 4 | 82.0 (15.73)
  Week 6 | 84.0 (14.89)
  Week 8 | 84.2 (14.18)

51. Secondary Outcome: EuroQoL EQ-5D Y VAS Scores in Participants Between 8-17 Years of Age : OL-Run-in Period
Description: EQ-5D Y VAS was used to record participant's rating for his/her current health-related quality of life state on vertical VAS (0-100);0 = worst imaginable health state and 100 = best imaginable health state.
Time Frame: Baseline (the last observation up to and including Day 1 of OL period), Weeks 2, 4, 6 and 8
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crisaborole 2% BID
Number analyzed (Participants) | 169
Units on a scale
  Baseline: number analyzed (Participants) | 164
  Baseline | 85.6 (16.27)
  Week 2: number analyzed (Participants) | 168
  Week 2 | 87.4 (11.91)
  Week 4 | 87.5 (12.92)
  Week 6 | 87.9 (12.72)
  Week 8 | 88.0 (12.93)

52. Secondary Outcome: EuroQoL EQ-5D Y Proxy VAS Scores in Participants Between 2-7 Years of Age: OL Run-in Period
Description: EQ-5D Y proxy VAS assessed the caregiver's impression of participants health state on a vertical VAS (range: 0 to 100), where, 0 (the worst imaginable health) to 100 (the best imaginable health).
Time Frame: Baseline (the last observation up to and including Day 1 of OL period), Weeks 2, 4, 6 and 8
Population: as for outcome 49
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crisaborole 2% BID
Number analyzed (Participants) | 136
Units on a scale
  Baseline | 86.0 (13.97) [lower limit 13.97]
  Week 2 | 87.6 (12.61) [lower limit 12.61]
  Week 4 | 90.0 (11.05) [lower limit 11.05]
  Week 6 | 90.4 (11.45) [lower limit 11.45]
  Week 8 | 90.8 (11.63) [lower limit 11.63]

53. Secondary Outcome: EuroQoL EQ-5D-5L Index Scores in Participants >= 18 Years of Age: DB Period
Description: as for outcome 47
Time Frame: as for outcome 32
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD | Crisaborole 2% BID: Flare Period
Number analyzed (Participants) | 46 | 48 | 35
Units on a scale
  Baseline: number analyzed (Participants) | 46 | 48 | 0
  Baseline | 0.9 (0.09) | 0.9 (0.11) |
  Week 4: number analyzed (Participants) | 23 | 30 | 35
  Week 4 | 0.9 (0.12) | 0.9 (0.10) | 0.9 (0.14)
  Week 8: number analyzed (Participants) | 25 | 31 | 28
  Week 8 | 0.9 (0.09) | 0.9 (0.10) | 0.9 (0.17)
  Week 12: number analyzed (Participants) | 23 | 28 | 24
  Week 12 | 0.9 (0.10) | 0.9 (0.18) | 0.9 (0.09)
  Week 16: number analyzed (Participants) | 31 | 33 | 13
  Week 16 | 0.9 (0.11) | 0.9 (0.15) | 0.9 (0.08)
  Week 20: number analyzed (Participants) | 15 | 13 | 6
  Week 20 | 0.9 (0.12) | 0.9 (0.15) | 0.9 (0.09)
  Week 24: number analyzed (Participants) | 26 | 30 | 8
  Week 24 | 0.9 (0.10) | 0.9 (0.21) | 0.9 (0.07)
  Week 28: number analyzed (Participants) | 12 | 11 | 5
  Week 28 | 0.9 (0.18) | 0.9 (0.14) | 1.0 (0.06)
  Week 32: number analyzed (Participants) | 23 | 27 | 5
  Week 32 | 0.9 (0.11) | 0.8 (0.22) | 0.9 (0.10)
  Week 36: number analyzed (Participants) | 11 | 11 | 4
  Week 36 | 0.9 (0.09) | 0.9 (0.13) | 1.0 (0.09)
  Week 40: number analyzed (Participants) | 23 | 28 | 5
  Week 40 | 0.9 (0.10) | 0.8 (0.24) | 1.0 (0.06)
  Week 44: number analyzed (Participants) | 12 | 11 | 6
  Week 44 | 0.9 (0.18) | 0.9 (0.14) | 1.0 (0.07)
  Week 48: number analyzed (Participants) | 22 | 24 | 7
  Week 48 | 0.9 (0.11) | 0.8 (0.23) | 1.0 (0.06)
  Week 52: number analyzed (Participants) | 25 | 23 | 7
  Week 52 | 0.9 (0.10) | 0.8 (0.24) | 0.9 (0.07)

54. Secondary Outcome: EuroQoL EQ-5D Y Index Scores in Participants Between 8-17 Years of Age: DB Period
Description: as for outcome 48
Time Frame: as for outcome 32
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD | Crisaborole 2% BID: Flare Period
Number analyzed (Participants) | 38 | 43 | 29
Units on a scale
  Baseline: number analyzed (Participants) | 38 | 43 | 0
  Baseline | 0.9 (0.08) | 0.9 (0.18) |
  Week 4: number analyzed (Participants) | 15 | 28 | 29
  Week 4 | 1.0 (0.07) | 1.0 (0.07) | 0.9 (0.21)
  Week 8: number analyzed (Participants) | 18 | 27 | 19
  Week 8 | 1.0 (0.07) | 1.0 (0.08) | 0.9 (0.10)
  Week 12: number analyzed (Participants) | 19 | 28 | 17
  Week 12 | 1.0 (0.06) | 1.0 (0.07) | 0.9 (0.10)
  Week 16: number analyzed (Participants) | 21 | 28 | 14
  Week 16 | 1.0 (0.08) | 1.0 (0.07) | 0.9 (0.09)
  Week 20: number analyzed (Participants) | 9 | 13 | 9
  Week 20 | 0.9 (0.09) | 1.0 (0.05) | 0.9 (0.09)
  Week 24: number analyzed (Participants) | 19 | 28 | 10
  Week 24 | 1.0 (0.07) | 1.0 (0.06) | 0.9 (0.12)
  Week 28: number analyzed (Participants) | 10 | 14 | 10
  Week 28 | 0.9 (0.09) | 0.9 (0.08) | 0.9 (0.14)
  Week 32: number analyzed (Participants) | 20 | 28 | 12
  Week 32 | 1.0 (0.06) | 1.0 (0.06) | 0.9 (0.11)
  Week 36: number analyzed (Participants) | 10 | 11 | 6
  Week 36 | 1.0 (0.08) | 1.0 (0.08) | 0.9 (0.09)
  Week 40: number analyzed (Participants) | 17 | 24 | 10
  Week 40 | 1.0 (0.07) | 0.9 (0.13) | 1.0 (0.08)
  Week 44: number analyzed (Participants) | 10 | 11 | 8
  Week 44 | 1.0 (0.08) | 0.9 (0.22) | 0.9 (0.09)
  Week 48: number analyzed (Participants) | 15 | 26 | 9
  Week 48 | 1.0 (0.07) | 0.9 (0.09) | 0.9 (0.09)
  Week 52: number analyzed (Participants) | 18 | 25 | 12
  Week 52 | 1.0 (0.07) | 1.0 (0.07) | 1.0 (0.08)

55. Secondary Outcome: EuroQoL EQ-5D Y Proxy Index Scores in Participants Between 2-7 Years of Age: DB Period
Description: as for outcome 49
Time Frame: as for outcome 32
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD | Crisaborole 2% BID: Flare Period
Number analyzed (Participants) | 41 | 30 | 34
Units on a scale
  Baseline: number analyzed (Participants) | 41 | 30 | 0
  Baseline | 1.0 (0.08) | 0.9 (0.12) |
  Week 4: number analyzed (Participants) | 17 | 14 | 34
  Week 4 | 0.9 (0.09) | 0.9 (0.14) | 0.8 (0.19)
  Week 8: number analyzed (Participants) | 22 | 14 | 25
  Week 8 | 0.9 (0.09) | 0.9 (0.09) | 0.8 (0.15)
  Week 12: number analyzed (Participants) | 18 | 17 | 22
  Week 12 | 1.0 (0.07) | 0.9 (0.13) | 0.8 (0.18)
  Week 16: number analyzed (Participants) | 16 | 17 | 19
  Week 16 | 1.0 (0.09) | 1.0 (0.07) | 0.9 (0.11)
  Week 20: number analyzed (Participants) | 13 | 10 | 12
  Week 20 | 0.9 (0.10) | 0.9 (0.15) | 0.8 (0.12)
  Week 24: number analyzed (Participants) | 20 | 15 | 15
  Week 24 | 1.0 (0.08) | 1.0 (0.07) | 0.9 (0.20)
  Week 28: number analyzed (Participants) | 13 | 9 | 12
  Week 28 | 0.9 (0.09) | 0.9 (0.09) | 0.9 (0.09)
  Week 32: number analyzed (Participants) | 17 | 11 | 14
  Week 32 | 1.0 (0.06) | 1.0 (0.07) | 0.9 (0.11)
  Week 36: number analyzed (Participants) | 10 | 8 | 12
  Week 36 | 1.0 (0.05) | 0.9 (0.10) | 0.9 (0.11)
  Week 40: number analyzed (Participants) | 15 | 9 | 15
  Week 40 | 0.9 (0.09) | 0.9 (0.08) | 0.9 (0.12)
  Week 44: number analyzed (Participants) | 10 | 6 | 6
  Week 44 | 1.0 (0.07) | 0.9 (0.10) | 0.9 (0.14)
  Week 48: number analyzed (Participants) | 16 | 12 | 11
  Week 48 | 1.0 (0.07) | 1.0 (0.07) | 0.9 (0.11)
  Week 52: number analyzed (Participants) | 19 | 13 | 8
  Week 52 | 1.0 (0.05) | 1.0 (0.00) | 0.9 (0.11)

56. Secondary Outcome: EuroQoL EQ-5D-5L VAS Scores in Participants >= 18 Years of Age: DB Period
Description: EQ-5D-5L VAS to record participant's rating for current health-related quality of life state on vertical VAS (0-100);0=worst imaginable health state;100=best imaginable health state.
Time Frame: as for outcome 32
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD | Crisaborole 2% BID: Flare Period
Number analyzed (Participants) | 46 | 48 | 35
Units on a scale
  Baseline: number analyzed (Participants) | 46 | 48 | 0
  Baseline | 88.3 (9.41) | 85.2 (15.56) |
  Week 4: number analyzed (Participants) | 23 | 30 | 35
  Week 4 | 89.9 (9.00) | 86.8 (10.74) | 81.9 (16.81)
  Week 8: number analyzed (Participants) | 25 | 31 | 28
  Week 8 | 90.7 (7.76) | 87.3 (12.02) | 83.8 (17.75)
  Week 12: number analyzed (Participants) | 23 | 28 | 24
  Week 12 | 88.5 (13.72) | 80.5 (21.68) | 88.1 (8.69)
  Week 16: number analyzed (Participants) | 31 | 33 | 13
  Week 16 | 88.1 (11.86) | 82.7 (18.94) | 88.7 (9.00)
  Week 20: number analyzed (Participants) | 15 | 13 | 6
  Week 20 | 87.1 (13.77) | 82.7 (14.47) | 85.3 (6.56)
  Week 24: number analyzed (Participants) | 26 | 30 | 8
  Week 24 | 89.2 (10.98) | 83.1 (19.39) | 88.0 (8.93)
  Week 28: number analyzed (Participants) | 12 | 11 | 5
  Week 28 | 88.3 (9.29) | 83.7 (16.57) | 81.2 (7.26)
  Week 32: number analyzed (Participants) | 23 | 27 | 5
  Week 32 | 90.0 (8.91) | 83.0 (20.02) | 83.2 (13.37)
  Week 36: number analyzed (Participants) | 11 | 11 | 4
  Week 36 | 90.8 (8.68) | 83.4 (12.80) | 86.8 (8.30)
  Week 40: number analyzed (Participants) | 23 | 28 | 5
  Week 40 | 88.9 (12.99) | 82.4 (20.68) | 93.8 (5.76)
  Week 44: number analyzed (Participants) | 12 | 11 | 6
  Week 44 | 87.2 (13.64) | 81.9 (13.96) | 87.0 (10.26)
  Week 48: number analyzed (Participants) | 22 | 24 | 7
  Week 48 | 88.8 (12.90) | 85.1 (20.92) | 86.9 (11.13)
  Week 52: number analyzed (Participants) | 25 | 23 | 7
  Week 52 | 90.0 (11.44) | 82.7 (20.98) | 83.7 (10.55)

57. Secondary Outcome: EuroQoL EQ-5D Y VAS Scores in Participants Between 8-17 Years of Age: DB Period
Description: EQ-5D Y VAS was a child-friendly version of EQ-5D questionnaire related to health status used to record participant's rating for his/her current health-related quality of life state on vertical VAS (0-100);0 = worst imaginable health state and 100 = best imaginable health state.
Time Frame: Baseline (the last observation up to and including Day 1 of OL period), Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD | Crisaborole 2% BID: Flare Period
Number analyzed (Participants) | 38 | 43 | 29
Units on a scale
  Baseline: number analyzed (Participants) | 38 | 43 | 0
  Baseline | 86.8 (14.86) | 91.1 (9.34) |
  Week 4: number analyzed (Participants) | 15 | 28 | 29
  Week 4 | 88.3 (11.29) | 91.6 (7.27) | 84.7 (14.13)
  Week 8: number analyzed (Participants) | 18 | 27 | 19
  Week 8 | 89.6 (9.52) | 88.6 (14.34) | 89.6 (8.36)
  Week 12: number analyzed (Participants) | 19 | 28 | 17
  Week 12 | 91.9 (9.18) | 89.1 (13.36) | 87.9 (13.50)
  Week 16: number analyzed (Participants) | 21 | 28 | 14
  Week 16 | 91.3 (8.20) | 88.9 (13.91) | 87.6 (9.87)
  Week 20: number analyzed (Participants) | 9 | 13 | 9
  Week 20 | 85.1 (10.89) | 87.8 (21.65) | 90.1 (9.43)
  Week 24: number analyzed (Participants) | 19 | 28 | 10
  Week 24 | 91.7 (10.92) | 89.3 (12.83) | 88.0 (11.94)
  Week 28: number analyzed (Participants) | 10 | 14 | 10
  Week 28 | 89.9 (12.09) | 90.4 (13.36) | 84.8 (12.56)
  Week 32: number analyzed (Participants) | 20 | 28 | 12
  Week 32 | 91.1 (9.40) | 91.5 (12.98) | 88.7 (9.89)
  Week 36: number analyzed (Participants) | 10 | 11 | 6
  Week 36 | 90.7 (10.34) | 91.7 (14.86) | 88.5 (10.88)
  Week 40: number analyzed (Participants) | 17 | 24 | 10
  Week 40 | 92.2 (9.03) | 89.8 (13.25) | 90.6 (10.02)
  Week 44: number analyzed (Participants) | 10 | 11 | 8
  Week 44 | 93.5 (8.70) | 88.3 (15.81) | 88.0 (11.16)
  Week 48: number analyzed (Participants) | 15 | 26 | 9
  Week 48 | 92.1 (9.75) | 91.3 (13.64) | 96.1 (5.18)
  Week 52: number analyzed (Participants) | 18 | 25 | 12
  Week 52 | 90.9 (13.75) | 92.6 (11.27) | 93.6 (7.91)

58. Secondary Outcome: EuroQoL EQ-5D Y Proxy VAS Scores in Participants Between 2-7 Years of Age: DB Period
Description: as for outcome 52
Time Frame: as for outcome 44
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD | Crisaborole 2% BID: Flare Period
Number analyzed (Participants) | 41 | 30 | 34
Units on a scale
  Baseline: number analyzed (Participants) | 41 | 30 | 0
  Baseline | 93.8 (9.97) | 94.3 (8.16) |
  Week 4: number analyzed (Participants) | 17 | 14 | 34
  Week 4 | 94.6 (5.86) | 96.3 (6.54) | 89.4 (11.28)
  Week 8: number analyzed (Participants) | 22 | 14 | 25
  Week 8 | 93.0 (7.39) | 96.3 (6.17) | 91.8 (7.49)
  Week 12: number analyzed (Participants) | 18 | 17 | 22
  Week 12 | 95.2 (5.47) | 96.8 (3.73) | 91.5 (10.81)
  Week 16: number analyzed (Participants) | 16 | 17 | 19
  Week 16 | 92.9 (7.08) | 96.5 (2.81) | 93.2 (6.29)
  Week 20: number analyzed (Participants) | 13 | 10 | 12
  Week 20 | 94.9 (5.09) | 93.4 (6.50) | 92.7 (5.07)
  Week 24: number analyzed (Participants) | 20 | 15 | 15
  Week 24 | 95.1 (5.62) | 95.7 (4.62) | 91.9 (7.77)
  Week 28: number analyzed (Participants) | 13 | 9 | 12
  Week 28 | 95.8 (5.60) | 97.1 (4.17) | 93.2 (5.65)
  Week 32: number analyzed (Participants) | 17 | 11 | 14
  Week 32 | 95.5 (5.70) | 96.9 (2.12) | 93.1 (6.98)
  Week 36: number analyzed (Participants) | 10 | 8 | 12
  Week 36 | 97.4 (2.99) | 97.8 (2.49) | 93.5 (5.71)
  Week 40: number analyzed (Participants) | 15 | 9 | 15
  Week 40 | 93.7 (7.76) | 96.8 (3.46) | 92.9 (5.28)
  Week 44: number analyzed (Participants) | 10 | 6 | 6
  Week 44 | 96.6 (4.60) | 97.8 (2.71) | 93.0 (5.14)
  Week 48: number analyzed (Participants) | 16 | 12 | 11
  Week 48 | 96.1 (5.15) | 96.9 (4.01) | 93.4 (5.57)
  Week 52: number analyzed (Participants) | 19 | 13 | 8
  Week 52 | 95.0 (5.51) | 96.7 (3.97) | 96.6 (3.11)

59. Secondary Outcome: EuroQoL EQ-5D-5L Index Scores in Participants >= 18 Years of Age: First Flare Period
Description: as for outcome 47
Time Frame: Weeks 0, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 27 | 28
Units on a scale
  Week 0 | 0.9 (0.11) | 0.9 (0.15)
  Week 4: number analyzed (Participants) | 14 | 15
  Week 4 | 1.0 (0.07) | 0.8 (0.19)
  Week 8: number analyzed (Participants) | 9 | 10
  Week 8 | 1.0 (0.06) | 0.8 (0.07)
  Week 12: number analyzed (Participants) | 3 | 3
  Week 12 | 0.9 (0.10) | 0.9 (0.10)

60. Secondary Outcome: EuroQoL EQ-5D Y Index Scores in Participants Between 8-17 Years of Age: First Flare Period
Description: as for outcome 48
Time Frame: Weeks 0, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 28 | 22
Units on a scale
  Week 0 | 0.9 (0.09) | 0.8 (0.25)
  Week 4: number analyzed (Participants) | 14 | 13
  Week 4 | 0.9 (0.09) | 0.9 (0.13)
  Week 8: number analyzed (Participants) | 9 | 9
  Week 8 | 0.9 (0.10) | 0.9 (0.11)
  Week 12: number analyzed (Participants) | 1 | 5
  Week 12 | 1.0 (NA) — Standard deviation could not be estimated due to less number of participants with events. | 0.9 (0.09)

61. Secondary Outcome: EuroQoL EQ-5D Y Proxy Index Scores in Participants Between 2-7 Years of Age: First Flare Period
Description: as for outcome 49
Time Frame: Weeks 0, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 30 | 23
Units on a scale
  Week 0 | 0.8 (0.22) | 0.8 (0.15)
  Week 4: number analyzed (Participants) | 19 | 15
  Week 4 | 0.9 (0.18) | 0.9 (0.16)
  Week 8: number analyzed (Participants) | 12 | 6
  Week 8 | 0.9 (0.11) | 0.8 (0.20)
  Week 12: number analyzed (Participants) | 4 | 1
  Week 12 | 0.9 (0.10) | 1.0 (NA) — Standard deviation could not be estimated due to less number of participants with events.

62. Secondary Outcome: EuroQoL EQ-5D-5L VAS Scores in Participants >= 18 Years of Age: First Flare Period
Description: EQ-5D-5L VAS was used to record participant's rating for his/her current health-related quality of life state on a vertical VAS (0-100), where 0 = worst imaginable health state and 100 = best imaginable health state.
Time Frame: Weeks 0, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 27 | 28
Units on a scale
  Week 0 | 84.1 (10.40) | 82.8 (17.81)
  Week 4: number analyzed (Participants) | 14 | 15
  Week 4 | 87.9 (8.02) | 81.1 (22.15)
  Week 8: number analyzed (Participants) | 9 | 10
  Week 8 | 88.6 (6.71) | 88.2 (9.25)
  Week 12: number analyzed (Participants) | 3 | 3
  Week 12 | 83.7 (11.85) | 85.0 (21.79)

63. Secondary Outcome: EuroQoL EQ-5D Y VAS Scores in Participants Between 8-17 Years of Age: First Flare Period
Description: as for outcome 57
Time Frame: Weeks 0, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 28 | 22
Units on a scale
  Baseline | 86.5 (10.87) | 88.7 (10.27)
  Week 4: number analyzed (Participants) | 14 | 13
  Week 4 | 91.5 (8.91) | 82.3 (18.55)
  Week 8: number analyzed (Participants) | 9 | 9
  Week 8 | 85.3 (17.58) | 87.0 (9.49)
  Week 12: number analyzed (Participants) | 1 | 5
  Week 12 | 100.0 (NA) — Standard deviation could not be estimated due to less number of participants with events. | 81.0 (4.18)

64. Secondary Outcome: EuroQoL EQ-5D Y Proxy VAS Scores in Participants Between 2-7 Years of Age: First Flare Period
Description: as for outcome 52
Time Frame: Weeks 0, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 30 | 23
Units on a scale
  Week 0 | 84.7 (21.55) | 91.0 (7.84)
  Week 4: number analyzed (Participants) | 19 | 15
  Week 4 | 90.3 (13.53) | 91.3 (7.69)
  Week 8: number analyzed (Participants) | 12 | 6
  Week 8 | 93.8 (5.29) | 93.0 (7.90)
  Week 12: number analyzed (Participants) | 4 | 1
  Week 12 | 90.0 (10.61) | 99.0 (NA) — Standard deviation could not be estimated due to less number of participants with events.

65. Secondary Outcome: EuroQoL EQ-5D Y Index Scores in Participants >= 18 Years of Age: First Flare Free Period
Description: as for outcome 48
Time Frame: Baseline (the last observation up to and including randomization day), Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 46 | 48
Units on a scale
  Baseline | 0.9 (0.09) | 0.9 (0.11)
  Week 4: number analyzed (Participants) | 22 | 30
  Week 4 | 0.9 (0.12) | 0.9 (0.10)
  Week 8: number analyzed (Participants) | 20 | 26
  Week 8 | 0.9 (0.10) | 0.9 (0.09)
  Week 12: number analyzed (Participants) | 15 | 21
  Week 12 | 1.0 (0.09) | 0.9 (0.09)
  Week 16: number analyzed (Participants) | 15 | 19
  Week 16 | 0.9 (0.11) | 0.9 (0.10)
  Week 20: number analyzed (Participants) | 7 | 6
  Week 20 | 0.9 (0.09) | 0.9 (0.15)
  Week 24: number analyzed (Participants) | 14 | 17
  Week 24 | 0.9 (0.10) | 0.9 (0.10)
  Week 28: number analyzed (Participants) | 7 | 4
  Week 28 | 1.0 (0.07) | 1.0 (0.00)
  Week 32: number analyzed (Participants) | 13 | 13
  Week 32 | 0.9 (0.10) | 0.9 (0.12)
  Week 36: number analyzed (Participants) | 6 | 3
  Week 36 | 0.9 (0.08) | 1.0 (0.00)
  Week 40: number analyzed (Participants) | 14 | 13
  Week 40 | 1.0 (0.08) | 0.9 (0.18)
  Week 44: number analyzed (Participants) | 7 | 4
  Week 44 | 1.0 (0.07) | 1.0 (0.07)
  Week 48: number analyzed (Participants) | 14 | 12
  Week 48 | 0.9 (0.11) | 0.9 (0.11)
  Week 52: number analyzed (Participants) | 13 | 12
  Week 52 | 0.9 (0.10) | 0.9 (0.12)

66. Secondary Outcome: EuroQoL EQ-5D Y Index Scores in Participants Between 8-17 Years of Age: First Flare Free Period
Description: as for outcome 48
Time Frame: Baseline (the last observation up to and including randomization day of DB period), Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 38 | 43
Units on a scale
  Baseline | 0.9 (0.08) | 0.9 (0.18)
  Week 4: number analyzed (Participants) | 13 | 28
  Week 4 | 1.0 (0.06) | 1.0 (0.07)
  Week 8: number analyzed (Participants) | 9 | 24
  Week 8 | 1.0 (0.05) | 1.0 (0.08)
  Week 12: number analyzed (Participants) | 10 | 25
  Week 12 | 1.0 (0.07) | 1.0 (0.06)
  Week 16: number analyzed (Participants) | 7 | 24
  Week 16 | 1.0 (0.07) | 1.0 (0.07)
  Week 20: number analyzed (Participants) | 2 | 11
  Week 20 | 0.8 (0.01) | 1.0 (0.05)
  Week 24: number analyzed (Participants) | 6 | 20
  Week 24 | 1.0 (0.07) | 1.0 (0.06)
  Week 28: number analyzed (Participants) | 1 | 9
  Week 28 | 1.0 (NA) — Standard deviation could not be estimated due to less number of participants with events. | 1.0 (0.07)
  Week 32: number analyzed (Participants) | 7 | 19
  Week 32 | 1.0 (0.07) | 1.0 (0.07)
  Week 36: number analyzed (Participants) | 0 | 7
  Week 36 |  | 1.0 (0.08)
  Week 40: number analyzed (Participants) | 6 | 17
  Week 40 | 0.9 (0.09) | 0.9 (0.14)
  Week 44: number analyzed (Participants) | 0 | 8
  Week 44 |  | 0.9 (0.25)
  Week 48: number analyzed (Participants) | 5 | 16
  Week 48 | 1.0 (0.08) | 0.9 (0.09)
  Week 52: number analyzed (Participants) | 4 | 15
  Week 52 | 1.0 (0.09) | 1.0 (0.07)

67. Secondary Outcome: EuroQoL EQ-5D Y Proxy Index Scores in Participants Between 2-7 Years of Age: First Flare Free Period
Description: as for outcome 49
Time Frame: as for outcome 66
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 41 | 30
Units on a scale
  Baseline | 1.0 (0.08) | 0.9 (0.12)
  Week 4: number analyzed (Participants) | 16 | 14
  Week 4 | 0.9 (0.10) | 0.9 (0.14)
  Week 8: number analyzed (Participants) | 11 | 10
  Week 8 | 1.0 (0.08) | 1.0 (0.08)
  Week 12: number analyzed (Participants) | 10 | 10
  Week 12 | 1.0 (0.09) | 1.0 (0.06)
  Week 16: number analyzed (Participants) | 7 | 6
  Week 16 | 0.9 (0.09) | 1.0 (0.00)
  Week 20: number analyzed (Participants) | 2 | 3
  Week 20 | 0.9 (0.12) | 1.0 (0.00)
  Week 24: number analyzed (Participants) | 4 | 6
  Week 24 | 0.9 (0.08) | 1.0 (0.00)
  Week 28: number analyzed (Participants) | 2 | 3
  Week 28 | 0.9 (0.12) | 0.9 (0.09)
  Week 32: number analyzed (Participants) | 4 | 4
  Week 32 | 0.9 (0.11) | 1.0 (0.00)
  Week 36: number analyzed (Participants) | 1 | 3
  Week 36 | 1.0 (NA) — Standard deviation could not be estimated due to less number of participants with events. | 1.0 (0.00)
  Week 40: number analyzed (Participants) | 4 | 3
  Week 40 | 0.9 (0.11) | 1.0 (0.00)
  Week 44: number analyzed (Participants) | 1 | 1
  Week 44 | 1.0 (NA) — Standard deviation could not be estimated due to less number of participants with events. | 1.0 (NA) — Standard deviation could not be estimated due to less number of participants with events.
  Week 48: number analyzed (Participants) | 4 | 3
  Week 48 | 0.9 (0.11) | 1.0 (0.00)
  Week 52: number analyzed (Participants) | 5 | 3
  Week 52 | 1.0 (0.06) | 1.0 (0.00)

68. Secondary Outcome: EuroQoL EQ-5D-5L VAS Scores in Participants >= 18 Years of Age: First Flare Free Period
Description: as for outcome 50
Time Frame: as for outcome 66
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 46 | 48
Units on a scale
  Baseline | 88.3 (9.41) | 85.2 (15.56)
  Week 4: number analyzed (Participants) | 22 | 30
  Week 4 | 89.6 (9.11) | 86.8 (10.74)
  Week 8: number analyzed (Participants) | 20 | 26
  Week 8 | 91.3 (7.44) | 88.5 (11.29)
  Week 12: number analyzed (Participants) | 15 | 21
  Week 12 | 91.9 (8.86) | 83.8 (15.36)
  Week 16: number analyzed (Participants) | 15 | 19
  Week 16 | 91.3 (9.74) | 86.1 (11.88)
  Week 20: number analyzed (Participants) | 7 | 6
  Week 20 | 88.1 (12.01) | 87.5 (14.01)
  Week 24: number analyzed (Participants) | 14 | 17
  Week 24 | 92.6 (8.26) | 88.1 (9.77)
  Week 28: number analyzed (Participants) | 7 | 4
  Week 28 | 91.9 (7.06) | 96.3 (2.75)
  Week 32: number analyzed (Participants) | 13 | 13
  Week 32 | 91.5 (6.70) | 89.5 (8.88)
  Week 36: number analyzed (Participants) | 6 | 3
  Week 36 | 91.3 (9.83) | 92.7 (10.12)
  Week 40: number analyzed (Participants) | 14 | 13
  Week 40 | 93.1 (7.95) | 87.2 (13.76)
  Week 44: number analyzed (Participants) | 7 | 4
  Week 44 | 91.1 (9.63) | 88.0 (11.78)
  Week 48: number analyzed (Participants) | 14 | 12
  Week 48 | 92.5 (9.28) | 92.4 (8.17)
  Week 52: number analyzed (Participants) | 13 | 12
  Week 52 | 93.7 (7.75) | 88.9 (9.70)

69. Secondary Outcome: EuroQoL EQ-5D Y VAS Scores in Participants Between 8-17 Years of Age: First Flare Free Period
Description: as for outcome 57
Time Frame: as for outcome 66
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 38 | 43
Units on a scale
  Baseline | 86.8 (14.86) | 91.1 (9.34)
  Week 4: number analyzed (Participants) | 13 | 28
  Week 4 | 87.7 (11.74) | 91.6 (7.27)
  Week 8: number analyzed (Participants) | 9 | 24
  Week 8 | 88.8 (10.96) | 87.6 (14.84)
  Week 12: number analyzed (Participants) | 10 | 25
  Week 12 | 89.8 (11.01) | 87.9 (13.70)
  Week 16: number analyzed (Participants) | 7 | 24
  Week 16 | 92.9 (8.01) | 87.9 (14.74)
  Week 20: number analyzed (Participants) | 2 | 11
  Week 20 | 84.0 (12.73) | 86.1 (23.22)
  Week 24: number analyzed (Participants) | 6 | 20
  Week 24 | 92.7 (12.04) | 89.8 (13.76)
  Week 28: number analyzed (Participants) | 1 | 9
  Week 28 | 96.0 (NA) — Standard deviation could not be estimated due to less number of participants with events. | 86.6 (15.40)
  Week 32: number analyzed (Participants) | 7 | 19
  Week 32 | 92.1 (8.43) | 88.8 (14.68)
  Week 36: number analyzed (Participants) | 0 | 7
  Week 36 |  | 89.0 (18.25)
  Week 40: number analyzed (Participants) | 6 | 17
  Week 40 | 95.2 (4.75) | 89.6 (14.01)
  Week 44: number analyzed (Participants) | 0 | 8
  Week 44 |  | 88.0 (16.46)
  Week 48: number analyzed (Participants) | 5 | 16
  Week 48 | 93.8 (7.50) | 89.1 (15.72)
  Week 52: number analyzed (Participants) | 4 | 15
  Week 52 | 98.5 (1.91) | 90.7 (13.53)

70. Secondary Outcome: EuroQoL EQ-5D Y Proxy VAS Scores in Participants Between 2-7 Years of Age: First Flare Free Period
Description: as for outcome 52
Time Frame: as for outcome 66
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 41 | 30
Units on a scale
  Baseline | 93.8 (9.97) | 94.3 (8.16)
  Week 4: number analyzed (Participants) | 16 | 14
  Week 4 | 94.6 (6.05) | 96.3 (6.54)
  Week 8: number analyzed (Participants) | 11 | 10
  Week 8 | 94.3 (7.06) | 96.0 (7.29)
  Week 12: number analyzed (Participants) | 10 | 10
  Week 12 | 94.4 (5.95) | 98.3 (2.26)
  Week 16: number analyzed (Participants) | 7 | 6
  Week 16 | 93.7 (8.22) | 98.2 (2.23)
  Week 20: number analyzed (Participants) | 2 | 3
  Week 20 | 96.5 (4.95) | 93.7 (10.97)
  Week 24: number analyzed (Participants) | 4 | 6
  Week 24 | 90.0 (8.49) | 95.7 (5.01)
  Week 28: number analyzed (Participants) | 2 | 3
  Week 28 | 100.0 (0.00) | 100.0 (0.00)
  Week 32: number analyzed (Participants) | 4 | 4
  Week 32 | 92.0 (8.45) | 97.8 (1.71)
  Week 36: number analyzed (Participants) | 1 | 3
  Week 36 | 100.0 (NA) — Standard deviation could not be estimated due to less number of participants with events. | 98.3 (2.89)
  Week 40: number analyzed (Participants) | 4 | 3
  Week 40 | 91.5 (9.33) | 99.3 (0.58)
  Week 44: number analyzed (Participants) | 1 | 1
  Week 44 | 100.0 (NA) — Standard deviation could not be estimated due to less number of participants with events. | 100.0 (NA) — Standard deviation could not be estimated due to less number of participants with events.
  Week 48: number analyzed (Participants) | 4 | 3
  Week 48 | 94.0 (5.35) | 99.0 (1.73)
  Week 52: number analyzed (Participants) | 5 | 3
  Week 52 | 96.4 (4.16) | 98.7 (2.31)

71. Secondary Outcome: Percent Work Time Missed Using Work Productivity and Activity Impairment (WPAI) Questionnaire Plus Classroom Impairment Questions (CIQ): OL Run-in Period
Description: WPAI plus CIQ was a 10-item questionnaire used to assess degree to which AD affected work productivity and regular activities over past 7 days. Questions were: Q1= currently employed; Q2= work hours missed due to health problems; Q3= work hours missed due to other reasons; Q4= hours actually worked; Q5= degree health affected productivity while working (0-10 scale, higher scores = less productivity); Q6= classes attended in academic setting or not; Q7= class hours missed due to health problems; Q8= class hours actually attended; Q9= degree health affected productivity while attending (0-10 scale, high scores= less productivity); Q10= degree health affected productivity in regular daily activities (0-10 scale, higher scores = less productivity). Percent work time missed was calculated as: Q2*100/(Q2+Q4) and score ranged from 0-100%, higher scores = greater impairment and less productivity.
Time Frame: Baseline (last observation up to and including Day 1 of OL period), Weeks 2, 4, 6 and 8
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Percentage of work time missed
Arm/Group | Crisaborole 2% BID
Number analyzed (Participants) | 135
Percentage of work time missed
  Baseline: number analyzed (Participants) | 125
  Baseline | 5.75 (16.796)
  Week 2: number analyzed (Participants) | 131
  Week 2 | 4.72 (15.553)
  Week 4: number analyzed (Participants) | 133
  Week 4 | 5.92 (16.487)
  Week 6: number analyzed (Participants) | 134
  Week 6 | 4.83 (14.801)
  Week 8 | 6.96 (18.080)

72. Secondary Outcome: Percent Impairment While Working Using Work Productivity and Activity Impairment (WPAI) Questionnaire Plus Classroom Impairment Questions (CIQ): OL Run-in Period
Description: WPAI+CIQ:10-item questionnaire used to assess degree to which AD affected work productivity and regular activities over past 7 days. Questions were:Q1= currently employed;Q2= work hours missed due to health problems; Q3=work hours missed due to other reasons; Q4= hours actually worked; Q5 = degree health affected productivity while working (0-10 scale, high scores=less productivity);Q6=classes attended in academic setting or not;Q7= class hours missed due to health problems; Q8= class hours actually attended; Q9= degree health affected productivity while attending(0-10 scale, high scores= less productivity); Q10= degree health affected productivity in regular daily activities (0-10 scale, high scores=less productivity). Percent impairment while working due to health problem was calculated as: 100*Q5/10 and score ranged from 0-100%,higher scores =greater impairment and less productivity.
Time Frame: Weeks 0, 2, 4, 6 and 8
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Percentage of work impairment
Arm/Group | Crisaborole 2% BID
Number analyzed (Participants) | 135
Percentage of work impairment
  Week 0: number analyzed (Participants) | 124
  Week 0 | 32.66 (28.602)
  Week 2: number analyzed (Participants) | 131
  Week 2 | 17.02 (21.293)
  Week 4: number analyzed (Participants) | 133
  Week 4 | 15.26 (20.285)
  Week 6: number analyzed (Participants) | 134
  Week 6 | 14.10 (20.417)
  Week 8 | 14.37 (20.898)

73. Secondary Outcome: Percent Overall Work Impairment Using Work Productivity and Activity Impairment (WPAI) Questionnaire Plus Classroom Impairment Questions (CIQ): OL Run-in Period
Description: WPAI+CIQ:10-item questionnaire to assess degree to which AD affected work productivity and regular activities over past 7 days.Questions:Q1=currently employed;Q2=work hours missed due to health problems;Q3=work hours missed due to other reasons;Q4=hours actually worked;Q5=degree health affected productivity while working(0-10 scale, high scores=less productivity);Q6=classes attended in academic setting or not;Q7=class hours missed due to health problems;Q8=class hours actually attended;Q9=degree health affected productivity while attending(0-10 scale, high scores= less productivity);Q10=degree health affected productivity: regular daily activities (0-10 scale, high scores =less productivity). Percent overall impairment while working due to health problem calculated as:100*{Q2/(Q2+Q4)+[(1- Q2/(Q2+Q4))×(Q5/10)]},score ranged:0-100%,high numbers=greater impairment and less productivity.
Time Frame: Weeks 0, 2, 4, 6 and 8
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Percentage of work impairment
Arm/Group | Crisaborole 2% BID
Number analyzed (Participants) | 135
Percentage of work impairment
  Week 0: number analyzed (Participants) | 124
  Week 0 | 34.77 (30.179)
  Week 2: number analyzed (Participants) | 131
  Week 2 | 20.10 (23.627)
  Week 4: number analyzed (Participants) | 133
  Week 4 | 19.30 (23.220)
  Week 6: number analyzed (Participants) | 134
  Week 6 | 17.43 (22.620)
  Week 8 | 19.36 (24.564)

74. Secondary Outcome: Percent Class Time Missed Using Work Productivity and Activity Impairment Questionnaire Plus Classroom Impairment Questions: OL Run-in Period
Description: WPAI+CIQ:10-item questionnaire to assess degree to which AD affected work productivity and regular activities over past 7 days. Questions: Q1=currently employed; Q2=work hours missed due to health problems; Q3=work hours missed due to other reasons; Q4=hours actually worked; Q5=degree health affected productivity while working (0-10 scale, high scores=less productivity); Q6=classes attended in academic setting or not; Q7=class hours missed due to health problems; Q8=class hours actually attended; Q9=degree health affected productivity while attending(0-10 scale, high scores= less productivity); Q10=degree health affected productivity in regular daily activities(0-10 scale, high scores =less productivity).Percent class time missed due to health problem calculated as: Q7*100/(Q7+Q8) and score ranged from 0-100% where higher numbers=greater impairment and less productivity.
Time Frame: Baseline (last observation up to and including Day 1 of OL period), Weeks 2, 4, 6 and 8
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Percent class time missed
Arm/Group | Crisaborole 2% BID
Number analyzed (Participants) | 118
Percent class time missed
  Baseline: number analyzed (Participants) | 83
  Baseline | 4.14 (14.982)
  Week 2: number analyzed (Participants) | 98
  Week 2 | 5.26 (16.664)
  Week 4: number analyzed (Participants) | 108
  Week 4 | 3.94 (12.968)
  Week 6: number analyzed (Participants) | 117
  Week 6 | 4.71 (13.991)
  Week 8 | 4.55 (14.584)

75. Secondary Outcome: Percent Impairment While in Class Using Work Productivity and Activity Impairment Questionnaire Plus Classroom Impairment Questions: OL Run-in Period
Description: WPAI+CIQ:10-item questionnaire used to assess degree to which AD affected work productivity and regular activities over past 7 days. Questions: Q1=currently employed; Q2=work hours missed due to health problems; Q3=work hours missed due to other reasons; Q4=hours actually worked; Q5 = degree health affected productivity while working (0-10 scale, high scores=less productivity); Q6=classes attended in academic setting or not; Q7=class hours missed due to health problems; Q8=class hours actually attended; Q9=degree health affected productivity while attending (0-10 scale, high scores= less productivity); Q10=degree health affected productivity in regular daily activities (0-10 scale, high scores =less productivity). Percent impairment while in class was calculated as: 100*Q9/10 and score ranged from 0-100% where higher numbers indicate greater impairment and less productivity.
Time Frame: Baseline (last observation up to and including Day 1 of OL period), Weeks 2, 4, 6 and 8
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Percent impairment in class
Arm/Group | Crisaborole 2% BID
Number analyzed (Participants) | 119
Percent impairment in class
  Baseline: number analyzed (Participants) | 82
  Baseline | 26.46 (22.683)
  Week 2: number analyzed (Participants) | 98
  Week 2 | 17.55 (19.639)
  Week 4: number analyzed (Participants) | 108
  Week 4 | 15.37 (19.879)
  Week 6: number analyzed (Participants) | 118
  Week 6 | 13.31 (19.527)
  Week 8 | 12.69 (17.789)

76. Secondary Outcome: Percent Overall Class Impairment Using Work Productivity and Activity Impairment Questionnaire Plus Classroom Impairment Questions: OL Run-in Period
Description: WPAI+CIQ:10-item questionnaire to assess degree to which AD affected work productivity and regular activities over past7days.Questions:Q1=currently employed;Q2=work hours missed due to health problems;Q3=work hours missed due to other reasons;Q4=hours actually worked;Q5=degree health affected productivity while working (0-10 scale, high scores=less productivity);Q6=classes attended in academic setting or not;Q7=class hours missed due to health problems;Q8=class hours actually attended;Q9=degree health affected productivity while attending(0-10 scale, high scores= less productivity);Q10=degree health affected productivity in regular daily activities(0-10 scale, high scores =less productivity).Percent overall class impairment due to health problem calculated as: 100*{Q7/(Q7+Q8)+[(1- Q7/(Q7+Q8))×(Q9/10)]},score range:0-100%,higher numbers=greater impairment and less productivity.
Time Frame: Baseline (last observation up to and including Day 1 of OL period), Weeks 2, 4, 6 and 8
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Percent overall class impairment
Arm/Group | Crisaborole 2% BID
Number analyzed (Participants) | 118
Percent overall class impairment
  Baseline: number analyzed (Participants) | 82
  Baseline | 28.20 (24.171)
  Week 2: number analyzed (Participants) | 98
  Week 2 | 20.27 (22.676)
  Week 4: number analyzed (Participants) | 108
  Week 4 | 18.13 (22.977)
  Week 6: number analyzed (Participants) | 117
  Week 6 | 17.01 (23.126)
  Week 8 | 16.20 (22.148)

77. Secondary Outcome: Percent Activity Impairment Using Work Productivity and Activity Impairment Questionnaire Plus Classroom Impairment Questions: OL Run-in Period
Description: WPAI+CIQ: 10-item questionnaire used to assess degree to which AD affected work productivity and regular activities over past 7 days. Questions:Q1=currently employed;Q2=work hours missed due to health problems; Q3=work hours missed due to other reasons; Q4=hours actually worked; Q5=degree health affected productivity while working (0-10 scale, high scores=less productivity); Q6=classes attended in academic setting or not; Q7=class hours missed due to health problems; Q8=class hours actually attended; Q9=degree health affected productivity while attending(0-10 scale, high scores= less productivity); Q10=degree health affected productivity in regular daily activities(0-10 scale, high scores =less productivity). Percent activity impairment due to health problem calculated as: 100*Q10/10, score ranged from 0-100%,higher numbers=greater impairment and less productivity.
Time Frame: Baseline (last observation up to and including Day 1 of OL period), Weeks 2, 4, 6 and 8
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Percent activity impairment
Arm/Group | Crisaborole 2% BID
Number analyzed (Participants) | 273
Percent activity impairment
  Baseline: number analyzed (Participants) | 268
  Baseline | 28.21 (28.766)
  Week 2: number analyzed (Participants) | 271
  Week 2 | 15.83 (20.036)
  Week 4 | 14.54 (20.162)
  Week 6 | 13.81 (20.547)
  Week 8 | 13.55 (19.783)

78. Secondary Outcome: Percent Work Time Missed Using Work Productivity and Activity Impairment Questionnaire Plus Classroom Impairment Questions: DB Period
Description: WPAI+CIQ:10-item questionnaire used to assess degree to which AD affected work productivity and regular activities over past 7 days. Questions were: Q1=currently employed; Q2=work hours missed due to health problems; Q3=work hours missed due to other reasons;Q4=hours actually worked; Q5 = degree health affected productivity while working (0-10 scale, high scores=less productivity);Q6=classes attended in academic setting or not;Q7=class hours missed due to health problems;Q8=class hours actually attended;Q9=degree health affected productivity while attending(0-10 scale, high scores = less productivity);Q10=degree health affected productivity in regular daily activities(0-10 scale, high scores=less productivity). Percent work time missed due to health problem calculated as: Q2*100/(Q2+Q4) and score ranged from 0-100%,higher numbers=greater impairment and less productivity.
Time Frame: as for outcome 65
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent work time missed
Arm/Group | Vehicle QD | Crisaborole 2% QD | Crisaborole 2% BID: Flare Period
Number analyzed (Participants) | 69 | 78 | 88
Percent work time missed
  Baseline: number analyzed (Participants) | 35 | 38 | 0
  Baseline | 4.77 (14.528) | 5.07 (14.128) |
  Week 4: number analyzed (Participants) | 11 | 18 | 23
  Week 4 | 5.67 (14.861) | 5.54 (15.120) | 2.80 (10.617)
  Week 8: number analyzed (Participants) | 13 | 17 | 16
  Week 8 | 5.48 (14.237) | 2.99 (12.345) | 1.41 (3.066)
  Week 12: number analyzed (Participants) | 13 | 15 | 9
  Week 12 | 3.98 (13.835) | 3.85 (12.970) | 6.81 (16.477)
  Week 16: number analyzed (Participants) | 18 | 21 | 8
  Week 16 | 14.84 (30.656) | 3.55 (10.903) | 6.25 (17.678)
  Week 20: number analyzed (Participants) | 8 | 6 | 5
  Week 20 | 4.34 (9.633) | 0.37 (0.898) | 10.00 (22.361)
  Week 24: number analyzed (Participants) | 15 | 18 | 5
  Week 24 | 0.37 (0.997) | 7.24 (17.750) | 18.76 (29.995)
  Week 28: number analyzed (Participants) | 5 | 5 | 4
  Week 28 | 0.36 (0.805) | 0.82 (1.834) | 4.73 (9.450)
  Week 32: number analyzed (Participants) | 13 | 18 | 3
  Week 32 | 5.55 (14.500) | 9.22 (25.636) | 18.27 (31.639)
  Week 36: number analyzed (Participants) | 5 | 5 | 4
  Week 36 | 5.00 (11.180) | 0.84 (1.878) | 3.58 (7.150)
  Week 40: number analyzed (Participants) | 15 | 18 | 3
  Week 40 | 1.91 (6.181) | 3.02 (11.770) | 0.00 (0.000)
  Week 44: number analyzed (Participants) | 6 | 6 | 4
  Week 44 | 0.27 (0.653) | 0.70 (1.715) | 2.08 (4.150)
  Week 48: number analyzed (Participants) | 12 | 15 | 6
  Week 48 | 1.44 (3.746) | 11.51 (21.033) | 5.55 (13.595)
  Week 52: number analyzed (Participants) | 15 | 16 | 3
  Week 52 | 11.27 (20.344) | 5.00 (12.884) | 0.00 (0.000)

79. Secondary Outcome: Percent Impairment While Working Using Work Productivity and Activity Impairment Questionnaire Plus Classroom Impairment Questions: DB Period
Description: WPAI+CIQ:10-item questionnaire used to assess degree to which AD affected work productivity and regular activities over past 7 days. Questions:Q1=currently employed; Q2=hours missed due to health problems; Q3=hours missed due to other reasons; Q4=hours actually worked; Q5=degree health affected productivity while working (0-10 scale, high scores=less productivity); Q6=classes attended in academic setting or not; Q7=hours missed due to health problems; Q8=hours actually attended; Q9=degree health affected productivity while attending(0-10 scale, high scores= less productivity); Q10=degree health affected productivity in regular daily activities(0-10 scale, high scores =less productivity). Percent impairment while working due to health problem calculated as: 100*Q5/10 score ranged from 0-100%,higher numbers=greater impairment and less productivity.
Time Frame: as for outcome 65
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent impairment while work
Arm/Group | Vehicle QD | Crisaborole 2% QD | Crisaborole 2% BID: Flare Period
Number analyzed (Participants) | 69 | 78 | 88
Percent impairment while work
  Baseline: number analyzed (Participants) | 35 | 38 | 0
  Baseline | 9.71 (15.432) | 10.26 (17.474) |
  Week 4: number analyzed (Participants) | 11 | 18 | 23
  Week 4 | 4.55 (12.136) | 10.56 (15.136) | 15.22 (25.561)
  Week 8: number analyzed (Participants) | 13 | 17 | 16
  Week 8 | 6.15 (7.679) | 5.29 (12.805) | 9.38 (16.520)
  Week 12: number analyzed (Participants) | 13 | 15 | 9
  Week 12 | 6.92 (8.549) | 8.00 (20.771) | 7.78 (13.017)
  Week 16: number analyzed (Participants) | 17 | 21 | 8
  Week 16 | 11.76 (15.506) | 5.24 (14.359) | 11.25 (21.002)
  Week 20: number analyzed (Participants) | 8 | 6 | 5
  Week 20 | 11.25 (15.526) | 3.33 (5.164) | 10.00 (12.247)
  Week 24: number analyzed (Participants) | 15 | 18 | 5
  Week 24 | 8.00 (8.619) | 8.89 (20.260) | 10.00 (17.321)
  Week 28: number analyzed (Participants) | 5 | 5 | 4
  Week 28 | 12.00 (13.038) | 0.00 (0.000) | 5.00 (5.774)
  Week 32: number analyzed (Participants) | 13 | 17 | 3
  Week 32 | 7.69 (8.321) | 9.41 (15.996) | 0.00 (0.000)
  Week 36: number analyzed (Participants) | 5 | 5 | 4
  Week 36 | 10.00 (10.000) | 10.00 (10.000) | 2.50 (5.000)
  Week 40: number analyzed (Participants) | 15 | 18 | 3
  Week 40 | 9.33 (10.998) | 10.56 (19.844) | 6.67 (11.547)
  Week 44: number analyzed (Participants) | 6 | 6 | 4
  Week 44 | 21.67 (32.506) | 11.67 (24.014) | 5.00 (10.000)
  Week 48: number analyzed (Participants) | 12 | 15 | 6
  Week 48 | 9.17 (9.003) | 13.33 (21.269) | 15.00 (22.583)
  Week 52: number analyzed (Participants) | 15 | 16 | 3
  Week 52 | 8.00 (9.411) | 10.63 (20.484) | 10.00 (10.000)

80. Secondary Outcome: Percent Overall Work Impairment Using Work Productivity and Activity Impairment Questionnaire Plus Classroom Impairment Questions: DB Period
Description: WPAI+CIQ:10-item questionnaire to assess degree to which AD affected work productivity and regular activities over past 7 days. Questions: Q1=currently employed;Q2=work hours missed due to health problems;Q3=work hours missed due to other reasons;Q4=hours actually worked;Q5=degree health affected productivity while working(0-10 scale, high scores=less productivity);Q6=classes attended in academic setting or not;Q7=class hours missed due to health problems;Q8=class hours actually attended;Q9=degree health affected productivity while attending(0-10 scale, high scores= less productivity);Q10=degree health affected productivity: regular daily activities(0-10 scale, high scores =less productivity). Percent overall impairment while working due to health problem calculated as:100*{Q2/(Q2+Q4)+[(1- Q2/(Q2+Q4))×(Q5/10)]}, score ranged: 0-100%, high numbers=greater impairment and less productivity.
Time Frame: as for outcome 65
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent overall work impairment
Arm/Group | Vehicle QD | Crisaborole 2% QD | Crisaborole 2% BID: Flare Period
Number analyzed (Participants) | 69 | 78 | 88
Percent overall work impairment
  Baseline: number analyzed (Participants) | 35 | 38 | 0
  Baseline | 14.04 (19.991) | 14.29 (21.183) |
  Week 4: number analyzed (Participants) | 11 | 18 | 23
  Week 4 | 10.20 (17.730) | 15.53 (20.088) | 15.80 (25.411)
  Week 8: number analyzed (Participants) | 13 | 17 | 16
  Week 8 | 11.46 (14.980) | 8.29 (16.813) | 10.73 (16.268)
  Week 12: number analyzed (Participants) | 13 | 15 | 9
  Week 12 | 10.11 (16.906) | 9.13 (23.216) | 14.04 (19.828)
  Week 16: number analyzed (Participants) | 17 | 21 | 8
  Week 16 | 21.06 (24.410) | 7.17 (19.121) | 17.50 (24.349)
  Week 20: number analyzed (Participants) | 8 | 6 | 5
  Week 20 | 15.15 (17.456) | 3.67 (5.715) | 19.00 (23.558)
  Week 24: number analyzed (Participants) | 15 | 18 | 5
  Week 24 | 8.33 (8.906) | 15.35 (25.202) | 22.76 (35.623)
  Week 28: number analyzed (Participants) | 5 | 5 | 4
  Week 28 | 12.32 (12.997) | 0.82 (1.834) | 9.25 (12.738)
  Week 32: number analyzed (Participants) | 13 | 17 | 3
  Week 32 | 12.69 (16.267) | 11.35 (20.568) | 18.27 (31.639)
  Week 36: number analyzed (Participants) | 5 | 5 | 4
  Week 36 | 14.50 (14.186) | 10.76 (10.143) | 5.73 (11.450)
  Week 40: number analyzed (Participants) | 15 | 18 | 3
  Week 40 | 11.01 (12.629) | 11.33 (21.941) | 6.67 (11.547)
  Week 44: number analyzed (Participants) | 6 | 6 | 4
  Week 44 | 21.93 (32.299) | 12.37 (23.664) | 7.08 (9.463)
  Week 48: number analyzed (Participants) | 12 | 15 | 6
  Week 48 | 10.36 (10.518) | 20.64 (28.599) | 20.55 (22.249)
  Week 52: number analyzed (Participants) | 15 | 16 | 3
  Week 52 | 17.91 (21.428) | 14.68 (23.128) | 10.00 (10.000)

81. Secondary Outcome: Percent Class Time Missed Using Work Productivity and Activity Impairment Questionnaire Plus Classroom Impairment Questions: DB Period
Description: WPAI+CIQ:10-item questionnaire to assess degree to which AD affected work productivity and regular activities over past 7 days. Questions: Q1=currently employed; Q2=work hours missed due to health problems; Q3=work hours missed due to other reasons; Q4=hours actually worked; Q5=degree health affected productivity while working(0-10 scale, high scores =less productivity); Q6=classes attended in academic setting or not;Q7=class hours missed due to health problems; Q8=class hours actually attended; Q9=degree health affected productivity while attending(0-10 scale, high scores= less productivity); Q10=degree health affected productivity in regular daily activities(0-10 scale, high scores =less productivity). Percent class time missed due to health problem calculated as: Q7*100/(Q7+Q8) and score ranged from 0-100% where higher numbers=greater impairment and less productivity.
Time Frame: as for outcome 65
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent class time missed
Arm/Group | Vehicle QD | Crisaborole 2% QD | Crisaborole 2% BID: Flare Period
Number analyzed (Participants) | 69 | 78 | 88
Percent class time missed
  Baseline: number analyzed (Participants) | 29 | 33 | 0
  Baseline | 0.04 (0.223) | 2.22 (9.030) |
  Week 4: number analyzed (Participants) | 12 | 22 | 15
  Week 4 | 0.89 (3.089) | 1.14 (5.330) | 5.96 (14.570)
  Week 8: number analyzed (Participants) | 12 | 19 | 12
  Week 8 | 0.00 (0.000) | 1.62 (6.735) | 7.95 (18.375)
  Week 12: number analyzed (Participants) | 8 | 18 | 7
  Week 12 | 11.36 (32.138) | 3.09 (11.781) | 7.14 (18.898)
  Week 16: number analyzed (Participants) | 9 | 14 | 7
  Week 16 | 0.00 (0.000) | 7.64 (23.561) | 0.81 (2.154)
  Week 20: number analyzed (Participants) | 7 | 9 | 4
  Week 20 | 7.79 (20.599) | 0.00 (0.000) | 25.00 (50.000)
  Week 24: number analyzed (Participants) | 8 | 20 | 4
  Week 24 | 0.00 (0.000) | 3.62 (9.881) | 0.00 (0.000)
  Week 28: number analyzed (Participants) | 5 | 7 | 7
  Week 28 | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
  Week 32: number analyzed (Participants) | 8 | 20 | 7
  Week 32 | 0.00 (0.000) | 5.83 (15.897) | 0.00 (0.000)
  Week 36: number analyzed (Participants) | 4 | 4 | 2
  Week 36 | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
  Week 40: number analyzed (Participants) | 5 | 14 | 0
  Week 40 | 0.00 (0.000) | 3.57 (13.363) |
  Week 44: number analyzed (Participants) | 5 | 6 | 3
  Week 44 | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
  Week 48: number analyzed (Participants) | 9 | 17 | 5
  Week 48 | 11.11 (33.333) | 0.00 (0.000) | 10.00 (22.361)
  Week 52: number analyzed (Participants) | 7 | 22 | 9
  Week 52 | 5.71 (15.119) | 9.09 (25.054) | 0.00 (0.000)

82. Secondary Outcome: Percent Impairment While in Class Using Work Productivity and Activity Impairment Questionnaire Plus Classroom Impairment Questions: DB Period
Description: WPAI+CIQ: 10-item questionnaire used to assess degree to which AD affected work productivity and regular activities over past 7 days. Questions: Q1=currently employed; Q2=work hours missed due to health problems; Q3=work hours missed due to other reasons; Q4=hours actually worked; Q5 = degree health affected productivity while working (0-10 scale, high scores=less productivity); Q6=classes attended in academic setting or not; Q7=class hours missed due to health problems; Q8=class hours actually attended; Q9=degree health affected productivity while attending(0-10 scale, high scores = less productivity); Q10=degree health affected productivity in regular daily activities (0-10 scale, high scores =less productivity). Percent impairment while in class was calculated as: 100*Q9/10 and score ranged from 0-100% where higher numbers indicate greater impairment and less productivity.
Time Frame: as for outcome 65
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent impairment while in class
Arm/Group | Vehicle QD | Crisaborole 2% QD | Crisaborole 2% BID: Flare Period
Number analyzed (Participants) | 69 | 78 | 88
Percent impairment while in class
  Baseline: number analyzed (Participants) | 29 | 33 | 0
  Baseline | 8.62 (14.072) | 7.88 (11.390) |
  Week 4: number analyzed (Participants) | 12 | 22 | 15
  Week 4 | 5.83 (12.401) | 6.36 (12.168) | 29.33 (26.583)
  Week 8: number analyzed (Participants) | 12 | 19 | 12
  Week 8 | 4.17 (7.930) | 5.79 (8.377) | 19.17 (23.916)
  Week 12: number analyzed (Participants) | 8 | 18 | 7
  Week 12 | 3.75 (7.440) | 2.22 (7.321) | 24.29 (17.182)
  Week 16: number analyzed (Participants) | 9 | 14 | 7
  Week 16 | 7.78 (16.415) | 8.57 (10.271) | 24.29 (29.358)
  Week 20: number analyzed (Participants) | 7 | 9 | 3
  Week 20 | 11.43 (16.762) | 11.11 (26.667) | 10.00 (10.000)
  Week 24: number analyzed (Participants) | 8 | 20 | 4
  Week 24 | 8.75 (18.077) | 4.00 (7.539) | 15.00 (23.805)
  Week 28: number analyzed (Participants) | 5 | 7 | 7
  Week 28 | 10.00 (22.361) | 7.14 (11.127) | 21.43 (21.157)
  Week 32: number analyzed (Participants) | 8 | 20 | 7
  Week 32 | 3.75 (10.607) | 3.50 (9.333) | 20.00 (25.166)
  Week 36: number analyzed (Participants) | 4 | 4 | 2
  Week 36 | 2.50 (5.000) | 2.50 (5.000) | 20.00 (28.284)
  Week 40: number analyzed (Participants) | 5 | 14 | 0
  Week 40 | 2.00 (4.472) | 8.57 (14.064) |
  Week 44: number analyzed (Participants) | 5 | 6 | 3
  Week 44 | 10.00 (14.142) | 6.67 (8.165) | 16.67 (5.774)
  Week 48: number analyzed (Participants) | 8 | 17 | 5
  Week 48 | 7.50 (13.887) | 7.06 (12.127) | 8.00 (8.367)
  Week 52: number analyzed (Participants) | 7 | 21 | 9
  Week 52 | 1.43 (3.780) | 7.62 (14.458) | 5.56 (8.819)

83. Secondary Outcome: Percent Overall Class Impairment Using Work Productivity and Activity Impairment Questionnaire Plus Classroom Impairment Questions: DB Period
Description: WPAI+CIQ: 10-item questionnaire to assess degree to which AD affected work productivity and regular activities over past 7 days. Questions: Q1=currently employed; Q2=work hours missed due to health problems; Q3=work hours missed due to other reasons; Q4=hours actually worked; Q5=degree health affected productivity while working (0-10 scale, high scores =less productivity); Q6=classes attended in academic setting or not; Q7=class hours missed due to health problems; Q8=class hours actually attended; Q9=degree health affected productivity while attending(0-10 scale, high scores = less productivity); Q10=degree health affected productivity in regular daily activities (0-10 scale, high scores =less productivity). Percent overall class impairment due to health problem calculated as: 100*{Q7/(Q7+Q8)+[(1- Q7/(Q7+Q8))×(Q9/10)]}, score range:0-100%, higher numbers=greater impairment and less productivity.
Time Frame: as for outcome 65
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent overall class impairment
Arm/Group | Vehicle QD | Crisaborole 2% QD | Crisaborole 2% BID: Flare Period
Number analyzed (Participants) | 69 | 78 | 88
Percent overall class impairment
  Baseline: number analyzed (Participants) | 29 | 33 | 0
  Baseline | 8.64 (14.136) | 10.10 (13.237) |
  Week 4: number analyzed (Participants) | 12 | 22 | 15
  Week 4 | 6.37 (14.034) | 7.50 (12.701) | 30.69 (27.265)
  Week 8: number analyzed (Participants) | 12 | 19 | 12
  Week 8 | 4.17 (7.930) | 7.40 (9.858) | 26.68 (25.384)
  Week 12: number analyzed (Participants) | 8 | 18 | 7
  Week 12 | 15.11 (31.477) | 5.28 (13.559) | 27.86 (24.471)
  Week 16: number analyzed (Participants) | 9 | 14 | 7
  Week 16 | 7.78 (16.415) | 14.06 (24.697) | 24.44 (29.707)
  Week 20: number analyzed (Participants) | 7 | 9 | 3
  Week 20 | 18.44 (24.535) | 11.11 (26.667) | 10.00 (10.000)
  Week 24: number analyzed (Participants) | 8 | 20 | 4
  Week 24 | 8.75 (18.077) | 7.20 (13.260) | 15.00 (23.805)
  Week 28: number analyzed (Participants) | 5 | 7 | 7
  Week 28 | 10.00 (22.361) | 7.14 (11.127) | 21.43 (21.157)
  Week 32: number analyzed (Participants) | 8 | 20 | 7
  Week 32 | 3.75 (10.607) | 9.06 (18.186) | 20.00 (25.166)
  Week 36: number analyzed (Participants) | 4 | 4 | 2
  Week 36 | 2.50 (5.000) | 2.50 (5.000) | 20.00 (28.284)
  Week 40: number analyzed (Participants) | 5 | 14 | 0
  Week 40 | 2.00 (4.472) | 11.79 (18.771) |
  Week 44: number analyzed (Participants) | 5 | 6 | 3
  Week 44 | 10.00 (14.142) | 6.67 (8.165) | 16.67 (5.774)
  Week 48: number analyzed (Participants) | 8 | 17 | 5
  Week 48 | 7.50 (13.887) | 7.06 (12.127) | 17.00 (22.804)
  Week 52: number analyzed (Participants) | 7 | 21 | 9
  Week 52 | 7.14 (14.960) | 11.90 (20.154) | 5.56 (8.819)

84. Secondary Outcome: Percent Activity Impairment Using Work Productivity and Activity Impairment Questionnaire Plus Classroom Impairment Questions: DB Period
Description: WPAI+CIQ:10-item questionnaire used to assess degree to which AD affected work productivity and regular activities over past 7 days. Questions: Q1=currently employed; Q2=work hours missed due to health problems; Q3=work hours missed due to other reasons; Q4=hours actually worked; Q5=degree health affected productivity while working (0-10 scale, high scores=less productivity); Q6=classes attended in academic setting or not; Q7=class hours missed due to health problems; Q8=class hours actually attended; Q9=degree health affected productivity while attending(0-10 scale, high scores= less productivity); Q10=degree health affected productivity in regular daily activities(0-10 scale, high scores =less productivity). Percent activity impairment due to health problem calculated as: 100*Q10/10, score ranged from 0-100%,higher numbers=greater impairment and less productivity.
Time Frame: as for outcome 65
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent activity impairment
Arm/Group | Vehicle QD | Crisaborole 2% QD | Crisaborole 2% BID: Flare Period
Number analyzed (Participants) | 69 | 78 | 88
Percent activity impairment
  Baseline: number analyzed (Participants) | 69 | 78 | 0
  Baseline | 8.99 (15.353) | 10.90 (16.763) |
  Week 4: number analyzed (Participants) | 32 | 51 | 51
  Week 4 | 10.31 (18.749) | 8.24 (13.222) | 15.88 (22.287)
  Week 8: number analyzed (Participants) | 36 | 50 | 38
  Week 8 | 8.61 (13.555) | 7.20 (12.784) | 16.58 (23.741)
  Week 12: number analyzed (Participants) | 32 | 49 | 32
  Week 12 | 10.31 (16.749) | 5.31 (13.087) | 13.44 (15.368)
  Week 16: number analyzed (Participants) | 42 | 52 | 21
  Week 16 | 10.00 (15.927) | 7.12 (14.731) | 16.19 (26.168)
  Week 20: number analyzed (Participants) | 21 | 21 | 11
  Week 20 | 16.19 (22.017) | 9.52 (21.089) | 13.64 (15.015)
  Week 24: number analyzed (Participants) | 37 | 47 | 14
  Week 24 | 8.38 (13.645) | 5.74 (12.810) | 16.43 (19.457)
  Week 28: number analyzed (Participants) | 18 | 17 | 14
  Week 28 | 11.67 (16.891) | 5.29 (12.805) | 22.14 (21.187)
  Week 32: number analyzed (Participants) | 34 | 45 | 13
  Week 32 | 9.12 (17.815) | 6.89 (14.744) | 26.92 (33.760)
  Week 36: number analyzed (Participants) | 17 | 17 | 7
  Week 36 | 11.18 (15.363) | 9.41 (13.449) | 7.14 (9.512)
  Week 40: number analyzed (Participants) | 34 | 47 | 8
  Week 40 | 10.59 (18.081) | 8.30 (17.235) | 8.75 (17.269)
  Week 44: number analyzed (Participants) | 18 | 17 | 11
  Week 44 | 13.33 (21.693) | 7.65 (16.781) | 16.36 (21.106)
  Week 48: number analyzed (Participants) | 30 | 43 | 12
  Week 48 | 11.00 (16.263) | 6.05 (13.997) | 10.00 (15.954)
  Week 52: number analyzed (Participants) | 32 | 43 | 15
  Week 52 | 7.50 (14.368) | 7.21 (15.480) | 8.00 (12.649)

85. Secondary Outcome: Percent Work Time Missed Using Work Productivity and Activity Impairment Questionnaire Plus Classroom Impairment Questions: First Flare Free Period
Description: WPAI+CIQ:10-item questionnaire used to assess degree to which AD affected work productivity and regular activities over past 7 days. Questions were: Q1=currently employed; Q2=work hours missed due to health problems;Q3=work hours missed due to other reasons; Q4=hours actually worked; Q5= degree health affected productivity while working (0-10 scale, high scores =less productivity); Q6=classes attended in academic setting or not; Q7=class hours missed due to health problems; Q8=class hours actually attended; Q9=degree health affected productivity while attending(0-10 scale, high scores = less productivity); Q10=degree health affected productivity in regular daily activities(0-10 scale, high scores =less productivity). Percent work time missed due to health problem calculated as: Q2*100/(Q2+Q4) and score ranged from 0-100%, higher numbers=greater impairment and less productivity.
Time Frame: as for outcome 65
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent work time missed
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 35 | 38
Percent work time missed
  Baseline | 4.77 (14.528) | 5.07 (14.128)
  Week 4: number analyzed (Participants) | 10 | 18
  Week 4 | 5.76 (15.662) | 5.54 (15.120)
  Week 8: number analyzed (Participants) | 9 | 14
  Week 8 | 7.50 (16.965) | 3.64 (13.604)
  Week 12: number analyzed (Participants) | 7 | 10
  Week 12 | 7.14 (18.898) | 5.77 (15.790)
  Week 16: number analyzed (Participants) | 7 | 14
  Week 16 | 23.49 (38.319) | 5.32 (13.142)
  Week 20: number analyzed (Participants) | 2 | 3
  Week 20 | 0.00 (0.000) | 0.73 (1.270)
  Week 24: number analyzed (Participants) | 7 | 10
  Week 24 | 0.34 (0.907) | 8.03 (18.722)
  Week 28: number analyzed (Participants) | 2 | 2
  Week 28 | 0.00 (0.000) | 2.05 (2.899)
  Week 32: number analyzed (Participants) | 6 | 11
  Week 32 | 11.75 (20.454) | 15.08 (31.936)
  Week 36: number analyzed (Participants) | 2 | 3
  Week 36 | 0.00 (0.000) | 1.40 (2.425)
  Week 40: number analyzed (Participants) | 7 | 11
  Week 40 | 0.69 (1.814) | 4.95 (15.001)
  Week 44: number analyzed (Participants) | 3 | 3
  Week 44 | 0.00 (0.000) | 1.40 (2.425)
  Week 48: number analyzed (Participants) | 7 | 10
  Week 48 | 1.79 (4.725) | 12.27 (21.541)
  Week 52: number analyzed (Participants) | 6 | 9
  Week 52 | 8.33 (20.412) | 3.33 (6.022)

86. Secondary Outcome: Percent Impairment While Working Using Work Productivity and Activity Impairment Questionnaire Plus Classroom Impairment Questions: First Flare Free Period
Description: WPAI+CIQ: 10-item questionnaire used to assess degree to which AD affected work productivity and regular activities over past 7 days. Questions: Q1=currently employed; Q2=hours missed due to health problems; Q3=hours missed due to other reasons; Q4=hours actually worked; Q5=degree health affected productivity while working (0-10 scale, high scores =less productivity); Q6=classes attended in academic setting or not; Q7=hours missed due to health problems; Q8=hours actually attended; Q9=degree health affected productivity while attending(0-10 scale, high scores = less productivity); Q10=degree health affected productivity in regular daily activities(0-10 scale, high scores =less productivity). Percent impairment while working due to health problem calculated as: 100*Q5/10 score ranged from 0-100%, higher numbers=greater impairment and less productivity.
Time Frame: as for outcome 65
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent impairment while work
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 35 | 38
Percent impairment while work
  Baseline | 9.71 (15.432) | 10.26 (17.474)
  Week 4: number analyzed (Participants) | 10 | 18
  Week 4 | 5.00 (12.693) | 10.56 (15.136)
  Week 8: number analyzed (Participants) | 9 | 14
  Week 8 | 4.44 (5.270) | 6.43 (13.927)
  Week 12: number analyzed (Participants) | 7 | 10
  Week 12 | 5.71 (7.868) | 12.00 (24.855)
  Week 16: number analyzed (Participants) | 6 | 14
  Week 16 | 8.33 (11.690) | 7.86 (17.177)
  Week 20: number analyzed (Participants) | 2 | 3
  Week 20 | 15.00 (21.213) | 6.67 (5.774)
  Week 24: number analyzed (Participants) | 7 | 10
  Week 24 | 8.57 (8.997) | 13.00 (25.408)
  Week 28: number analyzed (Participants) | 2 | 2
  Week 28 | 10.00 (14.142) | 0.00 (0.000)
  Week 32: number analyzed (Participants) | 6 | 10
  Week 32 | 8.33 (7.528) | 15.00 (19.003)
  Week 36: number analyzed (Participants) | 2 | 3
  Week 36 | 10.00 (14.142) | 10.00 (10.000)
  Week 40: number analyzed (Participants) | 7 | 11
  Week 40 | 12.86 (11.127) | 14.55 (23.394)
  Week 44: number analyzed (Participants) | 3 | 3
  Week 44 | 30.00 (43.589) | 23.33 (32.146)
  Week 48: number analyzed (Participants) | 7 | 10
  Week 48 | 11.43 (8.997) | 16.00 (24.585)
  Week 52: number analyzed (Participants) | 6 | 9
  Week 52 | 8.33 (7.528) | 15.56 (25.055)

87. Secondary Outcome: Percent Overall Work Impairment Using Work Productivity and Activity Impairment Questionnaire Plus Classroom Impairment Questions: First Flare Free Period
Description: WPAI+CIQ: 10-item questionnaire to assess degree to which AD affected work productivity and regular activities over past 7 days. Questions: Q1=currently employed; Q2=work hours missed due to health problems; Q3=work hours missed due to other reasons; Q4=hours actually worked; Q5=degree health affected productivity while working (0-10 scale, high scores =less productivity); Q6=classes attended in academic setting or not; Q7=class hours missed due to health problems; Q8=class hours actually attended; Q9=degree health affected productivity while attending (0-10 scale, high scores = less productivity); Q10=degree health affected productivity: regular daily activities(0-10 scale, high scores =less productivity). Percent overall impairment while working due to health problem calculated as:100*{Q2/(Q2+Q4)+[(1- Q2/(Q2+Q4))×(Q5/10)]}, score ranged:0-100%, high numbers=greater impairment and less productivity.
Time Frame: as for outcome 65
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent overall work impairment
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 35 | 38
Percent overall work impairment
  Baseline | 14.04 (19.991) | 14.29 (21.183)
  Week 4: number analyzed (Participants) | 10 | 18
  Week 4 | 10.74 (18.593) | 15.53 (20.088)
  Week 8: number analyzed (Participants) | 9 | 14
  Week 8 | 11.77 (16.662) | 10.06 (18.129)
  Week 12: number analyzed (Participants) | 7 | 10
  Week 12 | 11.43 (21.931) | 13.70 (27.729)
  Week 16: number analyzed (Participants) | 6 | 14
  Week 16 | 17.57 (23.791) | 10.75 (22.825)
  Week 20: number analyzed (Participants) | 2 | 3
  Week 20 | 15.00 (21.213) | 7.33 (6.429)
  Week 24: number analyzed (Participants) | 7 | 10
  Week 24 | 8.86 (9.442) | 19.63 (29.412)
  Week 28: number analyzed (Participants) | 2 | 2
  Week 28 | 10.00 (14.142) | 2.05 (2.899)
  Week 32: number analyzed (Participants) | 6 | 10
  Week 32 | 18.92 (20.929) | 18.29 (24.749)
  Week 36: number analyzed (Participants) | 2 | 3
  Week 36 | 10.00 (14.142) | 11.27 (10.238)
  Week 40: number analyzed (Participants) | 7 | 11
  Week 40 | 13.40 (11.616) | 15.82 (26.160)
  Week 44: number analyzed (Participants) | 3 | 3
  Week 44 | 30.00 (43.589) | 24.73 (30.679)
  Week 48: number analyzed (Participants) | 7 | 10
  Week 48 | 12.86 (11.127) | 23.46 (29.836)
  Week 52: number analyzed (Participants) | 6 | 9
  Week 52 | 15.83 (20.595) | 17.20 (25.996)

88. Secondary Outcome: Percent Class Time Missed Using Work Productivity and Activity Impairment Questionnaire Plus Classroom Impairment Questions: First Flare Free Period
Description: WPAI+CIQ:10-item questionnaire to assess degree to which AD affected work productivity and regular activities over past 7 days. Questions: Q1=currently employed; Q2=work hours missed due to health problems; Q3=work hours missed due to other reasons; Q4=hours actually worked; Q5=degree health affected productivity while working(0-10 scale, high scores =less productivity); Q6=classes attended in academic setting or not; Q7=class hours missed due to health problems; Q8=class hours actually attended; Q9=degree health affected productivity while attending(0-10 scale, high scores = less productivity); Q10=degree health affected productivity in regular daily activities(0-10 scale, high scores =less productivity). Percent class time missed due to health problem calculated as: Q7*100/(Q7+Q8) and score ranged from 0-100% where higher numbers=greater impairment and less productivity.
Time Frame: as for outcome 65
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent class time missed
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 29 | 33
Percent class time missed
  Baseline | 0.04 (0.223) | 2.22 (9.030)
  Week 4: number analyzed (Participants) | 11 | 22
  Week 4 | 0.97 (3.226) | 1.14 (5.330)
  Week 8: number analyzed (Participants) | 7 | 19
  Week 8 | 0.00 (0.000) | 1.62 (6.735)
  Week 12: number analyzed (Participants) | 4 | 17
  Week 12 | 0.00 (0.000) | 3.27 (12.118)
  Week 16: number analyzed (Participants) | 4 | 13
  Week 16 | 0.00 (0.000) | 8.22 (24.416)
  Week 20: number analyzed (Participants) | 1 | 7
  Week 20 | 0.00 (NA) — Standard deviation could not be estimated due to less number of participants with events. | 0.00 (0.000)
  Week 24: number analyzed (Participants) | 2 | 14
  Week 24 | 0.00 (0.000) | 0.71 (2.673)
  Week 28: number analyzed (Participants) | 0 | 4
  Week 28 |  | 0.00 (0.000)
  Week 32: number analyzed (Participants) | 2 | 13
  Week 32 | 0.00 (0.000) | 8.97 (19.226)
  Week 36: number analyzed (Participants) | 0 | 2
  Week 36 |  | 0.00 (0.000)
  Week 40: number analyzed (Participants) | 2 | 8
  Week 40 | 0.00 (0.000) | 0.00 (0.000)
  Week 44: number analyzed (Participants) | 1 | 3
  Week 44 | 0.00 (NA) — Standard deviation could not be estimated due to less number of participants with events. | 0.00 (0.000)
  Week 48: number analyzed (Participants) | 4 | 9
  Week 48 | 0.00 (0.000) | 0.00 (0.000)
  Week 52: number analyzed (Participants) | 2 | 9
  Week 52 | 0.00 (0.000) | 0.00 (0.000)

89. Secondary Outcome: Percent Impairment While in Class Using Work Productivity and Activity Impairment Questionnaire Plus Classroom Impairment Questions: First Flare Free Period
Description: WPAI+CIQ:10-item questionnaire used to assess degree to which AD affected work productivity and regular activities over past 7 days. Questions: Q1=currently employed; Q2=work hours missed due to health problems; Q3=work hours missed due to other reasons; Q4=hours actually worked; Q5 = degree health affected productivity while working (0-10 scale, high scores =less productivity); Q6=classes attended in academic setting or not; Q7=class hours missed due to health problems; Q8=class hours actually attended; Q9=degree health affected productivity while attending (0-10 scale, high scores = less productivity); Q10=degree health affected productivity in regular daily activities(0-10 scale, high scores =less productivity). Percent impairment while in class was calculated as: 100*Q9/10 and score ranged from 0-100% where higher numbers indicate greater impairment and less productivity.
Time Frame: as for outcome 65
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent impairment while in class
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 29 | 33
Percent impairment while in class
  Baseline | 8.62 (14.072) | 7.88 (11.390)
  Week 4: number analyzed (Participants) | 11 | 22
  Week 4 | 6.36 (12.863) | 6.36 (12.168)
  Week 8: number analyzed (Participants) | 7 | 19
  Week 8 | 1.43 (3.780) | 5.79 (8.377)
  Week 12: number analyzed (Participants) | 4 | 17
  Week 12 | 5.00 (10.000) | 2.35 (7.524)
  Week 16: number analyzed (Participants) | 4 | 13
  Week 16 | 2.50 (5.000) | 8.46 (10.682)
  Week 20: number analyzed (Participants) | 1 | 7
  Week 20 | 0.00 (NA) — Standard deviation could not be estimated due to less number of participants with events. | 14.29 (29.921)
  Week 24: number analyzed (Participants) | 2 | 14
  Week 24 | 10.00 (14.142) | 2.86 (6.112)
  Week 28: number analyzed (Participants) | 0 | 4
  Week 28 |  | 10.00 (14.142)
  Week 32: number analyzed (Participants) | 2 | 13
  Week 32 | 0.00 (0.000) | 3.85 (11.209)
  Week 36: number analyzed (Participants) | 0 | 2
  Week 36 |  | 5.00 (7.071)
  Week 40: number analyzed (Participants) | 2 | 8
  Week 40 | 5.00 (7.071) | 6.25 (9.161)
  Week 44: number analyzed (Participants) | 1 | 3
  Week 44 | 20.00 (NA) — Standard deviation could not be estimated due to less number of participants with events. | 10.00 (10.000)
  Week 48: number analyzed (Participants) | 4 | 9
  Week 48 | 7.50 (15.000) | 5.56 (11.304)
  Week 52: number analyzed (Participants) | 2 | 9
  Week 52 | 0.00 (0.000) | 3.33 (7.071)

90. Secondary Outcome: Percent Overall Class Impairment Using Work Productivity and Activity Impairment Questionnaire Plus Classroom Impairment Questions: First Flare Free Period
Description: WPAI+CIQ:10-item questionnaire to assess degree to which AD affected work productivity and regular activities over past 7 days. Questions: Q1=currently employed; Q2=work hours missed due to health problems; Q3=work hours missed due to other reasons; Q4=hours actually worked; Q5=degree health affected productivity while working (0-10 scale, high scores =less productivity); Q6=classes attended in academic setting or not; Q7=class hours missed due to health problems; Q8=class hours actually attended; Q9=degree health affected productivity while attending(0-10 scale, high scores = less productivity); Q10=degree health affected productivity in regular daily activities (0-10 scale, high scores =less productivity). Percent overall class impairment due to health problem calculated as: 100*{Q7/(Q7+Q8)+[(1- Q7/(Q7+Q8))×(Q9/10)]}, score range:0-100%,higher numbers=greater impairment and less productivity.
Time Frame: as for outcome 65
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent overall class impairment
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 29 | 33
Percent overall class impairment
  Baseline | 8.64 (14.136) | 10.10 (13.237)
  Week 4: number analyzed (Participants) | 11 | 22
  Week 4 | 6.95 (14.568) | 7.50 (12.701)
  Week 8: number analyzed (Participants) | 7 | 19
  Week 8 | 1.43 (3.780) | 7.40 (9.858)
  Week 12: number analyzed (Participants) | 4 | 17
  Week 12 | 5.00 (10.000) | 5.59 (13.910)
  Week 16: number analyzed (Participants) | 4 | 13
  Week 16 | 2.50 (5.000) | 14.37 (25.677)
  Week 20: number analyzed (Participants) | 1 | 7
  Week 20 | 0.00 (NA) — Standard deviation could not be estimated due to less number of participants with events. | 14.29 (29.921)
  Week 24: number analyzed (Participants) | 2 | 14
  Week 24 | 10.00 (14.142) | 3.50 (7.283)
  Week 28: number analyzed (Participants) | 0 | 4
  Week 28 |  | 10.00 (14.142)
  Week 32: number analyzed (Participants) | 2 | 13
  Week 32 | 0.00 (0.000) | 12.39 (21.847)
  Week 36: number analyzed (Participants) | 0 | 2
  Week 36 |  | 5.00 (7.071)
  Week 40: number analyzed (Participants) | 2 | 8
  Week 40 | 5.00 (7.071) | 6.25 (9.161)
  Week 44: number analyzed (Participants) | 1 | 3
  Week 44 | 20.00 (NA) — Standard deviation could not be estimated due to less number of participants with events. | 10.00 (10.000)
  Week 48: number analyzed (Participants) | 4 | 9
  Week 48 | 7.50 (15.000) | 5.56 (11.304)
  Week 52: number analyzed (Participants) | 2 | 9
  Week 52 | 0.00 (0.000) | 3.33 (7.071)

91. Secondary Outcome: Percent Activity Impairment Using Work Productivity and Activity Impairment Questionnaire Plus Classroom Impairment Questions: First Flare Free Period
Description: WPAI+CIQ:10-item questionnaire used to assess degree to which AD affected work productivity and regular activities over past 7 days. Questions: Q1=currently employed; Q2=work hours missed due to health problems; Q3=work hours missed due to other reasons; Q4=hours actually worked; Q5=degree health affected productivity while working (0-10 scale, high scores =less productivity); Q6=classes attended in academic setting or not; Q7=class hours missed due to health problems; Q8=class hours actually attended; Q9=degree health affected productivity while attending (0-10 scale, high scores = less productivity); Q10=degree health affected productivity in regular daily activities(0-10 scale, high scores =less productivity). Percent activity impairment due to health problem calculated as: 100*Q10/10, score ranged from 0-100%,higher numbers=greater impairment and less productivity.
Time Frame: as for outcome 65
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent activity impairment
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 69 | 78
Percent activity impairment
  Baseline | 8.99 (15.353) | 10.90 (16.763)
  Week 4: number analyzed (Participants) | 30 | 51
  Week 4 | 11.00 (19.182) | 8.24 (13.222)
  Week 8: number analyzed (Participants) | 25 | 44
  Week 8 | 10.00 (15.275) | 7.27 (13.005)
  Week 12: number analyzed (Participants) | 20 | 40
  Week 12 | 10.50 (18.202) | 5.50 (13.765)
  Week 16: number analyzed (Participants) | 19 | 37
  Week 16 | 8.95 (15.949) | 8.11 (15.958)
  Week 20: number analyzed (Participants) | 8 | 13
  Week 20 | 15.00 (16.903) | 9.23 (22.159)
  Week 24: number analyzed (Participants) | 17 | 31
  Week 24 | 8.24 (13.339) | 5.81 (13.850)
  Week 28: number analyzed (Participants) | 7 | 9
  Week 28 | 17.14 (17.995) | 3.33 (7.071)
  Week 32: number analyzed (Participants) | 16 | 27
  Week 32 | 11.88 (22.574) | 8.52 (17.255)
  Week 36: number analyzed (Participants) | 6 | 7
  Week 36 | 15.00 (13.784) | 8.57 (8.997)
  Week 40: number analyzed (Participants) | 17 | 26
  Week 40 | 12.35 (17.864) | 7.31 (16.385)
  Week 44: number analyzed (Participants) | 7 | 9
  Week 44 | 15.71 (17.182) | 8.89 (16.915)
  Week 48: number analyzed (Participants) | 17 | 24
  Week 48 | 11.18 (16.539) | 7.50 (16.485)
  Week 52: number analyzed (Participants) | 15 | 23
  Week 52 | 12.00 (17.403) | 6.52 (16.951)

92. Secondary Outcome: Percent Work Time Missed Using Work Productivity and Activity Impairment Questionnaire Plus Classroom Impairment Questions: First Flare Period
Description: WPAI+CIQ:10-item questionnaire used to assess degree to which AD affected work productivity and regular activities over past 7 days. Questions were: Q1=currently employed; Q2=work hours missed due to health problems; Q3=work hours missed due to other reasons; Q4=hours actually worked; Q5 = degree health affected productivity while working (0-10 scale, high scores =less productivity); Q6=classes attended in academic setting or not; Q7=class hours missed due to health problems; Q8=class hours actually attended; Q9=degree health affected productivity while attending (0-10 scale, high scores = less productivity); Q10=degree health affected productivity in regular daily activities (0-10 scale, high scores=less productivity). Percent work time missed due to health problem calculated as: Q2*100/(Q2+Q4) and score ranged from 0-100%, higher numbers=greater impairment and less productivity.
Time Frame: Weeks 0, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent work time missed
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 19 | 15
Percent work time missed
  Week 0 | 5.46 (14.226) | 6.99 (18.460)
  Week 4: number analyzed (Participants) | 10 | 5
  Week 4 | 1.49 (3.188) | 0.00 (0.000)
  Week 8: number analyzed (Participants) | 5 | 2
  Week 8 | 2.36 (5.277) | 0.00 (0.000)
  Week 12: number analyzed (Participants) | 2 | 1
  Week 12 | 34.40 (48.649) | 0.00 (NA) — Standard deviation could not be estimated due to less number of participants with events.

93. Secondary Outcome: Percent Impairment While Working Using Work Productivity and Activity Impairment Questionnaire Plus Classroom Impairment Questions: First Flare Period
Description: WPAI+CIQ: 10-item questionnaire used to assess degree to which AD affected work productivity and regular activities over past 7 days. Questions were: Q1=currently employed; Q2=hours missed due to health problems; Q3=hours missed due to other reasons; Q4=hours actually worked; Q5=degree health affected productivity while working (0-10 scale, high scores =less productivity); Q6=classes attended in academic setting or not; Q7=hours missed due to health problems; Q8=hours actually attended; Q9=degree health affected productivity while attending(0-10 scale, high scores = less productivity); Q10=degree health affected productivity in regular daily activities (0-10 scale, high scores =less productivity). Percent impairment while working due to health problem calculated as: 100*Q5/10 score ranged from 0-100%, higher numbers=greater impairment and less productivity.
Time Frame: Weeks 0, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent impairment while work
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 19 | 15
Percent impairment while work
  Week 0 | 11.05 (14.868) | 16.67 (31.547)
  Week 4: number analyzed (Participants) | 10 | 5
  Week 4 | 12.00 (18.738) | 10.00 (10.000)
  Week 8: number analyzed (Participants) | 5 | 2
  Week 8 | 8.00 (17.889) | 15.00 (21.213)
  Week 12: number analyzed (Participants) | 2 | 1
  Week 12 | 50.00 (14.142) | 0.00 (NA) — Standard deviation could not be estimated due to less number of participants with events.

94. Secondary Outcome: Percent Overall Work Impairment Using Work Productivity and Activity Impairment Questionnaire Plus Classroom Impairment Questions: First Flare Period
Description: WPAI+CIQ: 10-item questionnaire to assess degree to which AD affected work productivity and regular activities over past 7 days. Questions were: Q1=currently employed; Q2=work hours missed due to health problems; Q3=work hours missed due to other reasons; Q4=hours actually worked; Q5=degree health affected productivity while working(0-10 scale, high scores =less productivity); Q6=classes attended in academic setting or not; Q7=class hours missed due to health problems; Q8=class hours actually attended; Q9=degree health affected productivity while attending (0-10 scale, high scores = less productivity); Q10=degree health affected productivity in regular daily activities(0-10 scale, high scores =less productivity). Percent overall impairment while working due to health problem calculated as:100*{Q2/(Q2+Q4)+[(1- Q2/(Q2+Q4))×(Q5/10)]}, score ranged:0-100%, high numbers=greater impairment and less productivity.
Time Frame: Weeks 0, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent overall work impairment
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 19 | 15
Percent overall work impairment
  Week 0 | 16.21 (18.311) | 20.32 (32.634)
  Week 4: number analyzed (Participants) | 10 | 5
  Week 4 | 13.40 (18.431) | 10.00 (10.000)
  Week 8: number analyzed (Participants) | 5 | 2
  Week 8 | 10.36 (17.339) | 15.00 (21.213)
  Week 12: number analyzed (Participants) | 2 | 1
  Week 12 | 70.65 (15.061) | 0.00 (NA) — Standard deviation could not be estimated due to less number of participants with events.

95. Secondary Outcome: Percent Class Time Missed Using Work Productivity and Activity Impairment Questionnaire Plus Classroom Impairment Questions: First Flare Period
Description: WPAI+CIQ:10-item questionnaire to assess degree to which AD affected work productivity and regular activities over past 7 days. Questions were: Q1=currently employed; Q2=work hours missed due to health problems; Q3=work hours missed due to other reasons; Q4=hours actually worked; Q5=degree health affected productivity while working (0-10 scale, high scores =less productivity); Q6=classes attended in academic setting or not; Q7=class hours missed due to health problems; Q8=class hours actually attended; Q9=degree health affected productivity while attending(0-10 scale, high scores = less productivity); Q10=degree health affected productivity in regular daily activities(0-10 scale, high scores =less productivity). Percent class time missed due to health problem calculated as: Q7*100/(Q7+Q8) and score ranged from 0-100% where higher numbers=greater impairment and less productivity.
Time Frame: Weeks 0, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent class time missed
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 13 | 16
Percent class time missed
  Week 0 | 3.98 (12.314) | 11.53 (27.668)
  Week 4: number analyzed (Participants) | 6 | 12
  Week 4 | 0.00 (0.000) | 6.82 (16.215)
  Week 8: number analyzed (Participants) | 2 | 6
  Week 8 | 0.00 (0.000) | 8.33 (20.412)
  Week 12: number analyzed (Participants) | 0 | 4
  Week 12 |  | 1.43 (2.850)

96. Secondary Outcome: Percent Impairment While in Class Using Work Productivity and Activity Impairment Questionnaire Plus Classroom Impairment Questions: First Flare Period
Description: WPAI+CIQ:10-item questionnaire used to assess degree to which AD affected work productivity and regular activities over past 7 days. Questions:Q1=currently employed;Q2=work hours missed due to health problems;Q3=work hours missed due to other reasons;Q4=hours actually worked; Q5 = degree health affected productivity while working (0-10 scale, high scores =less productivity); Q6=classes attended in academic setting or not;Q7=class hours missed due to health problems;Q8=class hours actually attended;Q9=degree health affected productivity while attending(0-10 scale, high scores = less productivity);Q10=degree health affected productivity in regular daily activities(0-10 scale, high scores =less productivity). Percent impairment while in class was calculated as: 100*Q9/10 and score ranged from 0-100% where higher numbers indicate greater impairment and less productivity.
Time Frame: Weeks 0, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent impairment while in class
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 13 | 15
Percent impairment while in class
  Week 0 | 13.85 (17.578) | 24.67 (28.999)
  Week 4: number analyzed (Participants) | 6 | 12
  Week 4 | 16.67 (13.663) | 25.00 (25.761)
  Week 8: number analyzed (Participants) | 2 | 6
  Week 8 | 30.00 (14.142) | 30.00 (26.077)
  Week 12: number analyzed (Participants) | 0 | 4
  Week 12 |  | 40.00 (28.284)

97. Secondary Outcome: Percent Overall Class Impairment Using Work Productivity and Activity Impairment Questionnaire Plus Classroom Impairment Questions: First Flare Period
Description: WPAI+CIQ:10-item questionnaire to assess degree to which AD affected work productivity and regular activities over past 7 days. Questions were: Q1=currently employed; Q2=work hours missed due to health problems; Q3=work hours missed due to other reasons; Q4=hours actually worked; Q5=degree health affected productivity while working (0-10 scale, high scores =less productivity); Q6=classes attended in academic setting or not; Q7=class hours missed due to health problems; Q8=class hours actually attended; Q9=degree health affected productivity while attending (0-10 scale, high scores = less productivity); Q10=degree health affected productivity in regular daily activities(0-10 scale, high scores =less productivity). Percent overall class impairment due to health problem calculated as: 100*{Q7/(Q7+Q8)+[(1- Q7/(Q7+Q8))×(Q9/10)]}, score range:0-100%, higher numbers=greater impairment and less productivity.
Time Frame: Weeks 0, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent overall class impairment
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 13 | 15
Percent overall class impairment
  Week 0 | 17.49 (19.742) | 25.60 (30.354)
  Week 4: number analyzed (Participants) | 6 | 12
  Week 4 | 16.67 (13.663) | 30.21 (26.983)
  Week 8: number analyzed (Participants) | 2 | 6
  Week 8 | 30.00 (14.142) | 34.17 (31.371)
  Week 12: number analyzed (Participants) | 0 | 4
  Week 12 |  | 40.28 (28.803)

98. Secondary Outcome: Percent Activity Impairment Using Work Productivity and Activity Impairment Questionnaire Plus Classroom Impairment Questions: First Flare Period
Description: WPAI+CIQ:10-item questionnaire used to assess degree to which AD affected work productivity and regular activities over past 7 days. Questions: Q1=currently employed; Q2=work hours missed due to health problems; Q3=work hours missed due to other reasons; Q4=hours actually worked; Q5=degree health affected productivity while working (0-10 scale, high scores =less productivity); Q6=classes attended in academic setting or not; Q7=class hours missed due to health problems; Q8=class hours actually attended; Q9=degree health affected productivity while attending(0-10 scale, high scores = less productivity);Q10=degree health affected productivity in regular daily activities(0-10 scale, high scores =less productivity). Percent activity impairment due to health problem calculated as: 100*Q10/10, scores ranged from 0-100%,higher numbers=greater impairment and less productivity.
Time Frame: Weeks 0, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent activity impairment
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 43 | 44
Percent activity impairment
  Week 0 | 14.88 (20.745) | 17.27 (23.164)
  Week 4: number analyzed (Participants) | 21 | 24
  Week 4 | 15.24 (20.401) | 19.17 (21.653)
  Week 8: number analyzed (Participants) | 13 | 15
  Week 8 | 13.85 (17.578) | 26.00 (28.486)
  Week 12: number analyzed (Participants) | 3 | 7
  Week 12 | 16.67 (20.817) | 31.43 (29.681)

99. Secondary Outcome: Total Anxiety and Depression Scores Measured Using Hospital Anxiety and Depression Scale (HADS): OL Run-in Period
Description: HADS was a validated 14-item questionnaire to assess states of anxiety and depression over the past week. HADS consisted of 2 subscales: HADS-anxiety (HADS-A) and HADS-depression (HADS-D), each of which comprised of 7 items. Each item was rated on a 4-point scale, with scores ranging from 0 to 3, where higher scores indicated more anxiety/depression symptoms. HADS-A assessed state of generalized anxiety. HADS-A total score = sum of all 7 items with score ranging from 0 (no presence of anxiety) to 21 (severe feeling of anxiety); higher score indicated greater severity of anxiety. HADS-D assessed the state of lost interest and diminished pleasure response. HADS-D total score = sum of all 7 items with score ranging from 0 (no presence of depression) to 21 (severe feeling of depression); higher score indicated greater severity of depression symptoms.
Time Frame: Baseline (last observation up to and including Day 1 of OL period), Weeks 2, 4, 6 and 8
Population: as for outcome 49
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crisaborole 2% BID
Number analyzed (Participants) | 270
Units on a scale
  Anxiety: Baseline | 5.3 (3.70) [lower limit 3.70]
  Anxiety: Week 2 | 5.3 (3.73) [lower limit 3.73]
  Anxiety: Week 4 | 5.3 (3.72) [lower limit 3.72]
  Anxiety: Week 6 | 5.4 (3.79) [lower limit 3.79]
  Anxiety: Week 8 | 5.4 (3.81) [lower limit 3.81]
  Depression: Baseline | 3.2 (3.09) [lower limit 3.09]
  Depression: Week 2 | 3.2 (3.09) [lower limit 3.09]
  Depression: Week 4 | 3.2 (3.11) [lower limit 3.11]
  Depression: Week 6 | 3.3 (3.16) [lower limit 3.16]
  Depression: Week 8 | 3.3 (3.21) [lower limit 3.21]

100. Secondary Outcome: Total Anxiety and Depression Scores Measured Using Hospital Anxiety and Depression Scale: DB Period
Description: HADS was a validated 14-item questionnaire to assess states of anxiety and depression over the past week. HADS consisted of 2 subscales: HADS-A and HADS-D, each of which comprised of 7 items. Each item was rated on a 4-point scale, with scores ranging from 0 to 3, where higher scores indicated more anxiety/depression symptoms. HADS-A assessed state of generalized anxiety. HADS-A total score = sum of all 7 items with score ranging from 0 (no presence of anxiety) to 21 (severe feeling of anxiety); higher score indicated greater severity of anxiety. HADS-D assessed the state of lost interest and diminished pleasure response. HADS-D total score = sum of all 7 items with score ranging from 0 (no presence of depression) to 21 (severe feeling of depression); higher score indicated greater severity of depression symptoms.
Time Frame: Baseline (last observation up to and including randomization day), Week 8, 16, 32 and end of treatment [Week 52]
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD | Crisaborole 2% BID: Flare Period
Number analyzed (Participants) | 66 | 77 | 25
Units on a scale
  Anxiety: Baseline: number analyzed (Participants) | 66 | 77 | 0
  Anxiety: Baseline | 4.5 (3.50) | 4.5 (3.59) |
  Anxiety: Week 8: number analyzed (Participants) | 31 | 50 | 6
  Anxiety: Week 8 | 3.6 (3.23) | 4.5 (3.09) | 3.8 (2.71)
  Anxiety: Week 16: number analyzed (Participants) | 38 | 48 | 3
  Anxiety: Week 16 | 4.6 (3.83) | 4.7 (3.58) | 3.0 (2.65)
  Anxiety: Week 32: number analyzed (Participants) | 35 | 47 | 2
  Anxiety: Week 32 | 3.3 (3.42) | 4.4 (4.00) | 4.0 (5.66)
  Anxiety: End of treatment: number analyzed (Participants) | 35 | 49 | 19
  Anxiety: End of treatment | 4.0 (3.95) | 4.7 (3.62) | 4.7 (2.91)
  Depression: Baseline: number analyzed (Participants) | 66 | 77 | 0
  Depression: Baseline | 2.7 (2.36) | 2.8 (2.94) |
  Depression: Week 8: number analyzed (Participants) | 31 | 50 | 6
  Depression: Week 8 | 2.1 (2.00) | 2.5 (2.65) | 2.2 (1.72)
  Depression: Week 16: number analyzed (Participants) | 38 | 48 | 3
  Depression: Week 16 | 2.9 (2.65) | 3.5 (3.76) | 1.3 (1.53)
  Depression: Week 32: number analyzed (Participants) | 35 | 47 | 2
  Depression: Week 32 | 2.6 (2.82) | 3.3 (3.76) | 3.5 (3.54)
  Depression: End of treatment: number analyzed (Participants) | 35 | 49 | 19
  Depression: End of treatment | 2.8 (2.77) | 3.4 (3.23) | 2.6 (2.91)

101. Secondary Outcome: Total Anxiety and Depression Scores Measured Using Hospital Anxiety and Depression Scale: First Flare Period
Description: as for outcome 100
Time Frame: Weeks 0, 4, 8 and 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 15 | 18
Units on a scale
  Anxiety: Week 0: number analyzed (Participants) | 11 | 14
  Anxiety: Week 0 | 3.7 (3.52) | 4.9 (3.70)
  Anxiety: Week 4 | 4.3 (3.46) | 5.8 (4.19)
  Anxiety: Week 8: number analyzed (Participants) | 4 | 5
  Anxiety: Week 8 | 4.3 (1.89) | 8.0 (5.24)
  Anxiety: Week 12: number analyzed (Participants) | 3 | 6
  Anxiety: Week 12 | 6.0 (1.00) | 5.0 (4.73)
  Depression: Week 0: number analyzed (Participants) | 11 | 14
  Depression: Week 0 | 2.4 (3.07) | 2.5 (3.16)
  Depression: Week 4 | 3.1 (2.79) | 4.2 (5.19)
  Depression: Week 8: number analyzed (Participants) | 4 | 5
  Depression: Week 8 | 1.3 (1.26) | 4.8 (4.44)
  Depression: Week 12: number analyzed (Participants) | 3 | 6
  Depression: Week 12 | 1.0 (1.00) | 3.3 (2.16)

102. Secondary Outcome: Total Anxiety and Depression Scores Measured Using Hospital Anxiety and Depression Scale: First Flare Free Period
Description: as for outcome 100
Time Frame: Baseline (last observation up to and including the randomization day of DB period), Weeks 8, 16 and 32
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle QD | Crisaborole 2% QD
Number analyzed (Participants) | 66 | 77
Units on a scale
  Anxiety: Baseline | 4.5 (3.50) | 4.5 (3.59)
  Anxiety: Week 8: number analyzed (Participants) | 25 | 44
  Anxiety: Week 8 | 3.8 (3.28) | 4.1 (2.74)
  Anxiety: Week 16: number analyzed (Participants) | 19 | 38
  Anxiety: Week 16 | 3.9 (3.38) | 4.3 (3.49)
  Anxiety: Week 32: number analyzed (Participants) | 17 | 28
  Anxiety: Week 32 | 2.9 (2.47) | 4.2 (3.79)
  Depression: Baseline | 2.7 (2.36) | 2.8 (2.94)
  Depression: Week 8: number analyzed (Participants) | 25 | 44
  Depression: Week 8 | 2.2 (2.13) | 2.2 (2.29)
  Depression: Week 16: number analyzed (Participants) | 19 | 38
  Depression: Week 16 | 2.1 (1.91) | 3.1 (3.46)
  Depression: Week 32: number analyzed (Participants) | 17 | 28
  Depression: Week 32 | 1.9 (2.22) | 3.0 (3.00)

ADVERSE EVENTS:
Time Frame: From start of study intervention up to 8 weeks of OL period (OL: Crisaborole 2% BID arm); From start of study intervention in DB period to 28 days after last dose of study intervention (Up to 56 weeks) for DB: vehicle QD and DB: Crisaborole 2% QD arms
Description: Same event may appear as both AE and SAE, but are distinct events. An event may be categorized as serious in 1 participant and non-serious in another, or a participant may have experienced both SAE and non-SAE. Safety population comprised of all participants who received at least 1 dose of study intervention during the study.
Groups:
- OL: Crisaborole 2% BID: Participants with mild to moderate AD were administered crisaborole 2% ointment applied topically BID for maximum duration of up to 8 weeks in OL run-in period
- DB: Vehicle: Participants identified as responders during the OL period were randomized to receive vehicle applied topically QD for 52 weeks in the DB maintenance period. If a participant developed flares during the DB maintenance period, the participant was switched to receive flare rescue treatment with crisaborole 2% ointment BID in an open-label manner until resolution of flares following which DB treatment with vehicle was resumed.
- DB: Crisaborole 2% QD: Participants identified as responders during the OL period were randomized to receive crisaborole 2% ointment applied topically QD for 52 weeks in the DB maintenance period. If a participant developed flares during the DB maintenance period, the participant was switched to receive flare rescue treatment with crisaborole 2% ointment BID in an open-label manner until resolution of flares following which DB treatment with crisaborole 2% QD was resumed.
- DB Flare: Vehicle: Participants with an onset of flare (ISGA>=2) during DB maintenance period were switched to receive open-label crisaborole ointment 2%BID for up to 12 weeks until resolution of flares and resumption of DB maintenance treatment.
- DB Flare: Crisaborole 2% QD: Participants with an onset of flare (ISGA>=2) during DB maintenance period were switched to receive open-label crisaborole ointment 2% BID for up to 12 weeks until resolution of flares and resumption of DB maintenance treatment.
Arm/Group | OL: Crisaborole 2% BID | DB: Vehicle | DB: Crisaborole 2% QD | DB Flare: Vehicle | DB Flare: Crisaborole 2% QD
All-Cause Mortality (participants affected / at risk) | 0/497 | 0/135 | 0/135 | 0/89 | 0/78
Serious Adverse Events (participants affected / at risk) | 3/497 | 3/135 | 2/135 | 1/89 | 1/78
Other Adverse Events (participants affected / at risk) | 78/497 | 30/135 | 27/135 | 22/89 | 14/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OL: Crisaborole 2% BID (N=497) | DB: Vehicle (N=135) | DB: Crisaborole 2% QD (N=135) | DB Flare: Vehicle (N=89) | DB Flare: Crisaborole 2% QD (N=78)
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Application site infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Foreign body ingestion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
Paternal exposure during pregnancy (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OL: Crisaborole 2% BID (N=497) | DB: Vehicle (N=135) | DB: Crisaborole 2% QD (N=135) | DB Flare: Vehicle (N=89) | DB Flare: Crisaborole 2% QD (N=78)
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0
Application site erythema (General disorders) | 5 | 1 | 0 | 0 | 0
Application site pain (General disorders) | 28 | 2 | 0 | 1 | 1
Application site pruritus (General disorders) | 5 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 1 | 1 | 0
Allergy to animal (Immune system disorders) | 1 | 1 | 0 | 1 | 0
Application site infection (Infections and infestations) | 6 | 2 | 1 | 3 | 1
Bronchitis (Infections and infestations) | 2 | 3 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 5 | 1 | 1
Conjunctivitis (Infections and infestations) | 1 | 1 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 2 | 1 | 1 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 2 | 1 | 0
Influenza (Infections and infestations) | 4 | 1 | 3 | 0 | 0
Nasopharyngitis (Infections and infestations) | 4 | 5 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 2 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 2 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 10 | 2 | 4 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 1 | 0
Viral infection (Infections and infestations) | 2 | 2 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 3 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 12 | 3 | 0 | 2 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4 | 2 | 1 | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 4 | 1 | 1 | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Teething (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Application site acne (General disorders) | 0 | 0 | 0 | 0 | 1
Developmental delay (General disorders) | 0 | 0 | 0 | 1 | 0
Food allergy (Immune system disorders) | 3 | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Application site cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Tonsillitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 2 | 0 | 1 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Radial head dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/92/NCT04040192/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT04040192/SAP_001.pdf